# Statistical Analysis Plan

**Study ID:** 201791

**Official Title of Study:** Reporting and Analysis Plan for a 52-week, phase 3, multicentre, randomised, double blind, efficacy and safetystudy, comparing GSK3196165 with placebo and with tofacitinib in combination with conventional synthetic DMARDs, in participants with moderately to severely active rheumatoid arthritis who have an inadequate response to conventional synthetic DMARDs or biologic DMARDs.

**Date of Document:** 05 Aug 2022

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a 52-week, phase 3, multicentre, randomised, double blind, efficacy and safety study, comparing GSK3196165 with placebo and with tofacitinib in combination with conventional synthetic DMARDs, in participants with moderately to severely active rheumatoid arthritis who have an inadequate response to conventional synthetic DMARDs or biologic DMARDs. |
|---|---|---|
| <b>Compound Number</b> | : | GSK3196165 |
| <b>Compound Name</b> | : | Otilimab |
| <b>Effective Date</b> | : | 04 Aug 2022 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2018N385740\_02.
- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

# RAP Author(s):

| Approver | Date |
|-----------------------------------|-------------------|
| PPD | Refer to Document |
| Statistics Leader (Biostatistics) | Date |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **Biostatistics Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD (Biostatistics) | Refer to Document Date | eSignature |
| PPD Programming Leader (Biostatistics) | Refer to Document Date | eSignature |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| | 1.1. | RAP Amendments | 6 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 6 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | |
| 3. | DI AN | INED ANALYSES | 40 |
| ა. | | | |
| | 3.1.<br>3.2. | Interim Analyses | |
| | 3.2. | Final Analyses | 13 |
| 4. | ANAL | YSIS POPULATIONS | 14 |
| | 4.1. | Protocol Deviations | 15 |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | 16 |
| | | 5.1.1. Study Treatment & Sub-group Display Descriptors for | |
| | | Study Population Displays | 16 |
| | | 5.1.2. Study Treatment & Sub-group Display Descriptors for | |
| | | Efficacy Displays | 16 |
| | | 5.1.3. Study Treatment & Sub-group Display Descriptors for | |
| | | Safety Displays - Adverse Events (AEs) and Laboratory | 47 |
| | | Assessments | |
| | 5.2. | 5.1.4. Study Treatment descriptors used for Figures | |
| | 5.2. | 5.2.1. Baseline definition in Period 1 and Period 1+2 | |
| | | 5.2.2. Baseline definition in Period 1 and Period 1+2 | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | J. <del>4</del> . | 5.4.1. Covariates and Other Strata | 21 |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | 20 |
| | 0.0. | Conventions | 26 |
| 6. | | DY POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | 27 |
| 7. | EFFIC | CACY ANALYSES | 28 |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Primary Estimand Strategy | |
| | | 7.1.2. Supplementary Analyses | |
| | | 7.1.3. Statistical Analyses / Methods | |
| | 7.2. | Secondary Efficacy Analyses | |
| | - | 7.2.1. Estimand strategy | |
| | | 7.2.2. Supplementary Analysis | |

| | <b>T</b> | 7.2.3. Statistical Analyses / Methods | 35 |
|---|---|---|---|
| CC | | | |
| 0 | 0455 | TV ANALYOFO | 40 |
| 8. | 8.1. | TY ANALYSES | |
| | 8.1. | Adverse Events Analyses | |
| | 8.2. | 8.1.1. Adverse Events of Special Interest Analyses | |
| | 8.3. | Other Safety Analyses | |
| | 0.5. | 8.3.1. Immunogenicity Analyses | |
| CCI | | 0.0.1. Immunogenicity Analyses | |
| CCI | | | |
| 13. | REFE | RENCES | 50 |
| 14. | APPE | NDICES | 51 |
| | 14.1. | Appendix 1: Protocol Deviation Management and Definitions for Per | |
| | | Protocol Population | |
| | | 14.1.1. Exclusions from Per Protocol Population | 51 |
| | 14.2. | Appendix 2: Schedule of Activities | |
| | | 14.2.1. Protocol Defined Schedule of Events | |
| | 14.3. | Appendix 3: Assessment Windows | |
| | | 14.3.1. Definitions of Assessment Windows for Analyses | 55 |
| | 14.4. | Appendix 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | |
| | | 14.4.1. Study Phases | |
| | | 14.4.2. Treatment Emergent Flag for Adverse Events | |
| | 14.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | | 14.5.1. Reporting Process | |
| | | 14.5.2. Reporting Standards | 58 |

# CONFIDENTIAL

| 2 | <b>೧</b> 1 | 7 | a | • |
|---|------------|---|---|---|

| | 14.5.4. | Reporting Standards for Log-transformed Parameters | 59 |
|---|---|---|---|
| 14.6. | | x 6: Derived and Transformed Data | |
| | 14.6.1. | General | 60 |
| | 14.6.2. | Study Population | |
| | 14.6.3. | Efficacy | |
| | 14.6.4. | Safety | |
| 14.7. | Appendix | x 7: Reporting Standards for Missing Data | 83 |
| | 14.7.1. | Premature Withdrawals | |
| | 14.7.2. | | |
| 14.8. | Appendix | x 8: Values of Potential Clinical Importance | |
| | 14.8.1. | Laboratory Values Gradings | 85 |
| | 14.8.2. | Laboratory Values of Potential Clinical Importance | |
| | 14.8.3. | | |
| | 14.8.4. | Vital Signs Values of Potential Clinical Importance | |
| 14.9. | | x 9: List of Preferred Terms | |
| | 14.9.1. | Herpes Zoster | |
| | 14.9.2. | Mycobacterium Tuberculosis | |
| 14.10. | | x 10: Missing Data Imputation Strategies | |
| | 14.10.1. | Primary Estimand Strategy | 90 |
| | 14.10.2. | Supplemental Estimand 1 Strategy | 90 |
| | 14.10.3. | Supplemental Estimand 2 Strategy | 91 |
| | | Intermittent Missing Data Multiple Imputation | |
| 14.11. | | x 11: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | 14.11.2. | Trademarks | 94 |
| 14.12. | Appendix | x 12: List of Data Displays | 95 |
| | 14.12.1. | Data Display Numbering | 95 |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| 14.13. | Appendix | x 13: Example Mock Shells for Data Displays | 183 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2018N385740_00 | 06-Mar-2019 | Original |
| 2018N385740_01 | 22-May-2019 Correction of contraceptive requirements for Women of Child Bearing Potential (WOCBP) and additional clarifications. | |
| 2018N385740_02 | 21-Jan-2020 | <ul> <li>(1) To detail revised risks, entry and stopping criteria following the update to comparator drug (tofacitinib) label;</li> <li>(2) To introduce new medical device safety reporting wording, required in advance of roll out of pre-filled syringes to this study. (3) Other minor corrections and clarifications.</li> </ul> |

# 1.1. RAP Amendments

Revision chronology:

| RAP Section Amendment Details | |
|---|---|
| Statistical Analysis Plan F | Statistical Analysis Plan Final Reporting and Analysis Plan_201790_V1 [14-Feb-2022] |
| Statistical Analysis Plan F | inal Reporting and Analysis Plan Amendment_201790_V1 |
| Section 5.5 | Ordering of multiple testing procedure was amended. |
| Section 7.2 | Separate section for radiographic endpoints was removed and these endpoints were added into Section 7.2. |
| Section 14.6.2 | Correction to the Corticosteroid Scaling Factors. |
| Section 14.6.4 | Update to the derivation of Broad MACE and clarifications on CV events |
| | Addition of 3 tables and 3 figures for statistical analysis on radiographic endpoints |
| Section 14.12 | Addition of 4 tables and 1 figure for the COVID assessment on the Chinese population |
| | "Asia AAC" deliverable introduced to separate Asia-specific outputs from the AAC deliverable |
| General | Minor typos corrected |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol amendment 2 (Dated: 21/Jan/2020) are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| In order to preserve type 1 error, each of the primary and key secondary endpoints (ACR20, CDAI-LDA and HAQ- DI) will be assessed sequentially using a step-down approach. | <ul> <li>The step-down approach detailed in the protocol is extended to make use of a graphical multiple testing procedure and the principle of alphapropagation.</li> <li>The following are added into the multiplicity control: <ul> <li>Superiority versus placebo:</li></ul></li></ul> | To ensure that comparisons of interest for potential claims are controlled for multiplicity per the regulatory agency's feedback. |
| Major Secondary Efficacy Endpoints are CDAI-LDA and HAQ-DI. | CDAI total score, FACIT Fatigue and Pain VAS are added as Major Secondary Efficacy Endpoints. | Major Secondary Efficacy Endpoints aligned with the updated hierarchy (described on row above) |
| ACR20 and CDAI-LDA will be analysed using GEE | ACR20 and CDAI-LDA will<br>be analysed using Logistic<br>Regression | Missing data handling strategies will implement multiple imputation to generate full analysis datasets. GEE analysis provides no additional benefit over logistic regression when working with full datasets. |
| HAQ-DI will be analysed using MMRM | HAQ-DI will be analysed using ANCOVA | Missing data handling strategies will implement multiple imputation to generate full analysis datasets. MMRM analysis provides no additional benefit over ANCOVA when working with full datasets. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Intercurrent Event specified as discontinuation of study intervention | Additional intercurrent events specified: Discontinuation of study intervention for any reason Use of prohibited medication Change in stable dose of background medication | Following regulatory feedback |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the efficacy of GSK3196165 at doses of 90 mg and 150 mg weekly versus placebo for the treatment of participants with moderately to severely active RA who are on a stable background of csDMARDs and who have had an inadequate response to csDMARDs or bDMARDs. Secondary Objectives | Proportion of participants achieving ACR20 at Week 12 Secondary Endpoints |
| To compare: | Major Secondary Efficacy Endpoints |
| Efficacy of GSK3196165 at doses of 90 mg and 150 mg weekly versus tofacitinib for the treatment of participants with moderately to severely active RA who are on a stable background of csDMARDs and who have had an inadequate response to csDMARDs or bDMARDs. | <ul> <li>Week 12 versus placebo:</li> <li>Proportion of participants achieving CDAI total score ≤10 (CDAI LDA).</li> <li>Change from baseline in HAQ-DI.</li> <li>Change from baseline in FACIT-Fatigue</li> <li>Non-inferiority and superiority versus tofacitinib at Week 24:</li> <li>Proportion of participants achieving ACR20.</li> <li>Superiority versus tofacitinib at Week 24:</li> <li>Change from baseline in CDAI total Score</li> <li>Change from baseline in Pain VAS</li> <li>Proportion of participants achieving ACR20</li> <li>Change from baseline in FACIT Fatigue</li> <li>Other Secondary Efficacy Endpoints</li> <li>Week 12 (vs. placebo and vs. tofacitinib), Week 24 and Week 52 (vs. tofacitinib):</li> <li>Proportion of participant achieving:</li> <li>CDAI total score ≤10 (CDAI LDA).</li> <li>CDAI total score ≤2.8 (CDAI Remission).</li> <li>ACR20/50/70.</li> <li>DAS28-CRP &lt;3.2 and DAS28(ESR) &lt;3.2 (DAS28 LDA).</li> <li>DAS28-CRP &lt;2.6 and DAS28(ESR) &lt;2.6 (DAS28 Remission).</li> <li>A change from baseline in van der Heijde mTSS score of ≤0.5.</li> <li>Change from baseline in:</li> <li>CDAI total score.</li> <li>DAS28-CRP/DAS28-ESR.</li> <li>van der Heijde mTSS.</li> </ul> |
| Effect of GSK3196165 on Patient | Change from baseline at Week 12 (vs. placebo and vs. |
| Reported Outcomes (PROs) versus | tofacitinib), Week 24 and Week 52 (vs. tofacitinib) in: |

| Objectives | Endpoints |
|---|---|
| placebo and the active comparator tofacitinib | <ul> <li>HAQ-DI.</li> <li>Arthritis pain VAS.</li> <li>SF-36 physical and mental component scores, and domain scores.</li> <li>FACIT-Fatigue.</li> </ul> |
| Safety and tolerability of<br>GSK3196165 versus placebo and<br>the active comparator tofacitinib | <ul> <li>Incidence of AEs, SAEs and AESIs.</li> <li>Change from baseline in key laboratory parameters.</li> <li>Proportion of participants with NCI CTCAE ≥ Grade 3 haematological/clinical chemistry abnormalities.</li> </ul> |
| To determine the immunogenic potential of GSK3196165 | Safety Biomarker Endpoints |



# 2.3. Study Design



#### **Overview of Study Design and Key Features**

- key Asian country subgroups is not reached, then recruitment in these countries may continue.
- Participants who have already been enrolled from Asian country subgroups at the time of reaching the 1500 target will be included in the primary analysis. Doubleblinding will be maintained for any subjects continuing in the study at the time of the primary analysis. The primary analysis will be the basis of all inferences.
- If enrolment continues beyond the planned target of 1500 randomised participants, secondary analyses will be conducted upon completion of enrolment/follow-up for the entire study population, based on all randomised subjects.

# 2.4. Statistical Hypotheses

The primary objective of the study is to determine whether GSK3196165 is superior to placebo in the treatment of participants with moderately to severely active RA despite csDMARD treatment (i.e. csDMARD-IR), as assessed by the proportion of participants achieving ACR20 response at Week 12.

The study will test the null hypothesis that there is no difference between the 150mg dose of GSK3196165 and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 150mg dose of GSK3196165 differs from placebo in the proportion of participants achieving ACR20 response at Week 12.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

The primary analysis will be conducted when the planned target of 1500 randomised participants has been reached. No interim analysis with respect to this population is planned. However, if at the time of reaching approximately 1500 randomised participants a sufficient number of participants that are required for the key Asian country subgroups is not reached, then recruitment in these countries may continue. Participants who have already been enrolled from Asian country subgroups at the time of reaching the 1500 target will be included in the primary analysis. Double-blinding will be maintained for any subjects continuing in the study at the time of the primary analysis. The primary analysis will be the basis of all inferences. If enrolment continues beyond the planned target of 1500 randomised participants, secondary analyses will be conducted upon completion of enrolment/follow-up for the entire study population, based on all randomised subjects.

An Independent Data Monitoring Committee (IDMC) will be utilised in this study to ensure ongoing objective medical and/or statistical review of safety data in order to protect the welfare of participants in the study and the scientific validity of the study. Full details of the data to be reviewed, the frequency of review and members of the committee are included in the IDMC Charter [Version 1.0 09 May 2019]. Full details of the analyses are included in a separate IDMC RAP [ Version 1.0 30 Apr 2020]. Monthly Safety Review Team (SRT) reviews will be performed using blinded SDTM datasets and will be reviewed using Spotfire software.

# 3.2. Final Analyses

The final planned analyses on the primary analysis cohort (i.e. the first approximately 1500 participants) will be performed after the completion of the following sequential steps:

- 1. All participants to be included in the primary analyses have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Prior to unblinding, all protocol deviations that will result in an exclusion from the per-protocol population have been assigned in the analysis dataset.
- 5. Randomization codes have been distributed according to Cenduit Interactive Response Technology (C.I.R.T) system procedures.

If required, the final planned analyses on the full analysis set will be performed after the completion of the following sequential steps:

1. All participants from the key Asian country cohort have completed the study as defined in the protocol.

- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Prior to unblinding, all protocol deviations that will result in an exclusion from the per-protocol population have been assigned in the analysis dataset.
- 5. Randomization codes have been distributed according to Cenduit Interactive Response Technology (C.I.R.T) system procedures.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Study Population |
| Randomized | <ul> <li>All participants who were randomly assigned to treatment in the study.</li> <li>This population will be based on the treatment the participant was randomized to.</li> <li>Any participants who receives a treatment randomization number will be considered to have been randomized.</li> </ul> | Study Population |
| Enrolled | <ul> <li>All participants who passed screening and entered the study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population |
| Safety | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> <li>Note: Participants who were not randomized but received at least one dose of study treatment should be listed.</li> </ul> | <ul><li>Safety</li><li>Biomarker</li></ul> |
| Safety –<br>Subjects who<br>Entered Period 2 | <ul> <li>All participants randomized to a placebo switch treatment arm (i.e. Placebo to GSK3196165 90mg, Placebo to GSK3196165 150mg or Placebo to Tofacitinib 5mg) who received at least one dose of study treatment in period 2.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | Safety |
| Intent-To-Treat<br>(ITT) | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject was randomized to.</li> <li>Any participants who receives a treatment randomization number will be considered to have been randomized.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Per-Protocol | All participants in the ITT population who comply with the protocol. | Efficacy |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| (PP) | <ul> <li>Protocol deviations that would exclude participants from the PP population are defined in Section 4.1 (Protocol Deviations) and Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).</li> <li>The PP set will not be analysed if this population comprises more than 85% of the ITT population.</li> </ul> | |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised by IQVIA CTMS category. GSK subcategories will be included in individual subject listings.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by IQVIA and overseen by the GSK study team throughout the conduct of the study in accordance with the latest version of the Protocol Deviation Management Plan maintained by IQVIA in their TMF system.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised in the protocol deviations dataset.
- Deviations leading to exclusion from the Per Protocol Population will be identified in the ADDV dataset.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

Additional protocol deviations may be identified during the study and will be documented in protocol deviation adjudication meeting minutes prior to database freeze.

All violations will be discussed and adjudicated as important or not important. Only protocol deviations that have the potential to impact the efficacy evaluation (and are important) will lead to exclusion from the per-protocol population.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

# 5.1.1. Study Treatment & Sub-group Display Descriptors for Study Population Displays

Unless otherwise specified, all study population outputs will display the pooled placebo arm as follows:

| | Treatment Group Descriptions | | |
|---|---|---|---|
| Cenduit Interactive Response | | Data Displays for Reporting | |
| Technology (CIRT) Code Description | | Description | Order in TLF |
| 1 | | | Order in TEI |
| 1 | GSK3196165 150mg | OTI 150mg QW | 3 |
| 2 | GSK3196165 90mg | OTI 90mg QW | 2 |
| 3 | Tofacitinib BID | TOFA 5mg BID | 4 |
| 4+5+6 | Placebo to GSK3196165 150mg | Pooled PBO | 1 |
| | + Placebo to GSK3196165 90mg | | |
| | + Placebo to Tofacitinib BID | | |

All study population outputs required to be displayed by randomised treatment arm will display all randomised treatment arms as follows:

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Cenduit Interactive Response | | Data Displays for Reporting | |
| Technology (CIRT) Code Description | | Description Order in TL | |
| 1 | GSK3196165 150mg | OTI 150mg QW | 5 |
| 2 | GSK3196165 90mg | OTI 90mg QW | 4 |
| 3 | Tofacitinib BID | TOFA 5mg BID | 6 |
| 4 | Placebo to GSK3196165 150mg | PBO to OTI 150mg QW | 2 |
| 5 | Placebo to GSK3196165 90mg | PBO to OTI 90mg QW | 1 |
| 6 | Placebo to Tofacitinib BID | PBO to TOFA 5mg BID | 3 |

# 5.1.2. Study Treatment & Sub-group Display Descriptors for Efficacy Displays

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Cenduit Interactive Response Data Displays for Reporting | | | |
| Code | Technology (CIRT) Description | Description | Order in TLF |
| 1 | GSK3196165 150mg | OTI 150mg QW | 3 |
| 2 | GSK3196165 90mg | OTI 90mg QW | 2 |
| 3 | Tofacitinib BID | TOFA 5mg BID | 4 |
| 4 | Placebo to GSK3196165 150mg | PBO to OTI 150mg QW | 6 |
| 5 | Placebo to GSK3196165 90mg | PBO to OTI 90mg QW | 5 |

| Treatment Group Descriptions | | | |
|---|---|---|---|
| 6 | Placebo to Tofacitinib BID | PBO to TOFA 5mg BID | 7 |
| 4+5+6 | Placebo to GSK3196165 150mg | Pooled PBO | 1 |
| | + Placebo to GSK3196165 90mg | | |
| | + Placebo to Tofacitinib BID | | |

For the purpose of analyses up to week 12. the placebo-sequence groups will be pooled into a single placebo arm.

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. Otilimab 90mg vs Pooled Placebo
- 2. Otilimab 150mg vs Pooled Placebo
- 3. Tofacitinib 5mg vs Pooled Placebo
- 4. Otilimab 90mg vs Tofacitinib 5mg
- 5. Otilimab 150mg vs Tofacitinib 5mg

# 5.1.3. Study Treatment & Sub-group Display Descriptors for Safety Displays - Adverse Events (AEs) and Laboratory Assessments

Each AE display will be produced for the time periods below (see Figure 1 for graphical representation):

- 1. Period 1 up to week 12, to be displayed for all participants.
  - Period 1 (up to week 12) is defined as time from randomisation and first dose of treatment up to dosing of Period 2 treatment (Week 12) or date of study withdrawal or date of treatment withdrawal plus safety follow up, whichever is earlier. AEs that occur at week 12 visit i.e. AE start date is at week 12 visit will be assigned to Period.
  - The placebo-sequence groups up to week 12 will be pooled into a single placebo arm.
- 2. Period 2 post week 12, to be displayed for participants who were originally randomised to receive placebo and switched at week 12, only.
  - Period 2 is defined as time from first dose of treatment of period 2 (week 12) until date of study completion or date of study withdrawal or date of treatment withdrawal plus safety follow up, whichever is earlier.
- 3. Period 1+2 from week 0 to week 52, to be displayed for participants who were originally randomised to Otilimab 150mg, Otilimab 90mg or Tofacitinib 5mg, only.
  - Period 1+2 is defined as time from randomisation until date of study completion or date of study withdrawal or date of treatment withdrawal plus safety follow up, whichever is earlier.



Figure 1 Graphical Representation of Study Design with Periods and Treatment Arms within Each Period

For displays for Period 1 (up to week 12), the following treatment group descriptions will be used:

| | Treatment Group Descriptions | | |
|---|---|---|---|
| Cenduit Interactive Response | | Data Displays for Reporting | |
| | Technology (CIRT) | | |
| Code | Description | Description Order in T | |
| 1 | GSK3196165 150mg | OTI 150mg QW | 3 |
| 2 | GSK3196165 90mg | OTI 90mg QW | 2 |
| 3 | Tofacitinib BID | TOFA 5mg BID | 4 |
| 4+5+6 | Placebo to GSK3196165 150mg | Pooled PBO | 1 |
| | + Placebo to GSK3196165 90mg | | |
| | + Placebo to Tofacitinib BID | | |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. Otilimab 150mg vs Pooled Placebo
- 2. Otilimab 90mg vs Pooled Placebo
- 3. Tofacitinib 5mg vs Pooled Placebo
- 4. Otilimab 150mg vs Tofacitinib 5mg
- 5. Otilimab 90mg vs Tofacitinib 5mg
- 6. Otilimab 150mg vs Otilimab 90mg

For displays for Period 2 (post week 12), the following treatment group descriptions will be used:

| | Treatment Group Descriptions | | |
|---|---|---|---|
| C | Cenduit Interactive Response | Data Displays for Reporting | |
| Technology (CIRT) | | | |
| Code | Description | Description Order in T | |
| 4 | Placebo to GSK3196165 150mg | PBO to OTI 150mg QW | 2 |
| 5 | Placebo to GSK3196165 90mg | PBO to OTI 90mg QW | 1 |
| 6 | Placebo to Tofacitinib BID | PBO to TOFA 5mg BID | 3 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. Placebo to Otilimab 150mg vs Placebo to Tofacitinib 5mg
- 2. Placebo to Otilimab 90mg vs Placebo to Tofacitinib 5mg
- 3. Placebo to Otilimab 150mg vs Placebo to Otilimab 90mg

For displays for period 1+2 (Week 0 to Week 52), the following treatment group descriptions will be used:

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Ce | nduit Interactive Response<br>Technology (CIRT) | Data Displays for Reporting | |
| Code | Description | Description Order in TLF | |
| 1 | GSK3196165 150mg | OTI 150mg QW | 2 |
| 2 | GSK3196165 90mg | OTI 90mg QW | 1 |
| 3 | Tofacitinib BID | TOFA 5mg BID | 3 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. Otilimab 150mg vs Tofacitinib 5mg
- 2. Otilimab 90mg vs Tofacitinib 5mg
- 3. Otilimab 150mg vs Otilimab 90mg

# 5.1.4. Study Treatment descriptors used for Figures

Table 2 describes the format required for the reporting of figures.

Table 2 Treatment Descriptors, Colours, Line Style and Symbols to be used for Figures

| Treatment Description | Colour | SAS Colour | Marker | Line pattern |
|-----------------------|--------|------------|---------------|--------------|
| | | | Symbol | |
| Pooled PBO | Black | #333333 | X | 2 |
| PBO to OTI 90mg QW | Orange | #F36633 | SquareFilled | 2 |
| PBO to OTI 150mg QW | Green | #167716 | DiamondFilled | 2 |
| PBO to TOFA 5mg BID | Blue | #3131DD | CircleFilled | 2 |
| OTI 90mg QW | Orange | #F36633 | Square | 1 |
| OTI 150mg QW | Green | #167716 | Diamond | 1 |
| TOFA 5mg BID | Blue | #3131DD | Circle | 1 |

# 5.2. Baseline Definitions

# 5.2.1. Baseline definition in Period 1 and Period 1+2

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Assessments Considered as<br>Baseline | | Baseline Used in<br>Data Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Efficacy | | | |
| Tender Joint Count 28 | | X | Day 1 (Pre-Dose) |
| Tender Joint Count 68 | | X | Day 1 (Pre-Dose) |
| Swollen Joint Count 28 | | X | Day 1 (Pre-Dose) |
| Swollen Joint Count 66 | | X | Day 1 (Pre-Dose) |
| Pain VAS | | X | Day 1 (Pre-Dose) |
| Patient's Global Assessment of Arthritis (PtGA) | | Х | Day 1 (Pre-Dose) |
| Physician's Global Assessment of Arthritis (PhGA) | | Х | Day 1 (Pre-Dose) |
| CRP | | Х | Day 1 (Pre-Dose) |
| ESR | | Х | Day 1 (Pre-Dose) |
| HAQ-DI | | X | Day 1 (Pre-Dose) |
| DAS28-CRP Total Score | | Х | Day 1 (Pre-Dose) |
| DAS28-ESR Total Score | | Х | Day 1 (Pre-Dose) |
| Van der Heijde mTSS | Х | | Screening |
| SF-36 | | X | Day 1 (Pre-Dose) |
| FACIT-Fatigue | | Х | Day 1 (Pre-Dose) |

| Parameter | Study Assessments Considered as<br>Baseline | | Baseline Used in<br>Data Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Safety | | | |
| Vital Signs | X | X | Day 1 (Pre-Dose) [1] |
| ECG (12-lead) | X | Х | Day 1 (Pre-Dose) [1] |
| Laboratory | Х | Х | Day 1 (Pre-Dose) [1] |
| Pulmonary assessments | X | X | Day 1 (Pre-Dose) [1] |
| Immunogenicity | | X | Day 1 (Pre-Dose) |



Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.2.2. Baseline definition in Period 2

For all safety assessments the baseline value will be the latest pre-dose assessment before the first dose in period 2 with a non-missing value, including those from unscheduled visits.

#### 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site, country, and the regions.

| Region | Countries |
|---|---|
| US | United States |
| European Continent and Australia | Australia, Bulgaria, Estonia, France, Germany, Hungary, Poland, Russia, Spain, United Kingdom |
| Latin America | Argentina, Brazil, Colombia, Mexico |
| Asia | China, Japan, South Korea, Thailand |

# 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|------------|--------------------------------------------------------|
| Strata | Randomisation Stratification Factors: |
| | Previously failed medication: |
| | o csDMARD only |
| | o 1 bDMARD |
| | o >1 bDMARD |
| Covariates | Relevant baseline score, previously failed medication. |

# **5.4.2.** Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the study.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories | Overall Group |
|---|---|---|
| Prior Failed DMARD | csDMARD only, 1 bDMARD, >1 bDMARD | Disease<br>Characteristic |
| Region | US, European Continent and Australia, Latin America, Asia | Demographic |
| Specific Region | Europe, other | Demographic |
| Specific Region | USA, other | Demographic |
| Specific Region | Japan (Japan Region and Japanese Heritage Race), other | Demographic |
| Specific Region | China, other | Demographic |
| Age | <50 years, 50 to 64 years, ≥65 years | Demographic |
| Ethnicity | Hispanic or Latino, Not Hispanic or Latino | Demographic |
| Race | Black or African American/African Heritage,<br>Asian, White, Other (American Indian or Alaskan<br>Native, Native Hawaiian or Other Pacific<br>Islander, Multiple) | Demographic |
| Gender | Male, Female | Demographic |
| Baseline Body Weight | <60kg, 60-100kg, >100kg | Demographic |
| Baseline both RF Negative and Anti-CCP Negative | Both Negative, At Least One Positive | Disease<br>Characteristic |
| Baseline DAS28-CRP | <5.1, ≥5.1 | Disease<br>Characteristic |
| Baseline CDAI | <22, ≥22 | Disease<br>Characteristic |
| Duration of RA | ≤5 years, >5 to ≤10 years, >10 years | Disease<br>Characteristic |
| BMI | <25, ≥25 and <30, ≥30 | Demographic |

# 5.5. Multiple Comparisons and Multiplicity

The graphical multiple testing procedure described in (Bretz, 2009) will be used to control the type I error for the primary and key secondary endpoints.

Each hypothesis will be assessed sequentially using a step-down approach where testing of the second hypothesis will commence only if all null hypotheses of the prior steps are rejected. Additionally, as there are two doses of GSK3196165 within each test, this will also be incorporated into the step-down procedure.

A graphical presentation of the multiplicity control is provided in Figure 2.

If any of the hypotheses in the list are not rejected (i.e. the testing sequence fails at this step), the subsequent test(s) will still be performed but the results will be uncontrolled for multiplicity.

The proposed testing sequence of primary and key secondary hypotheses is:

- 1. ACR20 GSK3196195 vs. Placebo for Superiority at Week 12
- 2. CDAI-LDA GSK3196195 vs. Placebo for Superiority at Week 12
- 3. HAQ-DI GSK3196195 vs. Placebo for Superiority at Week 12
- 4. ACR20 GSK3196195 vs. Tofacitinib for Non-Inferiority at Week 24
- 5. FACIT-Fatigue GSK3196165 vs. Placebo for Superiority at Week 12
- 6. CDAI Total Score GSK3196195 vs. Tofacitinib for Superiority at Week 24
- 7. Pain VAS GSK3196195 vs. Tofacitinib for Superiority at Week 24
- 8. ACR20 GSK3196195 vs. Tofacitinib for Superiority at Week 24
- 9. FACIT-Fatigue GSK3196165 vs. Tofacitinib for Superiority at Week 24

The following steps will be followed to test the aforementioned hypotheses:

| Step | Test | Pre-requisite(s) | P-value (2-<br>sided) |
|---|---|---|---|
| 1 | ACR20 at week 12 for<br>GSK3196165 150mg vs.<br>placebo | None | 0.05 |
| 2a | CDAI-LDA at week 12 for<br>GSK3196165 150mg vs.<br>placebo | Step 1 passed | 0.025 |
| 2b | HAQ-DI at week 12 for<br>GSK3196165 150mg vs.<br>placebo | Step 2a passed | 0.025 |
| 3a | ACR20 at week 12 for<br>GSK3196165 90mg vs. placebo | Step 1 passed | 0.025 |
| 3b | CDAI-LDA at week 12 for<br>GSK3196165 90mg vs. placebo | Step 3a passed | 0.025 |
| 3c | HAD-DI at week 12 for GSK3196165 90mg vs. placebo | Step 3b passed | 0.025 |

| Step | Test | Pre-requisite(s) | P-value (2- |
|---|---|---|---|
| | | | sided) |
| 4 | ACR20 at week 24 for non- | Both step 2b and 3c passed | 0.05 |
| | inferiority of GSK3196165<br>150mg vs. tofacitinib | Step 2b passed and step 3c failed or not reached | 0.025 |
| | | Step 3c passed and step 2b failed or not reached | 0.025 |
| 5 | FACIT-Fatigue at week 12 for superiority of GSK3196165 | Step 4 tested at p=0.05 and passed | 0.05 |
| | 150mg vs. placebo | Step 4 tested at p=0.025 and passed | 0.025 |
| 6 | ACR20 at week 24 for non- | Step 5 tested at p=0.05 and passed | 0.05 |
| | inferiority of GSK3196165<br>90mg vs. tofacitinib | Step 5 tested at p=0.025 and passed | 0.025 |
| 7 | FACIT-Fatigue at week 12 for | Step 6 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>90mg vs. placebo | Step 6 tested at p=0.025 and passed | 0.025 |
| 8 | CDAI total score at week 24 for | Step 7 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>150mg vs. tofacitinib | Step 7 tested at p=0.025 and passed | 0.025 |
| 9 | Pain VAS at week 24 for superiority of GSK3196165 | Step 8 tested at p=0.05 and passed | 0.05 |
| | 150mg vs. tofacitinib | Step 8 tested at p=0.025 and passed | 0.025 |
| 10 | ACR20 at week 24 for | Step 9 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>150mg vs. tofacitinib | Step 9 tested at p=0.025 and passed | 0.025 |
| 11 | CDAI total score at week 24 for | Step 10 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>90mg vs. tofacitinib | Step 10 tested at p=0.025 and passed | 0.025 |
| 12 | Pain VAS at week 24 for | Step 11 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>90mg vs. tofacitinib | Step 11 tested at p=0.025 and passed | 0.025 |
| 13 | ACR20 at week 24 for | Step 12 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>90mg vs. tofacitinib | Step 12 tested at p=0.025 and passed | 0.025 |
| 14 | FACIT-Fatigue at week 24 for | Step 13 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>150mg vs. tofacitinib | Step 13 tested at p=0.025 and passed | 0.025 |
| 15 | FACIT-Fatigue at week 24 for | Step 14 tested at p=0.05 and passed | 0.05 |
| | superiority of GSK3196165<br>90mg vs. tofacitinib | Step 14 tested at p=0.025 and passed | 0.025 |

Analyses of other efficacy endpoints will not be subject to any multiplicity adjustment.



Figure 2 Graphical of the Multiple Testing Procedure

Note: The number in the circles refer to the initial weighting of alpha. The number along the arrows refer to the weighting of alpha which is passed along to the next test.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 14.3 | Appendix 3: Assessment Windows |
| Section 14.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| Section 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 14.5 | Appendix 6: Derived and Transformed Data |
| Section 14.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 14.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 14.9 | Appendix 9: List of Preferred Terms |
| Section 14.10 | Appendix 10: Missing Data Imputation Strategies. |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Screened", "Randomised", "Enrolled" or "ITT" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

All concomitant medications summaries will use the "while on treatment" approach, i.e. any concomitant medications which are taken post discontinuation of study intervention plus safety follow-up (+56 days), will be excluded.

Additional study population outputs relating to the COVID-19 pandemic will be based on GSK Core Data Standards, including:

- Baseline characteristics by pre and post COVID-19 pandemic measures
- Participant status and disposition by relationship to COVID-19 pandemic
- Treatment status and reasons for discontinuation of study treatment by relationship to COVID-19 pandemic
- Participants by country and site by implementation of pandemic measures
- Protocol deviations by relationship to COVID-19 pandemic
- COVID-19 Visits and Assessments Impacts
- Recruitment relative to COVID-19 pandemic measures

Details of the planned displays are presented in Appendix 12: List of Data Displays.

#### 7. EFFICACY ANALYSES

As discussed in the addendum ICH E9 (R1) [ICH, 2019] the specification of treatment effects to be estimated (the estimand) should include:

- The population of interest.
- The treatment condition of interest.
- The outcome variable of interest.
- The summary measure (which may be a model-based estimate or comparison).
- The identification and strategy for handling potential intercurrent events.

The following sections provide clarity on each of these components for the efficacy treatment effects to be estimated in this study and details on how missing outcomes will be handled.

# 7.1. Primary Efficacy Analyses

# 7.1.1. Primary Estimand Strategy

The primary estimand for this study is derived directly from the primary objective of the study to determine whether GSK3196165 150mg is superior to placebo in the treatment of participants with moderately to severely active RA despite csDMARD or bDMARD treatment (i.e. csDMARD-IR or bDMARD-IR). This will be assessed by the odds ratio of ACR20 response at Week 12 for GSK3196165 versus placebo, regardless of: IP discontinuation for any reason, prohibited medication use or change in stable dose of background therapy. Each component of this estimand is described below.

# **7.1.1.1.** Population

Participants with moderately to severely active RA despite csDMARD or bDMARD treatment, which is targeted using the inclusion and exclusion criteria.

#### **7.1.1.2.** Treatment

Those who receive at least one dose of GSK3196165 150mg, compared to those who receive at least one dose of placebo in addition to any other medication taken during the study.

#### 7.1.1.3. Outcome Variable

ACR20 response at week 12.

#### 7.1.1.4. Summary Measure

The odds ratio comparing GSK3196165 150mg arm with placebo. This measure will be derived from model-based adjusted estimates.

#### 7.1.1.5. Strategy for Intercurrent (Post-Randomization) Events

The intercurrent (post-randomisation) event (IE) anticipated to impact on the interpretation of the treatment effect for the primary objective are:

- 1. Discontinuation of study intervention for any reason
- 2. Use of prohibited medication
- 3. Change in stable dose of background medication

The handling strategy for all of these IEs will be based on a treatment policy approach; specifically, the effects estimated will be based on initial randomized treatment arm regardless of whether the participant had observed the IE. Data will continue to be collected after the occurrence of the IE, until the participant either completes the study or withdraws from the study before completion.

#### 7.1.1.6. Handling of Missing Data

Intermittent missing data (i.e. data between two non-missing assessments) for the ACR20 will be imputed under a missing at random (MAR) assumption.

If a participant experiences any of the IEs but efficacy data continues to be collected, their data will be analysed per their original randomised intervention.

Study withdrawal before the completion of the study will create missing outcome data. This may occur concurrently or after the IE. Missing data for the ACR20 response resulting from study withdrawal will be imputed using three possible MI models depending on the availability of off-treatment data (i.e. data that has been collected post discontinuation of study intervention), using principles introduced by Roger, 2019 (computational details are included in Section 14.10):

#### 1. MI using off-treatment data within randomised treatment arm:

If there is sufficient off-treatment data within a randomised treatment arm (i.e. at least 3 participants per arm per visit), then missing data will be imputed conditional on the participant's observed outcomes, using off-treatment data within randomised treatment arm. The use of this MI model assumes that missing outcomes resulting from participants withdrawing from the study would behave in a similar way to other participants who discontinued study intervention, were randomised to the same treatment arm, and continued providing data post-discontinuation of study intervention.

#### 2. MI using off-treatment data across all treatment arms:

If there is insufficient off-treatment data within a randomised treatment arm (i.e. failure of the imputation model in option 1) but there is sufficient off-treatment data across all treatment arms combined (i.e. at least 3 participants per visit), then missing data will be imputed conditional on the participant's observed outcomes, using off-treatment data across all treatment arms. The use of this MI model assumes that missing outcomes resulting from participants withdrawing from the study would behave in a similar way to other participants who discontinued study

intervention and continued providing data post-discontinuation of study intervention regardless of randomised treatment arm.

### 3. MI under MAR assumption:

If there is insufficient off-treatment data (i.e. neither option 1 nor 2 is feasible) then all missing data will be imputed under a MAR assumption. This MI model uses all available data collected on- and off-treatment within randomised treatment arm, and assumes missing outcomes resulting from participants withdrawing from the study would behave in a similar way to participants who were randomised to the same treatment arm and had data collected in the study, with no adjustment for values before or after intercurrent events.

Note: Week 1 data will not be included in any imputation models due to the unavailability of off-treatment data at this visit by design of the study.

#### 7.1.1.7. Sensitivity Analysis for the Handling of Missing Data

An additional tipping point analysis will be performed as sensitivity if the endpoint is statistically significant and it is plausible that the imputation strategy for missing data could alter the conclusions of the analysis. This will be performed at an ACR20 responder level assuming all possible ACR20 response rates from 0 to 100% amongst those with missing ACR20 response in GSK3196165 arm and pooled placebo arm, separately. Full details of this analysis will be included in a separate analysis plan and results included in a separate report.

#### 7.1.2. Supplementary Analyses

Two additional estimands for the primary objective will be considered and are described in this section. Computational details on both of these strategies are included in Section 14.10.

#### 7.1.2.1. Supplemental Estimand 1

As an additional estimand for the primary objective, a composite strategy will be considered for the handling of the IE of discontinuation of study intervention for any reason; specifically, a composite response definition will be used. A participant will be considered to be a non-responder if they do not meet the ACR20 response criterion or they discontinue study intervention for any reason. All other IEs will be handled using the same strategy as for the Primary Estimand Strategy (i.e. treatment policy).

# 7.1.2.2. Supplemental Estimand 2

As a second additional estimand for the primary objective, a hypothetical strategy will be considered for the handling of the IE of discontinuation of study intervention for any reason; specifically, the effects estimated will be under the hypothetical scenario where the IE did not occur.

Any efficacy data collected after the occurrence of this IE will be excluded from the analysis. All data for the treatment response after the occurrence of the IE will be

imputed conditional on the participant's observed outcomes, using on- and off-treatment data within randomised treatment arm. The use of this MI model assumes that missing outcomes would behave in a similar way to other participants who were randomised to the same treatment arm and had data collected in the study, with no adjustment for values before or after intercurrent events.

All other IEs will be handled using the same strategies as for the Primary Estimand Strategy (i.e. treatment policy).

# 7.1.2.3. Per-protocol Analysis

As a supportive analysis, the primary analyses may be repeated using the "Per-protocol" population (see Section 14.1 for the definition).

# 7.1.3. Statistical Analyses / Methods

The efficacy analyses will be based in the "Intent-to-Treat" population, unless otherwise specified.

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1.3 will be summarised using descriptive statistics and graphically presented (where appropriate).

# 7.1.3.1. Statistical Methodology Specification

### **Endpoint / Variables**

Proportion of participants with ACR20 response at week 12.

#### **Model Specification**

- Each estimate will be generated for each imputed dataset produced by the multiple imputation (MI) procedure described in Section 7.1.1.6, and the corresponding results will be combined using Rubin's rules.
- The proportion of participants with ACR20 response will be statistically analysed using a Logistic Regression model, comparing each randomised treatment arm with control group.
- The Logistic Regression model will be fitted including fixed effects for treatment arm (GSK3196165 150mg, GSK3196165 90mg, tofacitinib 5mg, pooled placebo), baseline swollen joint count 66, baseline tender joint count 68 and previously failed medication (csDMARD only, 1 bDMARD, >1 bDMARD).

#### **Model Checking & Diagnostics**

If the logistic model fails to converge (e.g. due to a small number of responders), the primary
endpoint will be analysed using an exact logistic regression. In case of response rates of 0%
or 100% in any of the treatment groups, confidence intervals for risk difference and p-values
from the t-test for the risk difference comparing to 0 will be provided.

#### **Model Results Presentation**

- Results will be summarised using proportions of subjects (after MI) achieving a response.
- Differences in the proportions of subjects (after MI) achieving response between each randomised treatment arm and pooled placebo will be summarised. 95% CI for the differences will be constructed using their asymptotic standard errors (asymptotic Wald confidence limits) without continuity correction.
- Estimates of the Odds Ratio (OR), corresponding 95% confidence intervals and p-values will be constructed using the least squared (LS) means estimates from the logistic regression model.
- Plots of the proportion of subjects (after MI) achieving a response and their corresponding asymptotic standard errors will be generated for each treatment group by time.

### **Subgroup Analyses**

See Section 5.4 for details on subgroup analyses.

#### **Sensitivity and Supportive Analyses**

- Sensitivity Analysis on the missing data imputation methods may be performed as described in Section 7.1.1.7.
- Supportive Analysis will be performed as described in Section 7.1.2.

# 7.2. Secondary Efficacy Analyses

# 7.2.1. Estimand strategy

The secondary efficacy analysis will use the same estimand as the primary efficacy analysis (see Section 7.1.1 for details).

#### **7.2.1.1.** Population

The population of interest for the secondary efficacy analysis is the same as is stated for the primary efficacy analysis (see Section 7.1.1.1).

#### **7.2.1.2.** Treatment

The treatment of interest for the secondary efficacy analysis is the same as is stated for the primary efficacy analysis (see Section 7.1.1.2).

#### 7.2.1.3. Outcome Variables

The key secondary outcomes of interest are:

- ACR20 response at week 12 (superiority of GSK3196165 90mg over placebo comparison) and at week 24 (non-inferiority and superiority over tofacitinib comparisons).
- CDAI-LDA (CDAI Total Score≤10) at week 12 (superiority over placebo comparisons).
- HAQ-DI at week 12 (superiority over placebo comparisons).
- CDAI Total Score at week 24 (superiority over tofacitinib comparisons).
- FACIT-Fatigue at week 12 (superiority over placebo comparison) and at week 24 (superiority over tofacitinib comparison).
- Pain VAS at week 24 (superiority over tofacitinib comparison).

#### Other Secondary:

- ACR20/50/70 response at each assessment visit.
- CDAI Remission (CDAI Total Score \( \leq 2.8 \)) at each assessment visit.
- DAS28-CRP LDA (DAS28-CRP\le 3.2) at each assessment visit.
- DAS28-ESR LDA (DAS28-ESR≤3.2) at each assessment visit.
- DAS28-CRP Remission (DAS28-CRP<2.6) at each assessment visit.
- DAS28-ESR Remission (DAS28-ESR<2.6) at each assessment visit.
- Good/moderate EULAR response at each assessment visit.
- Change from baseline in Van der Heijde mTSS \( \leq 0/0.5 \) at each assessment visit.
- ACR/EULAR Remission at each assessment visit.
- TJC28/68 and SJC28/66 at each assessment visit.
- CRP (mg/L) at each assessment visit.
- PtGA/PhGA at each assessment visit.
- DAS28-(CRP/ESR) at each assessment visit.
- Arthritis pain VAS at each assessment visit.
- SF-36 physical and mental component scores, and individual domain scores at each assessment visit.
- FACIT-Fatigue score at each assessment visit.
- Van der Heijde mTSS at each assessment visit.

#### 7.2.1.4. Summary Measure

The key secondary summary measures are:

- The odds ratio comparing GSK3196165 90mg arm with placebo in the proportion of participants achieving ACR20 at week 12.
- The odds ratio comparing GSK3196165 arms with placebo in the proportion of participants achieving CDAI-LDA at week 12.
- The difference between GSK3196165 arms and placebo in the change from baseline in HAQ-DI at week 12.
- The difference between GSK3196165 arms and tofacitinib in the change from baseline in CDAI Total Score at week 24.
- The difference between GSK3196165 arms and placebo in the change from baseline in FACIT-Fatigue Score at week 12.
- The difference between GSK3196165 arms and to facitinib in the proportion of participants achieving ACR20 at week 24.
- The difference between GSK3196165 arms and tofacitinib in the change from baseline in Arthritis Pain VAS at week 24.
- The odds ratio comparing GSK3196165 arms with tofacitinib in the proportion of participants achieving ACR20 at week 24.
- The difference between GSK3196165 arms and tofacitinib in the change from baseline in FACIT-Fatigue Score at week 24.

For all secondary endpoints (including the key secondary endpoints), the following summary measures are:

- Odds ratio and/or difference from placebo at all assessment visits up to week 12.
- Odds ratio and/or difference from tofacitinib at all assessment visits.

All summary measures will be derived from model-based adjusted estimates for each treatment arm.

#### 7.2.1.5. Strategy for Intercurrent (Post-Randomization) Events

The same strategy as the primary efficacy analysis will be implemented for all secondary efficacy analyses (See Section 7.1.1.5 for full details)

#### 7.2.1.6. Handling of Missing Data

The same missing data handling strategy as the primary efficacy analysis will be implemented for all secondary efficacy analyses (See Section 7.1.1.6 for full details)

#### 7.2.1.7. Sensitivity Analysis for the Handling of Missing Data

A tipping point analysis will be performed as sensitivity of the key secondary efficacy analyses if the endpoints are statistically significant and it is plausible that the imputation strategy for missing data could alter the conclusions of the analysis. For binary endpoints, the same tipping point strategy as for the primary endpoint will be implemented (see Section 7.1.1.7 for full details). For continuous endpoints, this will be performed by

applying a shift parameter to the mean for the participants with missing outcomes in the GSK3196165 arms and the control arm, separately. Full details of this analysis will be included in a separate analysis plan and results included in a separate report.

### 7.2.2. Supplementary Analysis

The same supplemental strategies as the primary efficacy analysis will be implemented for the key secondary efficacy endpoint analyses as follows:

- Supplemental estimand 1 will be applied to ACR20 and CDAI-LDA (see Section 7.1.2.1 for details).
- Supplemental estimand 2 will be applied to ACR20, CDAI Total score and Pain VAS (see Section 7.1.2.2 for details).

# 7.2.3. Statistical Analyses / Methods

The secondary efficacy analyses will be based in the "Intent-to-Treat" population, unless otherwise specified.

Details of the planned displays are provided in Appendix 12: List of Data Displays, and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1.3 will be summarised using descriptive statistics and graphically presented (where appropriate).
# 7.2.3.1. Statistical Methodology Specification

#### **Binary Endpoints**

#### **Endpoint / Variables**

- Proportion of participants achieving ACR20 response.
- Proportion of participants achieving CDAI-LDA (CDAI Total Score≤10).
- Proportion of participants achieving ACR50/70 response.
- Proportion of participants achieving CDAI Remission (CDAI Total Score≤2.8).
- Proportion of participants achieving DAS28-(CRP/ESR) LDA (DAS28-CRP≤3.2 or DAS28-ESR≤3.2).
- Proportion of participants achieving DAS28-(CRP/ESR) remission (DAS28-CRP<2.6 or DAS28-ESR<2.6).</li>
- Proportion of participants achieving good/moderate EULAR response.
- Proportion of participants achieving change from baseline in Van der Heijde mTSS≤0.5/0.

## **Model Specification**

- Each estimate will be generated for each imputed dataset produced by the multiple imputation (MI) procedure described in Section 7.1.1.6, and the corresponding results will be combined using Rubin's rules.
- Binary Endpoints will be statistically analysed using the same methods as for the primary endpoint (see Section 7.1.3.1 for full details) however the model will be adjusted for the following baseline values:

| Binary Endpoint | Baseline adjustment |
|----------------------------------------|---------------------|
| ACR20 | TJC68, SJC66 |
| ACR50 | TJC68, SJC66 |
| ACR70 | TJC68, SJC66 |
| CDAI-LDA | CDAI Total Score |
| CDAI Remission | CDAI Total Score |
| DAS28-CRP LDA | DAS28-CRP |
| DAS28-CRP Remission | DAS28-CRP |
| DAS28-ESR LDA | DAS28-ESR |
| DAS28-ESR Remission | DAS28-ESR |
| Good/Moderate EULAR (CRP) | DAS28-CRP |
| Change from baseline in Van der | mTSS |
| Heijde mTSS≤0.5 | |
| change from baseline in Van der Heijde | mTSS |
| mTSS≤0 | |

- A separate logistic regression model will be fitted for each assessment time point. For time points up to week 12, all treatment arms will be included in the model (i.e. pooled placebo, GSK3196165 150mg, GSK3196165 90mg, tofacitinib 5mg). For time points beyond week 12, only GSK3196165 150mg, GSK3196165 90mg and tofacitinib 5mg randomised treatment arms will be included in the model.
- If at any time point the convergence criterion is not satisfied or maximum likelihood estimates do not exist, then the results of this model will not be reported.

## Model Checking & Diagnostics

• The same model checking and diagnostics will be used as for the primary endpoint. See Section 7.1.3.1 for full details.

#### **Model Results Presentation**

- Binary Endpoints will be presented using the same methods as the primary endpoint. See Section 7.1.3.1 for full details.
- The results from each assessment time point model will be presented within the same output.
- Non-inferiority over tofacitinib on ACR20 will be concluded if the lower limit of the multiplicity corrected 95% CI in the difference in proportions (GSK3196165 minus tofacitinib) is greater than -12% (Note: non-inferiority was calculated using the FDA fixed margin approach [FDA, 2016]).

## **Subgroup Analyses**

See Section 5.4 for details on subgroup analyses.

#### **Sensitivity and Supportive Analyses**

- Sensitivity Analysis on the missing data imputation methods may be performed as described in Section 7.2.1.7.
- Supportive Analysis may be performed as described in Section 7.2.2.

## **Continuous Endpoints**

#### **Endpoint / Variables**

- Change from baseline in HAQ-DI.
- Change from baseline in CDAI Total Score.
- Change from baseline in FACIT-Fatigue score.
- Change from baseline in arthritis pain VAS.
- Change from baseline in TJC28/68 and SJC28/66.
- Change from baseline in CRP (mg/L)
- Change from baseline in PtGA/PhGA.
- Change from baseline in DAS28-(CRP/ESR).
- Change from baseline in SF-36 physical and mental component scores.
- Change from baseline in Van der Heijde mTSS.

## **Model Specification**

- Each estimate will be generated for each imputed dataset produced by the multiple imputation (MI) procedure described in Section 7.1.1.6, and the corresponding results will be combined using Rubin's rules.
- Continuous endpoints will be statistically analysed using an analysis of covariance (ANCOVA)
  comparing each randomised treatment arm with control groups when controlling for treatment
  arm, respective baseline value and previously failed medication (csDMARD only, 1 bDMARD,
  >1 bDMARD).
- A separate ANCOVA will be conducted for each assessment time point.
  - o For time points up to week 12, all treatment arms will be included in the model (i.e. pooled placebo, GSK3196165 150mg, GSK3196165 90mg, tofacitinib 5mg).
  - For time points beyond week 12, only GSK3196165 150mg, GSK3196165 90mg and tofacitinib 5mg randomised treatment arms will be included in the model.
  - For time points beyond week 12, estimates of the least squares means for the placebo switch treatment arms (i.e. placebo to GSK3196165 150mg, placebo to GSK3196165 90mg and placebo to tofacitinib 5mg) will be derived from the model including all six randomised treatment arms.

## **Model Checking & Diagnostics**

• If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### Model Results Presentation

- The results from each assessment time point will be presented within the same output.
- Point estimates and corresponding 95% confidence intervals will be constructed for the treatment differences over placebo and over tofacitinib at each visit using the least squared (LS) means estimates.
- Plots of LS means and corresponding standard errors from the model will be generated for each treatment group by visit.
- Non-inferiority over tofacitinib on change from baseline in CDAI Total score will be concluded
  if the upper limit of the multiplicity corrected 95% CI in the treatment difference (GSK3196165
  minus tofacitinib) is less than 3.5 (Note: non-inferiority was calculated using the FDA fixed
  margin approach [FDA, 2016]).
- Non-inferiority over tofacitinib on change from baseline in Pain VAS will be concluded if the upper limit of the multiplicity corrected 95% CI in the treatment difference (GSK3196165 minus tofacitinib) is less than 5.3 (Note: non-inferiority was calculated using the FDA fixed margin approach [FDA, 2016]).

## **Subgroup Analyses**

See Section 5.4 for details on subgroup analyses.

# Sensitivity and Supportive Analyses

- Sensitivity Analysis on the missing data imputation methods may be performed as described in Section 7.2.1.7.
- Supportive Analysis may be performed as described in Section 7.2.2.
- Non-parametric analyses may be conducted if the normality assumption does not hold.









#### 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Safety analysis will be displayed in three different ways (see Section 5.1.3 for details).

All primary safety analysis will use the "while on treatment" approach, i.e. any safety events which occur post discontinuation of study intervention which are not classified as treatment emergent under the definition specified in Section 14.4.2 will be excluded. A sensitivity analysis will be performed on key safety outputs using the "treatment policy" approach, i.e. all safety events reported in the study will be included.

Missing safety data will not be imputed.

The details of the planned displays are provided in Appendix 12: List of Data Displays.

# 8.1. Adverse Events Analyses

- Adverse events analyses including the analysis of adverse events (AEs), Serious adverse events (SAEs) and other important adverse events will be based on GSK Core Data Standards.
- All AEs will be classified using the current standard GSK Medical Dictionary for Regulatory Activities (i.e. MedDRA version in use at the time of reporting), and grouped by SOC and PT, unless otherwise stated. The MedDRA version will be detailed on every table that uses MedDRA.
- Exposure adjusted event rates per 100 patient years by treatment group will be presented separately for AEs and SAEs.
- Common AEs will be defined as ≥ 5% incidence in any treatment group, unless otherwise specified. Relative risks, based on observed frequencies, for the proportions of subjects with common AEs will be calculated for the comparisons specified in Section 5.1.3.
- AEs with missing intensity will be considered severe.
- Additional safety outputs relating to COVID-19 adverse events including COVID-19 assessments and symptom assessments will be based on GSK Core Data Standards.

# 8.1.1. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.

The details regarding the derivations of adverse events of special interest (AESI) and other important AEs are provided in Section 14.6.4.

Exposure adjusted event rates per 100 patient-years by treatment group will be calculated for each category of AESI and other important AE.

Relative risks, based on observed frequencies, for the proportions of subjects with AESIs will be calculated for the comparisons specified in Section 5.1.3.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, fasting lipids, and liver function tests will be based on GSK Core Data Standards. All laboratory parameters will be summarised, but only laboratory parameters of interest with available CTCAE grades will be used in summary table by grades.

Laboratory parameters of interest are:

- WBCs
- Neutrophils
- Lymphocytes
- Hemoglobin
- Platelets
- ALT
- AST
- ALP
- Bilirubin
- Creatinine
- eGFR
- Total cholesterol
- Low-density lipoprotein (LDL)
- High-density lipoprotein (HDL)
- Triglycerides

Local laboratory parameters will not be included in any summaries and will appear in the listing only.

# 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified.

## 8.3.1. Immunogenicity Analyses

An immune response to GSK3196165 can lead to generation of anti-drug antibodies (ADA). For the immunogenicity assessment, two types of antibody assays will be performed, a binding antibody assay and a neutralizing antibody assay.

For the binding antibody assay, there will be three testing steps: screening, confirmation and titration. The screening assay produces a result of positive or negative relative to a screening cut point. Positive samples continue with the confirmation assay, which also produces a result of positive or negative relative to a confirmation cut point. For samples with a positive confirmation result, a titre value will also be obtained to quantify the degree of binding in a titration assay. Subjects with confirmed positive results, will also be tested in the neutralizing antibody assay, which also reports results as positive or negative.

Subjects will be categorized as positive or negative based on confirmation step and a positive ADA event will further be categorized as transient positive or persistent positive at each visit and for anytime post baseline visit. Transient positive is defined as a single positive immunogenic response where the previous visit is negative, that does not occur at the final study assessment and persistent positive is defined as a positive immunogenic response where the previous visit is positive, or the final study assessment is positive. Titers will be summarized by median, minimum and maximum.

A summary of treatment emergent positive confirmation binding ADA assay results in the subset of subjects who did not have a positive confirmation binding ADA assay result prior to the dosing of study treatment will also be presented.

Neutralizing antibody assay results will be summarised by visit. For anytime post baseline visit, highest result will be used, i.e. according to the following hierarchy: ADA result will be Persistent Positive > Transient Positive > Negative, NAB result will be Positive > Negative and highest titer value.









# 13. REFERENCES

Bretz F, Maurer W, Brannath W, Posch M. A graphical approach to sequentially rejective multiple test procedures. Stat Med. 2009;28(4):586-604.

FDA (Food and Drug Administration). Guidance for Industry: Non-Inferiority Clinical Trials to Establish Effectiveness. 2016. https://www.fda.gov/media/78504/download

Freynhagen R, Baron R, Gockel U, Tölle T.R, CurrMed ResOpin Vol 22, 2006, 1911-1920 © 2006 Pfizer Pharma GmbH, Pfizerstr.1, 76139 Karlsruhe, Germany.

ICH HARMONISED GUIDELINE. Addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials E9(R1). 2019. https://database.ich.org/sites/default/files/E9-R1\_Step4\_Guideline\_2019\_1203.pdf

NCI. National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 NCI, NIH, DHHS. 2017

 $https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/CTCAE\_v5\_Q\\uick\_Reference\_5x7.pdf$ 

Roger JH, Bratton DJ, Mayer B, Abellan JJ, Keene ON. Treatment policy estimands for recurrent event data using data collected after cessation of randomised treatment. Pharmaceutical Statistics. 2019;18:85–95.

# 14. APPENDICES

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 14.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| 01 | Participant was randomised despite not meeting an eligibility criteria which, in the judgement of the clinical team, constitutes an exclusion from the Per protocol population (Subset of Important Protocol Deviations with GSK category 2) |
| 02 | Medication/Vaccine excluded by the protocol was administered, including those restricted prior to the study, during the study and/or during the safety follow-up of the study (Important Protocol Deviations with GSK categories 4A or 4B) |
| 03 | Participant substantially did not receive medication as planned per protocol (Important Protocol Deviations with GSK category 7A). |
| 04 | Participant received medication while in contraindication (Important Protocol Deviations with GSK category 7B) |
| 05 | Participant received wrong study treatment or assignment (Important Protocol Deviations with GSK category 7C) |
| 06 | Participant had significant non-compliance or dose modification of background treatment (Important Protocol Deviations with GSK category 7OT) |
| 07 | Participant developed withdrawal criteria specified in the protocol but were not withdrawn and continued dosing (Important Protocol Deviations with GSK category 3A, 3B or 3OT) |
| 08 | Study blind/unblind procedures: Investigator/site staff/participant/GSK Clinical team did not remain blinded to treatment assignment through Week 52 Exit visit efficacy evaluation, includes emergency unblinding for medical reasons (Important Protocol Deviations with GSK category 8B) |
| 09 | Other: a deviation that does not satisfy the above criteria, however, in the judgment of the clinical team, including the medical monitor, constitutes an exclusion from the Per Protocol population. |

# 14.2. Appendix 2: Schedule of Activities

# 14.2.1. Protocol Defined Schedule of Events

# SoA – Screening Period

| | Participant Screening Task List |
|---|---|
| | (after informed consent, all screening assessments must be completed within the 42 days prior to Randomisation) |
| | Day -42 to Day -1 |
| | $\downarrow$ |
| | Informed Consent and optional Genetics consent |
| | Inclusion/exclusion criteria |
| | Participant Demographics |
| | Medical, disease and therapy history Review of asthma/COPD/pulmonary disease |
| | history |
| | Concomitant Medication Review |
| | 12-lead ECG1 |
| | Vital signs |
| w | Full Physical Exam |
| ent | Dyspnoea & Cough assessment, Lung |
| Sm | Auscultation, Pulse Oximetry |
| Assessments | TB evaluation |
| As | SAE assessment |
| | Swollen (66) & Tender (68) joint count <sup>2</sup> |
| | Hands and feet X-ray³ |
| | Chest X-ray (posteroanterior) <sup>4</sup> |
| | Haematology, Chemistry, Urinalysis (dip stick) |
| abs. | HIV, TB, Hepatitis B & Hepatitis C screen hsCRP |
| La | Serum pregnancy test <sup>5</sup> |
| | Lipid profile <sup>6</sup> |
| | Lipia promo |

#### Screening assessment notes

- 1) ECGs should be performed before vital signs and blood draws.
- 2) Joint assessments should be performed by an independent assessor. Where possible the same assessor should perform all joint assessments for an individual participant.
- 3) Will be read centrally & imaging CRO will assess presence or absence of erosion(s).
- 4) Unless performed within previous 12 weeks.
- 5) For women of child-bearing potential.
- 6) Fasting is not required, but 6hr fasting status at time of blood draw must be noted on requisition form.

| SoA – Treatment Period | | | | | | | | | 96165<br>V0-11) | | | | • | Tofac | itin | on GSI<br>ib (W1 | 2-52 | ) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week | | | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13 | 14-15 | 16 | 17-23 | 24 | 25-35 | 36 3 | 7-47 | 48 | 49-51 | 52 |
| | Assessment visit Day Study activities <sup>1</sup> | Baseline Day 1 | Day 8 (±2d) | Day 15 (±2d) | Day 22 (±2d) | Day 29 (±2d) | | Day 57 (±2d) | | Primary endpoint<br>Day 85 (±3d) | Day 92 (±3d) | | Day 113 (±5d) | | Day 169 (±7d) | | Day 253 (±7d) | | Day 337 (±7d) | | End of treatment<br>Day 365 (± 7d) |
| | Randomisation | Χ | | | | | | | | | | | | | | | | | | | |
| | Arthritis pain VAS, PtGA, HAQ-DI | Χ | Χ | Χ | | Х | | Χ | | Х | Χ | | Χ | | Χ | | Х | | | | X |
| | PROMIS Pain Interference | Х | Χ | | | Χ | | | | Χ | | | Χ | | Χ | | Х | | | | Χ |
| S | PainDETECT | Χ | | | | | | | | | | | | | | | | | | | |
| PR0s1 | RA Symptom & Impact questionnaire | Χ | Х | | | Χ | | | | Χ | | | Χ | | Χ | | Х | | | | X |
| - | FACIT-Fatigue, SF-36, PROMIS Sleep | Χ | | | | Χ | | | | Χ | | | Χ | | Χ | | Х | | | | X |
| | Participant Feedback questionnaire | | | | | | | | | Χ | | | | | | | | | | | Χ |
| | 12-lead ECG2 (S=single, T=triplicate) | | | | | | | | | S | | | | | | | | | | | Т |
| | Vital signs | Χ | | Χ | | Χ | | Χ | | Χ | Χ | | Χ | | Χ | | X | | | | X |
| | Brief Physical Exam | Χ | | Χ | | | | | | Χ | Χ | | Χ | | Χ | | Х | | | | X |
| Assessments | Dyspnoea & Cough assessment, Lung<br>Auscultation, Pulse Oximetry | Х | Х | Х | | Χ | | Х | | X | Χ | | Χ | | Χ | | Х | | | | Х |
| ess | Pulmonary function tests (FEV <sub>1</sub> , FVC) | X17 | | | | | | | | | | | | | | | | | | | |
| Ass | Swollen (66) & Tender (68) joint count <sup>3</sup> | Χ | Χ | Χ | | Χ | | Χ | | Χ | Χ | | Χ | | Χ | | X | | | | X |
| | Physician Global Assessment <sup>4</sup> | Χ | Χ | Χ | | Χ | | Χ | | X | X | | Χ | | Χ | | X | | | | X |
| | Hands and Feet X-ray⁵ | | | | | | | | | Χ | | | | | Χ | | | | | | X |
| | Chest x-ray (posteroanterior) | | | | | | | | | | | | X6 | | | | | | | | |
| | Haematology, Chemistry, Urinalysis | Χ | | Χ | | Χ | | Χ | | Χ | Χ | | Χ | | Χ | | X | | Χ | | X |
| | Lipid profile <sup>7</sup> | | | | | Χ | | | | | | | Χ | | | | | | | | X7 |
| draws | Urine pregnancy test8 | Χ | | | | Χ | | Χ | | Χ | | | Χ | | _ | Ev | - 1 | weel | (S - | > | X |
| <del>L</del> a | hsCRP, ESR9 | Χ | Χ | Χ | | Χ | | Χ | | Χ | Χ | | Χ | | Χ | | X | | | | X |
| poold | RF, ACPA (anti-CCP) | Χ | | | | | | | | | | | | | | | | | | | |
| ğ | TB testing | | | | | | | | | | | | | | | | | | Χ | | |
| and | Pre-dose PK sample (& GMCSF complex) | | | Χ | | Χ | | Χ | | X | | | Χ | | Χ | | X | | | | X |
| Labs | Immunogenicity blood sampling | X10 | | Χ | | Χ | | | | Χ | | | Χ | | Χ | | X | | | | X |
| 2 | Genetic sample <sup>11</sup> | Χ | | | | | | | | | | | | | | | | | | | |
| | Sampling for RNA analysis <sup>12</sup> | X | | | | Χ | | | | X | | | | | Χ | | | | | | |
| | Blood PD & Biomarkers <sup>12</sup> | Χ | Χ | Χ | | Χ | | | | Χ | | | | | Χ | | | | | | |
| Dose | Dispense: Weekly SC injection <sup>13,14</sup> | | X13 | Χ | < | | X <sup>14</sup> | | > | X13 X13 <> | | | | | | | | | | | |
| ŏ | Dispense: BID oral intervention <sup>15</sup> | X X X X < Every 4 weeks | | | | | | | | | | | | | | | | | | | |
| | SAE/AE review <sup>16</sup> | < | | | | | | | | | | | | | | | | | | | |
| | Concomitant medication review <sup>16</sup> < | | | | | X> | | | | | | > | | | | | | | | | |
| | AE/conmed phone call if no site visit 16 | visit 16 Weekly to Week 12 Every two weeks to W36, every four weeks to W52 | | | | | | | | | | | | | | | | | | | |

#### Notes

- PROs should be completed first, before any other assessments, procedures or consultations, to avoid influencing participants' perception.
- ECGs should be performed before vital signs and blood draws, where possible.
- Joint assessments should be performed by an independent assessor. Where possible the same assessor should perform all joint assessments for an individual participant.
- Where possible, the same individual should perform all physician global assessments for an individual participant.
- Will be centrally read & assessed for presence or absence of erosion(s).
- . Schedule X-ray between Weeks 48-51.
- Fasting is not required, but 6hr fasting status at time of blood draw must be noted on requisition form.
- For women of child-bearing potential.
- ESR measured locally (using kit provided) by unblind site staff.
- Day 1 sample includes anti-GM-CSF autoantibody and free GM-CSF analysis.
- Genetics consenting participants only.
- Selected sites only. Refer to site information and laboratory manual.
- Monitor participants for 1 hour after SC dosing at site at Weeks 0, 1, 12 and 13.
   SC injection must be administered at site when dosing on assessment visit days.
- Dispense weekly for site administration;
   OR if available, dispense PFS in boxes of 4, every 4 weeks, for home SC dosing.
- Dispense 2 bottles of oral intervention every 4 weeks.
- Minimum weekly review to Week 12, then every two weeks to Week 36, then every four weeks to Week 52. A phone call is acceptable if a site visit is not scheduled.
- 17. May be performed before Day 1 if required.

# SoA - Safety Follow-up Visit

| | Safety follow-up visit procedures |
|---|---|
| | (Follow-up visit only for participants who do not transition into LTE study 209564) |
| | Week 59 (Day 414 $\pm$ 14 days) |
| | $\downarrow$ |
| | Vital signs |
| Assessments | Full Physical Exam |
| l sme | Dyspnoea & Cough assessment, Lung Auscultation, |
| ess | Pulse Oximetry |
| Ass | Concomitant Medication Review |
| , | SAE/AE review |
| | Haematology, Chemistry, Urinalysis (dip stick) |
| -abs | Urine pregnancy test (for women of child bearing |
| La | potential only) |
| | Immunogenicity blood sampling |

# **Assessments for Early Withdrawal from Study**

Follow the Week 52 procedures\* at the time of withdrawal from the study, or within 1 week of withdrawal, and schedule a safety follow-up visit 8 weeks post last dose of SC administered study intervention.

\*Note: A hands/feet x-ray should not be performed at early withdrawal if the participant's last dose of study drug was prior to week 8, OR if a hands/feet x-ray has been carried out within 8 weeks of the early withdrawal date, as part of study assessments.

# 14.3. Appendix 3: Assessment Windows

# 14.3.1. Definitions of Assessment Windows for Analyses

Data will be analysed as per the planned visit assignment.

Early withdrawal and unscheduled visits will be slotted to the appropriate planned visit. The assigned visit will be based on the interval in which the Study Day for the early withdrawal or unscheduled visit falls according to intervals provided below.

| Analysis Set / Domain | Target | Analysis | Window | Analysis |
|---|---|---|---|---|
| | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | Day-1 | Day -42 | Day -1 | Screening |
| All [1] | Day 1 | Day 1 | Day 1 | Baseline |
| All (Efficacy, lung auscultation and pulse oximetry) [1] | Day 8 | Day 2 | Day 11 | Week 1 |
| All (Safety) [2] | Day 15 | Day 2 | Day 22 | Week 2 |
| All (Efficacy, lung auscultation and pulse oximetry) [1] | Day 15 | Day 12 | Day 22 | Week 2 |
| All [1] | Day 29 | Day 23 | Day 43 | Week 4 |
| All [1] | Day 57 | Day 44 | Day 71 | Week 8 |
| Imaging | Day 85 | Day 2 | Day 127 | Week 12 |
| All [1] | Day 85 | Day 72 | Day 88 | Week 12 |
| All [1] | Day 92 | Day 89 | Day 95 | Week 13 |
| All [1] | Day 113 | Day 96 | Day 141 | Week 16 |
| All [1] | Day 169 | Day 142 | Day 211 | Week 24 |
| Imaging | Day 169 | Day 128 | Day 267 | Week 24 |
| All (Safety) | Day 253 | Day 212 | Day 295 | Week 36 |
| All (Efficacy) [1] | Day 253 | Day 212 | Day 309 | Week 36 |
| All (Safety) | Day 337 | Day 296 | Day 351 | Week 48 |
| All (Safety) | Day 365 | Day 352 | Day 399 | Week 52 |
| All (Efficacy) [1] | Day 365 | Day 310 | Day 399 | Week 52 |
| Imaging | Day 365 | Day 268 | Day 399 | Week 52 |
| All (Safety) | Day 414 | Day 400 | Day 400+ | 8 week Follow-<br>up (for<br>participants<br>who don't<br>transition into<br>LTE study) |
| Safety (participants withdrawn early from treatment) | 56 days after last treatment | 42 days after last treatment | 70 days after last treatment | 8 Week Follow<br>Up |

#### NOTES:

- If there are two slotted values within a time window, the value closest to the target day for that window will be used except for ECGs and X-Rays where multiple measures are expected. If values are the same distance from the target, then the mean will be taken.
- [1] Excluding Imaging.
- [2] Excluding lung auscultation and pulse oximetry

# 14.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 14.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date.

On-Treatment AEs well be reported as treatment emergent AEs (TEAE). Definition for TEAE can be found in Section 14.4.2.

If an AE happened at week 12 visit, it will be assigned to Period 2.

# For Placebo:

| Study Phase | Period | Definition |
|---|---|---|
| Pre-Treatment | | Date ≤ Study Treatment Start Date |
| On-Treatment | Period 1 | Study Treatment Start Date < Date ≤ Week 12 Visit Date or Early Withdrawal (if before Week 12) Visit Date |
| Off-Treatment | | Study Treatment Stop Date < Date ≤ Study Treatment Stop Date + |
| Safety Follow-Up[1] | | 56 days |
| Off-Treatment | | Date ≥ Study Treatment Stop Date + 56 days |

<sup>[1]</sup> The safety follow up definition for Placebo is only valid for participants who withdraw early. The participants that are on placebo who complete Period 1, will continue into Period 2.

#### For GSK3196165:

| Study Phase | Period | Definition |
|---|---|---|
| Pre-Treatment | | Date ≤ Study Treatment Start Date |
| On-Treatment | Period 1 | Study Treatment Start Date < Date ≤ Week 12 Visit Date or Early Withdrawal (if before week 12) Visit Date+ 7 days |
| | Period 2 | Week 12 Visit Date < Date ≤ Study Treatment Stop Date + 7 days or Early Withdrawal (if after week 12) Visit Date + 7 days |
| Off-Treatment<br>Safety Follow-Up | | Study Treatment Stop Date + 7 days < Date ≤ Study Treatment Stop Date + 56 days |
| Off-Treatment | | Date ≥ Study Treatment Stop Date + 56 days |

#### For Tofacitinib:

| Study Phase | Period | Definition |
|---|---|---|
| Pre-Treatment | | Date ≤ Study Treatment Start Date |
| On-Treatment | Period 1 | Study Treatment Start Date < Date ≤ Week 12 Visit Date or Early Withdrawal (if before week 12) Visit Date+ 1 day |
| | Period 2 | Week 12 Visit Date< Date ≤ Study Treatment Stop Date + 1 day or Early Withdrawal (if after week 12) Visit Date + 1 day |
| Off-Treatment<br>Safety Follow-Up | | Study Treatment Stop Date + 7 days < Date ≤ Study Treatment Stop Date + 56 days |

| Study Phase | Period | Definition |
|---------------|--------|--------------------------------------------|
| Off-Treatment | | Date ≥ Study Treatment Stop Date + 56 days |

## 14.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | Any medication that started before first dose of study treatment |
| Concomitant | Any medication that is taken post first dose of study treatment, regardless of whether it was started prior to the first dose of study treatment or not |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 14.4.1.2. Study Phases for Efficacy Assessments

| Study Phase | Definition |
|------------------|-------------------------------------------|
| Pre Early | |
| Treatment | Date ≤ Study Treatment Stop Date + 7 days |
| Withdrawal | |
| Post Early | |
| Treatment | Date ≥ Study Treatment Stop Date +7 days |
| Withdrawal (Off- | Date 2 Study Treatment Stop Date +7 days |
| Treatment) | |

# 14.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | • Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 56 |
| Emergent | days. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.
- If AE happens on the week 12 visit date, it will be assigned to period 2.

# 14.5. Appendix 5: Data Display Standards & Handling Conventions

# 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software 9.4 will be used. | |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound | : GSK3196165/MID201791 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for the final reporting effort for tables and listings. | |

# 14.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DPs) will be adopted for reporting
  of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DPs.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be slotted as stated in Section 14.3.1 unless otherwise stated.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7 01 to 7 13 | |



# 14.5.4. Reporting Standards for Log-transformed Parameters

| Reporting of Log-Transformed Parameters | |
|---|---|
| Descriptive | N, n, geometric mean, 95% CI of geometric mean, geometric coefficient of |
| Summary Statistics | variation (CV <sub>b</sub> (%)) will be reported. |
| | [1] $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| Figures | Axes will be presented with actual values with an appropriate log-scale (either |
| | base 2 or base 10) depending on range of values |

# 14.6. Appendix 6: Derived and Transformed Data

#### 14.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Data will be analysed as per the planned visit assignment.
- Early withdrawal and unscheduled visits will be slotted to the appropriate planned visit (as per Section 14.3.1). If there are two slotted values within a time window the value closest to the target day for that window will be used except for ECGs and X-Rays where multiple measures are expected. If values are the same distance from the target, then the mean will be taken.
- In the instance of both local and central labs being collected at the same timepoint, only the central labs will be used in any analysis.
- Triplicate ECG measures will be averaged for each subject and visit prior to generating summary tables
- Multiple X-Ray measures from multiple readers will be handled as described in Section 14.6.3.10.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### Period 1 (Up to Week 12)

- Period 1 (up to week 12) is defined as time from randomisation up to dosing of period 2 study medication (week 12) or date of study withdrawal or date of treatment withdrawal plus follow up, whichever is earlier.
- A participant completed 12 weeks of treatment if study medication (injection) was administered at week 11 visit or later up to next study medication administration or study medication (capsule) was administered at week 11 plus 6 days or later up to next study medication administration
- A participant completed week 12 if week 12 assessments were performed and study medication of the next period was administered.
- A participant withdrew from the study if the withdrawal date is < date of study medication administration of next period (week 12)

# Period 2 (Post Week 12)

- Period 2 (post week 12) is defined as time from first dose of study medication of period 2 (Week 12)
  until date of study completion or date of study withdrawal or date of treatment withdrawal plus safety
  follow up whichever is earlier.
- A participant withdrew from the study if the withdrawal date > date of study medication administration of period 2

#### **Study Completion**

- For subjects not entering LTE study: completion of study is defined as completion of treatment plus follow up period.
- For subjects entering LTE: completion of study is defined as completion of the week 52 visit.

#### 14.6.2. Study Population

#### **Treatment Compliance**

• Treatment compliance will be calculated based on the formula:

For GSK3196165:

#### Treatment Compliance =

(Number of Actual Doses / Planned Treatment Duration in Weeks) \*100

For tofacitinib:

# **Treatment Compliance =**

# (Number of Actual Doses / (Planned Treatment Duration in Weeks\*14)) \*100

- Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is 52 weeks.
- Compliance for early treatment discontinuation participants will only be calculated up until the date of early treatment discontinuation.

## Date of Birth and Age

- Only the year of birth will be captured, and therefore the date of birth is then derived as follows:
   Year of birth = YYYY → Date of birth = 30th June YYYY
- Age in years will be calculated as integer part of (latest of (randomisation date, screening date)— date of birth). Birth date will be presented in listings as 'YYYY'.

## **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

For GSK3196165:

Duration of Exposure in Days = I/Treatment stop date - treatment start d

Duration of Exposure in Days = [(Treatment stop date – treatment start date) + 7][(Number of missed injections) \* 7]

For Tofacitinib:

# Duration of Exposure in Days =(Total capsules consumed/2) + 1

 Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure. The cumulative dose will be based on the formula:

**Cumulative Dose = Sum of Total Dose at Each Visit** 

#### **Disease History/Duration**

• RA duration since diagnosis in years will be calculated based on the formula:

RA Duration Since Diagnosis in Years =

(Date of First Dose of Study Treatment - Start date of RA diagnosis + 1)/365.25

RA duration since first symptoms in years will be calculated based on the formula:

RA Duration Since First Symptoms in Years =

• (Date of First Dose of Study Treatment - Start date of first symptoms + 1)/365.25

#### **Stratification Stratum (Previously Failed Medication)**

• Stratification stratum will be derived from the randomisation numbers as follows:

| Randomization Numbers | Stratum |
|--------------------------------|--------------|
| 10001 – 12700<br>18101 – 20800 | csDMARD only |

| | 12701 – 15400<br>20801 – 23500 | 1 bDMARD |
|---|--------------------------------|-----------|
| • | 15401 – 18100<br>23501 – 26200 | >1 bDMARD |

# **Corticosteroid Scaling Factor**

- To assess corticosteroid use and determine average daily corticosteroid dose, all
  corticosteroid dosages will be converted to a prednisone equivalent in milligrams by
  multiplying the dose of the steroid (using the coded term from GSKDrug) by the conversion
  factor to get prednisone equivalent units.
- The following conversion factors will be used:

| Corticosteroid | Scaling Factor |
|--------------------------------|----------------|
| Betamethasone | 8.333 |
| Dexamethasone | 6.667 |
| Meprednisone | 1.25 |
| Methylprednisolone | 1.25 |
| Methylprednisolone Sodium | 1.25 |
| Succinate | |
| Prednisolone | 1 |
| Prednisone, Prednisone Acetate | 1 |
| Triamcinolone | 1.25 |
| Predmet (NOS) | 1.25 |
| Deflazacort | 0.833 |

#### **Prior and Concomitant Medication**

#### RA Concomitant medication will be split into following categories:

- DMARDs
  - Methotrexate (all methotrexate medications combined into one category)
  - Other csDMARDs (not Methotrexate)
  - csDMARDs > 1
  - bsDMARDs/boDMARDs/tsDMARDs
- Corticosteroids (the following groups will be derived by route)
  - -Oral
  - -Intra-Articular
- Other RA medications

#### Prior RA medications will be split into following categories:

- -DMARDs
  - Methotrexate (all methotrexate medications combined into one category)
  - Other csDMARDs (not Methotrexate)
  - csDMARDs >1
  - -bsDMARDs/boDMARDs/tsDMARDs
    - ->=1 of the above
    - -=1 of the above
    - ->1 of the above

#### **Prior and Concomitant Medication**

- -Inadequate response to >=1 bs/boDMARD
- -Inadequate response to >=1 tsDMARD
- -Inadequate response to >1 bsDMARD/boDMARD/tsDMARD
- -Oral corticosteroids
- -Other RA medications

#### RA Concomitant medication will be derived as following:

Follow Section 14.4.1.1 for definition of "concomitant" medication.

#### o DMARDs:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using all "medication type" which includes C1SCAT="CONVENTIONAL SYNTHETIC DMARDS", C1SCAT="BIOLOGICAL ORIGINATOR DMARDS", C1SCAT="BIOSIMILAR DMARDS", and C1SCAT="TARGETED SYNTHETIC DMARDS".

#### Methotrexate:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG", using C1SCAT="CONVENTIONAL SYNTHETIC DMARDS" where ingredient/CMDECOD contains "METHOTREXATE". All methotrexate medications will be combined together into one category called "Methotrexate"

Other csDMARDs (not methotrexate):

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG", using C1SCAT="CONVENTIONAL SYNTHETIC DMARDS", but excluding methotrexate (where ingredient/CMDECOD contains "METHOTREXATE")

#### o csDMARDs > 1:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using C1SCAT="CONVENTIONAL SYNTHETIC DMARDS" where a participant has taken more than 1 csDMARD (2 or more).

#### bsDMARDs/boDMARDs/tsDMARDs:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using "medication type" which includes C1SCAT="BIOLOGICAL ORIGINATOR DMARDS", C1SCAT="BIOSIMILAR DMARDS" and C1SCAT="TARGETED SYNTHETIC DMARDS".

#### Corticosteroids Oral:

Derived from "RA other medication" page in eCRF, C1CAT="OTHER RHEUMATOID ARTHRITIS MEDICATION" using C1SCAT= "CORTICOSTEROID" and C1ROUTE="ORAL"

#### Corticosteroids IA:

Derived from "Intra-Articular Corticosteroids" page in eCRF,C1CAT="OTHER RHEUMATOID ARTHRITIS MEDICATION" using C1SCAT="CORTICOSTEROID" and C1ROUTE = "INTRA-ARTICULAR"

#### Other RA medication:

Derived from "RA other medication" page in eCRF, C1CAT="OTHER RHEUMATOID ARTHRITIS MEDICATION" using all "medication type" which includes C1SCAT="Corticosteroid" all routes except

#### **Prior and Concomitant Medication**

C1ROUTE="ORAL" and C1ROUTE="INTRA-ARTICULAR", C1SCAT="OPIOID" and C1SCAT="OTHER".

#### Non-RA Concomitant medication will be derived as following:

Follow Section 14.4.1.1 for definition of "concomitant" medication.

Non RA medication is derived from "Non-RA concomitant medications" page in eCRF, C1CAT="NON RHEUMATOID ARTHRITIS MEDICATION".

Uncoded concomitant medication will be combined together in one category called "Uncoded"

#### Prior RA medication will be derived as following:

Follow Section 14.4.1.1 for definition of "prior" medication.

#### DMARDs:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using all "medication type" which includes C1SCAT="CONVENTIONAL SYNTHETIC DMARDS", C1SCAT="BIOLOGICAL ORIGINATOR DMARDS", C1SCAT="BIOSIMILAR DMARDS" and C1SCAT="TARGETED SYNTHETIC DMARDS".

#### Methotrexate:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using C1SCAT="CONVENTIONAL SYNTHETIC DMARDS" where ingredient/CMDECOD contains "METHOTREXATE". All methotrexate medications will be combined together into one category called "Methotrexate"

#### Other csDMARDs (not methotrexate):

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using C1SCAT="CONVENTIONAL SYNTHETIC DMARDS" where ingredient/ CMDECOD contains "METHOTREXATE".

#### o csDMARDs > 1:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using C1SCAT="CONVENTIONAL SYNTHETIC DMARDS" where a participant has taken more than 1 csDMARD.

#### bsDMARDS/boDMARDs/tsDMARDs:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" using C1SCAT="BIOSIMILAR DMARDS", C1SCAT="BIOLOGICAL ORIGINATOR DMARDS" and C1SCAT="TARGETED SYNTHETIC DMARDS".

- >=1 of the above is derived as above for participants that have taken at least one of the bsDMARDS, boDMARDs or tsDMARDs
- =1 of the above is derived as above for participants that have taken one of the bsDMARDS, boDMARDs or tsDMARDs
- >1 of the above is derived as above for participants that have taken more than one of the bsDMARDS, boDMARDs or tsDMARDs

#### **Prior and Concomitant Medication**

o Inadequate response to >=1 bs/boDMARD:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" where a subject had at least one of the following: C1SCAT="BIOSIMILAR DMARDS" or C1SCAT="BIOLOGICAL ORIGINATOR DMARDS", with one or more of the following selected "lack of initial efficacy" or "loss of efficacy" or "adverse event", QNAM="PRSMEDEN" and QVAL contains "ADVERSE EVENT", "LACK OF INITIAL EFFICACY", or "LOSS OF EFFICACY".

Inadequate response to >=1 tsDMARD:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" where a subject had at least one C1SCAT="TARGETED SYNTHETIC DMARDS", with one or more of the following selected "lack of initial efficacy" or "loss of efficacy" or "adverse event", QNAM="PRSMEDEN" and QVAL contains "ADVERSE EVENT", "LACK OF INITIAL EFFICACY", or "LOSS OF EFFICACY".

Inadequate response to >1 bsDMARD/boDMARD/tsDMARD:

Derived from "RA Medications MTX, csDMARD and bDMARD" page in eCRF, C1CAT="DISEASE-MODIFYING ANTIRHEUMATIC DRUG" where a subject had at least two of the following: C1SCAT= "BIOSIMILAR DMARDS" or C1SCAT="BIOLOGICAL ORIGINATOR DMARDS" or "C1SCAT=TARGETED SYNTHETIC DMARDS", with one or more of the following selected "lack of initial efficacy" or "loss of efficacy" or "adverse event", QNAM="PRSMEDEN" and QVAL contains "ADVERSE EVENT", "LACK OF INITIAL EFFICACY", or "LOSS OF EFFICACY".

Corticosteroids Oral:

Derived from "RA other medication" page in eCRF, C1CAT="OTHER RHEUMATOID ARTHRITIS MEDICATION" using C1SCAT= "CORTICOSTEROID" and C1ROUTE= "ORAL".

Other RA medication:

Derived from "RA other medication" page in eCRF, C1CAT="OTHER RHEUMATOID ARTHRITIS MEDICATION" using all "medication type" which includes C1SCAT="corticosteroid" which includes all routes except C1ROUTE="ORAL", C1SCAT="OPIOID" and C1SCAT="OTHER".

The following medications will be combined into one category:

- All Methotrexate medications will be combined into one category called "Methotrexate"
- Hydroxychloroguine and Hydroxychloroguine Sulfate will be combined into "Hydroxychloroguine"
- Chloroquine, Chloroquine Phosphate and Chloroquine Sulfate will be combined into "Chloroquine"
- Filgotinib and Filgotinib Maleate will be combined into "Filgotinib"
- Tofacinitib and Tofacitinib Citrate will be combined into "Tofacitinib"

#### **Concomitant COVID-19 Vaccine**

 COVID-19 Vaccines will be derived from the most recent list of terms provided by GSK Medical Dictionary at the time of reporting

## 14.6.3. **Efficacy**

#### 14.6.3.1. ACR20/50/70

#### ACR20/50/70

#### Proportion of ACR20/50/70 responders

- The American College of Rheumatology's (ACR) definition for calculating improvement in RA is calculated as a 20% improvement (ACR20) in both tender and swollen joint counts and 20% improvement in 3 of the 5 remaining ACR-core set measures: patient and physician global assessments, patient's assessment of arthritis pain, disability, and an acute-phase reactant (i.e. CRP value). Similarly, ACR50 and ACR70 are calculated with the respective percent improvement. This efficacy measurement will be made at every post-baseline study assessment time point.
- The specific components of the ACR Assessments that will be used in this study are:
  - Tender/Painful Joint count 68 (TJC68)
  - Swollen Joint Count 66 (SJC66)
  - o Patient's Assessment of Arthritis Pain
  - Patient's Global Assessment of Arthritis Disease Activity
  - Physician's Global Assessment of Arthritis
  - CRP (mg/L)
  - Health Assessment Questionnaire Disability Index (HAQ-DI)
- Individual components collected outside of a +/- 2 day window from visit date will be considered missing for the purpose of the ACR calculation.
- For all visits, if any of the component scores are missing, then those scores will be considered as not having met the criteria for improvement. Therefore, if TJC68 or SJC66 or 3 or more of the 5 remaining ACR-core set measures are missing, ACR20/ ACR50/ ACR70 will each be considered missing.
- For component scores with missing Baseline values or a Baseline value of 0, the percentage
  improvement can't be calculated, and the component will be considered as missing for all visits. If
  the baseline value is missing, do not use screening visit data for imputation.

#### 14.6.3.2. Tender/Painful and Swollen Joint Counts

#### Tender/Painful Joint Count (TJC) and Swollen Joint Count (SJC)

#### TJC28/68 and SJC28/66

- Four different scores will be calculated to evaluate swelling and tenderness of joints. TJC28 and SJC28 will take 28 joints into account, SJC66 and TJC68 will use 66 and 68 joints, respectively.
- The assessment for swelling is the total number of joints with a present swelling and ranges from 0 to 28 for SJC28 and 0 to 66 for SJC66.
- The assessment for tenderness is the total number of joints with a present tenderness and ranges from 0 to 28 for TJC28 and 0 to 68 for TJC68.
- The following 28 joints will be taken into account for TJC28 and SJC28: Shoulder (2 joints), Knee (2), Elbow (2), Wrist (2), Fingers (PIP, MCP: 20).
- Additionally, the following joints will be taken into account for SJC66/TJC68: Temporomandibular (2), Sternoclavicular (2), Acromioclavicular (2), Fingers (DIP: 8), Ankle (2), Tarsus (2), Toes (PIP, MTP: 20), Hip (2, only for TJC).

- Replaced or fused joints are considered non-evaluable in the swelling and tenderness assessment.
- If there are missing observations for tender or swollen joints, then the remaining observations will be assessed and weighted by dividing the number presented by number of non-missing and by multiplying by 28/66/68 for the joint count.
- If a joint has undergone inter-articular injection of corticosteroid during the course of the study, this joint is recorded in the concomitant medication dataset. The joint will be considered to be tender and swollen for 8 weeks post IA corticosteroid injection.

#### 14.6.3.3. Pain VAS

#### Patient's assessment of Arthritis Pain VAS

#### Pain VAS

• Subjects will assess the severity of their current arthritis pain using a continuous visual analog scale (VAS) with anchors "0" (CCL COLORS).

# 14.6.3.4. Patient's/Physician's Global Assessment of Arthritis Disease Activity

## Patient's/Physician's Global Assessment of Arthritis Disease Activity (PtGA/PhGA)

#### **PtGA**

• Subjects will complete a global assessment of disease activity using the patient global assessment of disease activity (PtGA) item, a continuous VAS with anchors "0" (CCI COLORS) to "100" (CCI COLORS).

#### **PhGA**

 Physicians will complete a global assessment of disease activity using the physician global assessment of disease activity item (PhGA), a continuous VAS with anchors "0" (CCI) to "100"

#### 14.6.3.5. HAQ-DI Questionnaire

#### HAQ-DI

#### HAQ-DI

- The functional status of the subject will be assessed by means of the Disability Index of the Stanford Health Assessment Questionnaire (HAQ-DI). This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas:
  - Dressing & grooming (HAQ0201, HAQ0202)
  - Arising (HAQ0203, HAQ0204)
  - Eating (HAQ0205, HAQ0206, HAQ0207)
  - Walking (HAQ0208, HAQ0209)
  - Hygiene (HAQ0223, HAQ0224, HAQ0225)
  - Reach (HAQ0226, HAQ0227)
  - Grip (HAQ0228, HAQ0229, HAQ0230)
  - Common daily activities (HAQ0231, HAQ0232, HAQ0233)
- Each functional area contains at least two questions. For each question, there is a four-level response set that is scored from 0 (CCI) to 3 (CCI). Each functional area is scored as the maximum value of their component activities (0,1,2 or 3).
- If aids/devices or help from another person are used for a specific functional area and the maximum response of this functional area is 0 or 1 the according value is increased to a score of 2. If "other" is

#### HAQ-DI

marked as an aid or equipment, then this can be assigned to a group of four functional areas and will be handled as an aid or equipment for each of the four functional areas. Therefore, if the maximum score of a functional area is 0 or 1 that value is increased to a score of 2 for each of the four functional areas:

| Aid/device | Will be associated with functional area |
|---|---|
| Cane (HAQ0210) | Walking |
| Walker (HAQ0211) | |
| Crutches (HAQ0212) | |
| Wheelchair (HAQ0213) | |
| Devices used for dressing (HAQ0214) | Dressing and grooming |
| Built Up or Special Utensils (HAQ0215) | Eating |
| Special or Built Up Chair (HAQ0216) | Arising |
| Raised toilet seat (HAQ0234) | Hygiene |
| Bathtub bar (HAQ0237) | |
| Bathtub seat (HAQ0235) | |
| Long-handled appliance in bathroom (HAQ0239) | |
| Long-handled appliance for reaching (HAQ0238) | Reach |
| Jar opener (HAQ0236) | Grip |
| Other Aid (Dress/Arising/Eat/Walk) (HAQ0217) | Dressing & grooming, Arising, Eating, Walking |
| Other Aid (Hygiene/Reach/Grip/Act) (HAQ0240) | Hygiene, Reach, Grip, Common daily activities |

| Help from another person | Will be associated with functional area |
|-----------------------------------|-----------------------------------------|
| Walking (HAQ0222) | Walking |
| Dressing and Grooming (HAQ0219) | Dressing and grooming |
| Eating (HAQ0221) | Eating |
| Arising (HAQ0220) | Arising |
| Hygiene (HAQ0242) | Hygiene |
| Reach (HAQ0243) | Reach |
| Grip (HAQ0244) | Grip |
| Common daily activities (HAQ0245) | Common daily activities |

- After these corrections, the highest response within each functional area determines the final score
  of that specific functional area. If no questions within a given functional area were answered, no
  score will be provided for that category (even if answers on aids or equipment are available).
- HAQ-DI is only calculated if there are at least 6 functional area scores available.
- The average of these non-missing functional area scores defines the continuous HAQ-DI score ranging from 0 to 3. If there are less than 6 functional area scores available, no imputation will be done, and the HAQ-DI will be set to missing for the according assessment.

#### 14.6.3.6. CDAI

#### CDAI

#### **CDAI Total Score**

- The Clinical Disease Activity Index (CDAI) is a composite score consisting of the sum of SJC28, TJC28, PtGA and PhGA. Since PtGA and PhGA are both collected on a VAS scale 0-100, the respective scores will be divided by 10 before computing the CDAI total score.
- CDAI ranges from 0 to 76 with higher values representing higher disease activity.

- Individual components collected outside of a +/- 2 day window from visit date will be considered missing for the purpose of the CDAI calculation.
- If one of the components is missing at an individual assessment point the CDAI value for that assessment will be set to missing.

### CDAI Low disease activity (CDAI-LDA)

Low Disease Activity is achieved for a non-missing CDAI total score ≤10.

#### **CDAI Remission**

Remission is achieved for a non-missing CDAI total score ≤2.8.

#### 14.6.3.7. DAS28-CRP and DAS28-ESR

#### DAS28-CRP

#### DAS28-CRP

- The components of the DAS28-CRP arthritis assessment include:
  - Tender Joint Count 28 (TJC28)
  - Swollen Joint Count 28 (SJC28)
  - C-reactive protein (CRP) (in mg/L)
  - o Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=ccl to 100=ccl )
- The DAS28-CRP score will be calculated using the following formula:

#### DAS28-CRP=0.56\*\TJC28+0.28\*\SJC28+0.36\*In(CRP+1)+0.014\*PtGA+0.96

- Individual components collected outside of a +/- 2 day window from visit date will be considered missing for the purpose of the DAS28 calculation.
- If one of the components is missing at an individual assessment point, no imputations will be done and the DAS28 value for that assessment will be set to missing.

#### DAS28-CRP Low disease activity (LDA)

Low Disease Activity is achieved for a DAS28-CRP ≤3.2.

#### **DAS28-CRP Remission**

Remission is achieved for a DAS28-CRP < 2.6</li>

#### DAS28-ESR

#### DAS28-ESR

- The components of the DAS28-ESR arthritis assessment includes:
  - Tender Joint Count 28 (TJC28)
  - Swollen Joint Count 28 (SJC28)
  - Erythrocyte sedimentation rate (ESR) (in mm/hr)
  - o Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=ccl to 100=ccl)
- The DAS28-ESR score will be calculated using the following formula:

#### DAS28(ESR)=0.56\*\(\sqrt{TJC28+0.28\*\sqrt{SJC28+0.7\*In(ESR)+0.014\*PtGA}\)

- Individual components collected outside of a +/- 2 day window from visit date will be considered missing for the purpose of the DAS28 calculation.
- If one of the components is missing at an individual assessment point, no imputations will be done and the DAS28 value for that assessment will be set to missing.
- An ESR value of 0 will be substituted with ESR=1 for the calculation of DAS28(ESR).

#### DAS28-ESR Low disease activity (LDA)

Low Disease Activity is achieved for a DAS28-ESR ≤3.2.

#### **DAS28-ESR Remission**

Remission is achieved for a DAS28-ESR <2.6</li>

#### 14.6.3.8. EULAR Response

#### **EULAR Response**

## **EULAR Good/Moderate Response**

DAS28-CRP and DAS28-ESR scores will each be categorised using EULAR response criteria.
 Response at a given time point is defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to baseline. The definition of no response, moderate response and good response is captured in the following table:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

 If the post-baseline DAS28 value is missing, then the corresponding EULAR category will be set to missing.

#### 14.6.3.9. ACR/EULAR Remission

#### **ACR/EULAR Remission**

#### **Boolean-based ACR/EULAR Remission**

- Boolean-based remission is achieved if all of the following requirements are met at the same time:
  - o TJC68 ≤ 1
  - o SJC66 ≤ 1
  - CRP ≤ 1mg/dl
  - o PtGA ≤ 10
- Individual components collected outside of a +/- 2 day window from visit date will be considered missing for the purpose of the calculation.
- If one of the components is missing at an individual assessment point, the Boolean-based remission for that assessment will be set to missing.

#### Index-based ACR/EULAR Remission

- The Simple Disease Activity Index (SDAI) is a composite score consisting of the sum of SJC28, TJC28, PtGA, PhGA, and CRP (mg/dl). Since PtGA and PhGA are both collected on a VAS scale 0-100, the respective scores will be divided by 10 before computing the SDAI total score.
- Index-based remission is achieved if the following requirement is met:
  - o SDAI ≤ 3.3
- Individual components collected outside of a +/- 2 day window from visit date will be considered missing for the purpose of the calculation.

#### ACR/EULAR Remission

• If one of the components is missing at an individual assessment point, the Index-based remission for that assessment will be set to missing.

# 14.6.3.10. Van der Heijde Modified Total Sharp Score


#### Van der Heijde Modified total Sharp Score (mTSS)

#### Erosion Grading Scheme of the Foot

Similar erosion grading method will be used in the foot as previously described for the hand, except
the scale extends from 0 to 10 per joint. This method gives relatively more weight to the joints of the
feet, because of the higher maximum erosion score.

#### **Total Joint Erosion Score**

- The total joint erosion score will be calculated using a summation of the scores of all locations (both hands and feet) at each time point.
- If an individual location is scored either "Not Assessable" or "Surgically Modified" then the score for that location will be set to missing before calculating the total score.
- If an individual location has a missing score, then the score will be imputed using the average score across all available evaluable locations.
- If data for more than 50% of locations are missing at the time of a given assessment, then the total individual component score will be set to missing for that visit.

## Joint Space Narrowing (JSN) Score

- The JSN score summarizes the severity of JSN in 15 locations in each hand/wrist (30 locations in total) and 6 locations in each foot (12 locations in total).
- Assessment of JSN for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, is scored from 0 to 4, with 0 indicating columns and 4 indicating columns and 4 indicating columns is 168 (120 for both hands/wrists and 48 for both feet) at a time point.
- JSN for each hand and foot joint is graded on the following scale:
   CCI This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

#### Total Joint Space Narrowing Score

- The total joint space narrowing score will be calculated using a summation of the scores of all locations (both hands and feet) at each time point.
- If an individual location is scored either "Not Assessable" or "Surgically Modified" then the score for that location will be set to missing before calculating the total score.
- If an individual location has a missing score, then the score will be imputed using the average score across all available evaluable locations.
- If data for more than 50% of locations are missing at the time of a given assessment, then the total individual component score will be set to missing for that visit.

#### Modified Total Sharp Score (mTSS)

- The total mTSS score at a time point is the sum of the erosion (maximum of 280) and JSN (maximum of 168) scores, for a maximum score of 448.
- The van der Heijde modified sharp scoring method is summarised below:

| | Joint/Bone | Erosion | Joint | JSN |
|------|------------|---------|-------|-----|
| Hand | MCP1 | 0-5 | MCP1 | 0-4 |
| | MCP2 | 0-5 | MCP2 | 0-4 |
| | MCP3 | 0-5 | MCP3 | 0-4 |

| | MCP4 | 0-5 | MCP4 | 0-4 |
|------|--------------------------|-------|------------------------|-------|
| | MCP5 | 0-5 | MCP5 | 0-4 |
| | PIP2 | 0-5 | PIP2 | 0-4 |
| | PIP3 | 0-5 | PIP3 | 0-4 |
| | PIP4 | 0-5 | PIP4 | 0-4 |
| | PIP5 | 0-5 | PIP5 | 0-4 |
| | IP1 | 0-5 | CMC3 | 0-4 |
| | CMC1 | 0-5 | CMC4 | 0-4 |
| | Radius | 0-5 | CMC5 | 0-4 |
| | Ulna | 0-5 | Trapezium-navicular | 0-4 |
| | Multangular bones | 0-5 | Capitate-navicular | 0-4 |
| | Navicular | 0-5 | Radio-carpal | 0-4 |
| | Lunate | 0-5 | | |
| Foot | MTP1 | 0-10 | MTP1 | 0-4 |
| | MTP2 | 0-10 | MTP2 | 0-4 |
| | MTP3 | 0-10 | MTP3 | 0-4 |
| | MTP4 | 0-10 | MTP4 | 0-4 |
| | MTP5 | 0-10 | MTP5 | 0-4 |
| | IP1 Toe | 0-10 | IP1 Toe | 0-4 |
| | Total score one hand | 0-80 | Total score one hand | 0-60 |
| | Total score one foot | 0-60 | Total score one foot | 0-24 |
| | Total score both hands | 0-160 | Total score both hands | 0-120 |
| | Total score both feet | 0-120 | Total score both feet | 0-48 |
| | Score range for erosions | 0-280 | Score range for JSN | 0-168 |
| | Score range mTSS | | | 0-448 |

## 14.6.3.11. SF-36

## **SF-36**

## SF-36

Health-related quality of life will be assessed using the subject-completed Medical Outcomes Study Short-Form 36 (SF-36) which is a generic health survey that contains 36 questions covering eight domains of health. The SF-36 yields an eight-scale profile of functional health and well-being scores as well as physical and mental component health summary scores. The version 2, 1-week recall questionnaire will be used. Recoding, calculations and standardisation will be done using Quality Metrics SF-36 scoring software.

•

## SF-36 Domain Scores

- Individual question responses will be inputted into the Quality Metrics SF-36 scoring software to compute the eight domain scores:
  - Physical functioning (PF)
  - Role function Physical aspect (RP)
  - o Bodily Pain (BP)
  - General health perception (GH)
  - Mental Health (MH)
  - o Role function Emotional aspect (RE)
  - Social functioning (SF)
  - Vitality (VT)
- Higher scores represent better health status.

## SF-36 Physical and Mental component scores

• Individual question responses will be inputted into the Quality Metrics SF-36 scoring software to compute the physical and mental component scores.



## CONFIDENTIAL

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third p | arty |
|---|---|
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third p copyright laws and therefore have been excluded. | |
| CCL - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third of | arty |
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third p copyright laws and therefore have been excluded. | urty |





# 14.6.4. Safety

# **Adverse Events**

# AE event rates per 100 patient-years of exposure

AE event rates per 100 patient-years of exposure will be calculated as:
 (Sum of occurrences of adverse event/ Sum of exposure duration [in years]) \* 100

# Adverse Events of Special Interest (AESI)

# **AEs of Special Interest (AESI)**

 Adverse events of special interest (AESI) and other important adverse events will be derived using MEDRA and Common Terminology Criteria for Adverse Events v5.0 (NCI, 2017) and will include:

| AESI | for Adverse Events v5.0 (NCI, 2017) and will include<br>Programmatical Derivation |
|---|---|
| Serious infections and Serious infections excluding COVID-19 infections | Serious infections: Filter on Infections and Infestations SOC, limited to serious. |
| | Serious infections excluding COVID-19 infections: Filter on Infections and Infestations SOC, limited to serious and exclude the following PTs: Suspected COVID-19", "COVID-19", "COVID-19" pneumonia" or "Asymptomatic COVID-19". |
| Opportunistic infections | Opportunistic infections will be derived using the "Opportunistic infections" (Broad) SMQ and adjudicated by the SRT. Adjudicated opportunistic infections will be summarised. |
| Active TB, latent TB and TB reactivation | Derived from preferred terms of "Tuberculosis". Use HLT: 'Tuberculous Infections'. |
| | All tuberculosis infections will be adjudicated by SRT. The outcome of the adjudication will be Active TB, latent TB, or TB reactivation which will be summarised. |
| Neutropenia | Derived using PT of "Neutropenia" and/or "neutrophil count decreased" and/or "neutrophil percentage decreased". Only AEs/SAEs of neutropenia and/or neutrophil count decreased and/or neutrophil percentage decreased where the corresponding absolute neutrophil count (from laboratory data) are CTCAE grade 3 or 4 will be reported as AESI. |
| Persistent Cough | Cough CTCAE ≥ Grade 2 recorded for 3 consecutive weeks (≥21 Days). |
| | Identified from: Cough 'Yes' entered in the eCRF with Grade determined from AE reporting with the following definition: CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |

| Persistent dyspnoea | Persistent dyspnoea grade ≥ 2 for three consecutive weeks (≥21 days). |
|---|---|
| | Identified from: |
| | Dyspnoea rating scale on the pulmonary assessment eCRF page with the following grading: |
| | CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
| PAP (Pulmonary alveolar proteinosis) | Derived using preferred term (PT) "alveolar |
| | proteinosis'. (LLT of 'pulmonary alveolar proteinosis' maps to PT of 'alveolar proteinosis'). All cases adjudicated by Pulmonary Adjudication Committee (PAC). |
| | The adjudicated PAP outcome will be summarised. |
| Serious Hypersensitivity reactions, including anaphylaxis | Serious hypersensitivity reactions will be adjudicated using "Hypersensitivity" (Broad) SMQ, 'Anaphylactic reaction' (Broad) SMQ and 'anaphylactic/anaphylactoid shock condition' (Broad) SMQ based on SAE listings. |
| | Final adjudication will be conducted by SRT and the adjudicated hypersensitivity reactions will be summarised. |
| Injection site reactions | Derived from HLT term "injection site reactions", HLT term "administration site reaction NEC" and PT term "injection related reaction". |

#### Other Important AEs

#### Protocol defined cardiovascular (CV) events and adjudicated CV events

#### CV Events

CV events as reported in the database will be included in the summary table for all AEs.

#### Adjudicated CV Events

Endpoints of interest: cardiovascular (CV) death, myocardial infarction (MI), hospitalisation for unstable angina, stroke, hospitalisation for heart failure, deep vein thrombosis (DVT) and pulmonary embolism (PE). These will be derived using PT terms listed in clinical events classification (CEC) Charter and adjudicated by Duke Clinical Research Institute (DCRI) CEC group. Adjudicated CV endpoints will be summarised.

Adjudicated CV Events will also be reported as the following categories:

- o MACE: CV death, non-fatal MI, non-fatal stroke
- Broad MACE: CV death, MI, hospitalisation for unstable angina, stroke and hospitalisation for heart failure.
- VTE (DVT and/or PE)
- o DVT only
- PE only

#### Note:

- CV categories include both fatal and non-fatal events.
- Fatal CV events will be captured in two categories, respective CV category and CV death.
- A subject can have an event in more than one category.
- CV death includes death due to CV causes (cardiogenic shock, HF, arrhythmia/sudden death, MI, cardiac rupture, ischemic stroke, PE, venous/arterial thrombotic events) and any other unobserved deaths for which an alternative cause has not been identified
- In the broad MACE category, if a subject has a CV event that resulted in death, it will only be counted as one MACE event. This will be derived by cross referencing the adjudication outcomes with the outcomes of the CV event reported by the investigator.

#### GI Perforation and Adjudicated GI perforation

## GI perforation Events

GI perforation events as reported in the database will be included in the summary table for all AEs.

## • Adjudicated GI perforation

This will be adjudicated by CEC. Data reported in EDC and the adjudicated GI Perforation will be used in the outputs.

#### Malignancy

- Malignancies will be reported as the following categories:
  - Any Malignancy derived from the preferred terms in the below SMQs.
    - Solid, excluding non-melanoma skin cancer (NMSC) derived from Non-haematological malignant tumours (SMQ) and Non-haematological tumours of unspecified malignancy (SMQ) and excluding NMSC terms identified below
    - NMSC PTs derived from Skin neoplasms, malignant and unspecified (SMQ):
      - Atypical fibroxanthoma
      - Basal cell carcinoma
      - Basosquamous carcinoma of skin
      - Bowen's disease
      - Carcinoma in situ of skin
      - Keratoacanthoma
      - Marjolin's ulcer

#### Other Important AEs

- Skin squamous cell carcinoma metastatic
- Skin squamous cell carcinoma recurrent
- Squamous cell carcinoma of skin
- Hematologic derived from Haematological malignant tumours (SMQ) and Haematological tumours of unspecified malignancy (SMQ)
- Lymphoma derived from Malignant Lymphomas (broad SMQ)

#### **Herpes Infections**

- Derived from HLT term "Herpes Viral Infections" excluding the following terms: Human herpesvirus 6 encephalitis, Human herpesvirus 6 infection, Human herpesvirus 7 infection, Human herpesvirus 8 infection, Exanthema subitum
- They will be further categorised as Herpes Zoster, Herpes Simplex and Non-Specific using preferred terms from the most recent version of MedDRA at the time of reporting.

## **All-Cause Mortality**

Any SAE with a fatal outcome

#### **Serious Pulmonary infections**

Any SAE in HLGT "respiratory tract infections"

# Serious Pulmonary infections excluding COVID-19 Infections

 Any SAE in HLGT "respiratory tract infections" excluding the following PTs: Suspected COVID-19", "COVID-19", "COVID-19 pneumonia" or "Asymptomatic COVID-19".

## Pneumonia (serious and non-serious)

Derived from Infective pneumonia (narrow SMQ)

## Pneumonia (serious and non-serious) excluding COVID-19 Infections

 Derived from Infective pneumonia (narrow SMQ) excluding the following PTs: Suspected COVID-19", "COVID-19", "COVID-19 pneumonia" or "Asymptomatic COVID-19".

#### **Hepatitis B and Hepatitis B Reactivation**

AEs and SAEs using PTs 'hepatitis B' and 'hepatitis B reactivation'

#### Thromboembolic events

AEs and SAEs using 'Embolic and thrombotic events' (Broad) SMQ

## **COVID-19 Infections and Adjudicated COVID-19 Infections**

COVID-19 Infections

COVID-19 infections will be derived from the following PTs: "Suspected COVID-19", "COVID-19", "COVID-19". "COVID-19".

All events will be split into serious or non-serious based on how they are reported i.e. all COVID-19 SAEs will be categorised as serious and all COVID-19 AEs will be categorised as non-serious. Non-serious cases of COVID-19 will be split into confirmed, suspected or probable cases based on the eCRF and cases for each category will be displayed.

The serious adverse events of COVID-19 will be adjudicated by PAC and only the adjudicated events summarised.

Adjudicated COVID-19 Infections

Each case that is adjudicated to confirmed case of COVID-19 or probable case of COVID-19 will also be assigned a grade based on World Health Organisation (WHO) original scale.

All adjudicated confirmed cases of COVID-19 and all adjudicates probable cases of COVID-19 will be split into 3 categories (see the categorisation below) and cases for each category will be summarised:

Non hospitalised includes the following WHO grades: grade 1-no limitation of activity and grade
 2-limation of activity.

#### Other Important AEs

- Hospitalised includes the following WHO grades: grade 3-no oxygen therapy; grade 4-low-flow oxygen by mask or nasal prongs; grade 5-high-flow oxygen (≥15L/min), CPAP, BIPAP, non-invasive ventilation; grade 6- intubation and mechanical ventilation and grade 7- mechanical ventilation plus additional organ support (ECMO and vasopressors).
- Death

## **Laboratory Parameters**

#### **eGFR**

• This will be provided in the dataset by Q<sup>2</sup>

#### **Laboratory Results**

If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

- Example 1: 2 Decimal Places= '< x ' becomes x 0.01</li>
- Example 2: 1 Decimal Place= '> x' becomes x + 0.1
- Example 3: 0 Decimal Places= '< x' becomes x − 1

#### **Immunogenicity**

- Positive binding antibody assay results are to be categorised as transient positive or persistent positive accordingly to the following definitions:
- For all post-baseline visits, other than final study assessment
  - Transient positive = a single positive immunogenic response at a visit, where the previous visit was negative
  - Persistent positive = a positive immunogenic response at a visit, where the previous visit was also positive

# 14.7. Appendix 7: Reporting Standards for Missing Data

# 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all phases of the study including the follow up.</li> <li>Withdrawn subjects were not replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |
| | If a scheduled visit and an EW visit occur within the same visit window and are both available, the scheduled visit will be used for any summaries/analyses. The EW visit will appear in listing only. |
| | • For efficacy analyses, if an EW visit is assigned to a non-standard efficacy visit, i.e., a visit at which efficacy assessments are not scheduled per the Time and Events Table, then these EW data will be ignored in the statistical analysis, but all data will be listed. |

# 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Adverse<br>Events | AEs with missing intensity will be considered as severe. |

# 14.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>Although every effort will be made to prevent and eliminate partial dates, the eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| RA diagnosis<br>and<br>symptom<br>onset | <ul> <li>Missing day, but month and year present: <ul> <li>Date is set to the first day of the month (e.g., XX-Sep-2010 is considered as 01-Sep-2010).</li> </ul> </li> <li>Missing day and month, but year present: <ul> <li>Date is set to 01 January (e.g., XX-XXX-2010 is considered as 01-Jan-2010)</li> </ul> </li> </ul> |

# 14.7.2.2. Handling of Missing Efficacy Data

Unless otherwise stated, apply the missing data imputation strategies detailed in Section 7.1.1.6 and Section 7.2.1.6.

# 14.8. Appendix 8: Values of Potential Clinical Importance

# 14.8.1. Laboratory Values Gradings

Laboratory value gradings will be derived using the most recent version of CTCAE at the time of reporting.

# 14.8.2. Laboratory Values of Potential Clinical Importance

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Ratio of | Male | 0.2 | 0.6 |
| | | Female | 0.2 | 0.6 |
| Hematocrit | | Change<br>from<br>baseline | ↓0.075 | |
| | g/L | Male | 80 | 180 |
| | | Female | 80 | 180 |
| Hemoglobin | | Change<br>from<br>baseline | ↓20 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.75 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.0 | 16 |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 2.0 | 20 |
| Eosinophils | x10 <sup>9</sup> / L | | | 1 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | 55 |
| Calcium | mmol/L | | 2 | 2.75 |
| | µmol/L | | | 150 |
| Creatinine | µmol/L | Change<br>from<br>baseline | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 11 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 160 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| GFR from Creatinine<br>Adjusted for BSA | mL/min/1.73<br>m <sup>2</sup> | | 60 | |
| Cholesterol | mmol/L | | | 6.5 |
| Triglycerides | mmol/L | | | 2.3 |
| Urea | mmol/L | | | 10.5 |

| Liver Function | | | |
|----------------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| Creatinine Kinase | U/L | High | ≥ 2x ULN |
| Gamma Glutamyl Transferase | U/L | High | ≥ 2x ULN |
| Lactate Dehydrogenase | U/L | High | ≥ 2x ULN |

| Urinalysis | |
|----------------------------|------------------------|
| Test Analyte | Clinical Concern Range |
| Bacteria | Moderate |
| Bacteria | Many |
| Caucamous Enithelial Colle | Moderate (6-20) |
| Squamous Epithelial Cells | Many (21 or greater) |
| | 1+ OR 1/4 G/DL (%) |
| Glucose | 2+ OR 1/4 G/DL (%) |
| Gladode | |
| | 3+ OR 1/4 G/DL (%) |
| | 4. |
| Doctor | 1+ |
| Protein | 2+ |
| | 3+ |
| | 10-15 |
| | 12-25 |
| Erythrocytes | 25-50 |
| | 50-100 |
| | >100 |
| | 10-15 |
| Leukocytes | 12-25 |
| | 25-50 |

| Urinalysis | |
|--------------|------------------------|
| Test Analyte | Clinical Concern Range |
| | 50-100 |
| | >100 |
| Veest Calle | Moderate |
| Yeast Cells | Many |

For the listing of Laboratory Data for Subjects with any value of Potential Clinical Important, only include the following laboratory data:

- Alanine Aminotransferase
- Albumin
- Albumin/Globulin
- Alkaline Phosphate
- Aspartate Aminotransferase
- Basophils
- Bilirubin
- C Reactive Protein
- Calcium
- Cholesterol
- Creatinine Kinase
- Creatinine
- Cyclic Citrullinated Peptide Antibody
- Direct Bilirubin
- Eosinophils
- Erythrocyte Sedimentation Rate
- Erythrocytes
- GFR from Creatinine Adjusted for BSA
- Gamma Glutamyl Transferase
- Glucose
- HDL Cholesterol, Direct
- Hematocrit
- Hemoglobin
- Hepatitis B Core Antibody Total, Qual
- Hepatitis B Virus DNA
- Hepatitis B Virus DNA, copies
- Hepatitis B Virus DNA, log
- Hepatitis B Virus Surface Antibody, Qual
- Hepatitis B Virus Surface Antigen, Qual
- Hepatitis C Antibody, Qual
- Hepatitis C Virus RNA
- Hepatitis C Virus RNA, log
- Interferon Gamma, Qualitative
- LDL Cholesterol
- Lactate Dehydrogenase

- Leukocytes
- Lymphocytes
- Monocytes
- Neutrophils
- Platelets
- Potassium
- Protein
- Prothrombin Intl. Normalized Ratio
- Reticulocytes/Erythrocytes
- Rheumatoid Factor
- Theophylline
- Triglycerides
- Urea

# 14.8.3. ECG Values of Potential Clinical Importance

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | >450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >30↑ |

# 14.8.4. Vital Signs Values of Potential Clinical Importance

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
| Change from Baseline | | | |
| Systolic Blood Pressure | mmHg | ≥ 20↓ | ≥ 20↑ |
| Diastolic Blood Pressure | mmHg | ≥ 10↓ | ≥ 10↑ |
| Heart Rate | bpm | ≥ 15↓ | ≥ 15↑ |

# 14.9. Appendix 9: List of Preferred Terms

## 14.9.1. Herpes Zoster

Adjudication by GSK SRT will identify events that are recurrent or disseminated. Herpes Zoster is considered disseminated if there is involvement of other organs other than the skin or if skin lesions (1) cross the midline of the body or (2) are in non-adjacent dermatomes or (3) are located in more than three adjacent dermatomes. Herpes zoster is considered an opportunistic infection if it is adjudicated as recurrent or disseminated. However, there may be some uncommon occurrences of a herpes zoster case that is adjudicated as an OI but is neither recurrent nor disseminated.

## 14.9.2. Mycobacterium Tuberculosis

Tuberculosis (TB) cases are reviewed by the GSK SRT to determine if a case is an OI. The following principles are applied: Pulmonary TB in an endemic area is not considered an OI. Pulmonary TB in a non-endemic area would be considered an OI unless the participant had close contact with a person infected with TB. Extra pulmonary TB is generally considered an OI unless the affected extra pulmonary area followed a wound or trauma.

## 14.10. Appendix 10: Missing Data Imputation Strategies

## 14.10.1. Primary Estimand Strategy

## 14.10.1.1. Multiple Imputation using off-treatment data within treatment arm

- 1. Exclude week 1 data and participants with missing baseline values.
- 2. Generate 1000 multiply imputed datasets using a monotone logistic imputation with augmentation (binary endpoints) or a monotone regression imputation (continuous endpoints) including terms for baseline value, all previous visit values, treatment group, treatment discontinuation and treatment group-by-treatment discontinuation interaction, i.e. a model of the form  $y_i = \alpha_{1i} + \alpha_{2i}base + \alpha_{3i}TD_i + \alpha_{4i}trt + \alpha_{5i}(trt * TD_i) + \beta_{i-1}y_{i-1} + \cdots + \beta_1y_1$  where  $y_i$  is the result at visit i and  $TD_i$  is the treatment discontinuation indicator at visit i.
- 3. Perform statistical analysis as detailed in Section 7.1.3 and Section 7.2.3.

#### 14.10.1.2. Multiple Imputation using off-treatment data across all treatment arms

- 1. Exclude week 1 data and participants with missing baseline values.
- 2. Generate 1000 multiply imputed datasets using a monotone logistic imputation with augmentation (binary endpoints) or monotone regression imputation (continuous endpoints) including terms for baseline value, all previous visit values, treatment group and treatment discontinuation, i.e. a model of the form

 $y_i = \alpha_{1i} + \alpha_{2i}base + \alpha_{3i}TD_i + \alpha_{4i}trt + \beta_{i-1}y_{i-1} + \cdots + \beta_1y_1$ where  $y_i$  is the result at visit i and  $TD_i$  is the treatment discontinuation indicator at visit i.

3. Perform statistical analysis as detailed in Section 7.1.3 and Section 7.2.3.

#### 14.10.1.3. Multiple imputation under MAR assumption

- 1. Exclude week 1 data and participants with missing baseline values.
- 2. Generate 1000 multiply imputed datasets using a monotone logistic imputation with augmentation (binary endpoints) or monotone regression imputation (continuous endpoints) including terms for baseline value, all previous visit values, and treatment group, i.e. a model of the form

$$y_i = \alpha_{1i} + \alpha_{2i}base + \alpha_{3i}trt + \beta_{i-1}y_{i-1} + \dots + \beta_1y_1$$
 where  $y_i$  is the result at visit  $i$ .

3. Perform statistical analysis as detailed in Section 7.1.3 and Section 7.2.3.

# 14.10.2. Supplemental Estimand 1 Strategy

- 1. Impute all data for each visit following the intercurrent event for categorical variables to be non-response.
- 2. Exclude week 1 data and participants with missing baseline values.
- 3. In order to impute intermittent missing data, generate 1000 multiply imputed datasets using a monotone logistic imputation with augmentation (binary endpoints) or monotone regression imputation (continuous endpoints) including

terms for baseline value, all previous visit values, and treatment group, i.e. a model of the form

$$y_i = \alpha_{1i} + \alpha_{2i}base + \alpha_{3i}trt + \beta_{i-1}y_{i-1} + \dots + \beta_1y_1$$
 where  $y_i$  is the result at visit  $i$ 

4. Perform statistical analysis as detailed in Section 7.1.3 and Section 7.2.3.

## 14.10.3. Supplemental Estimand 2 Strategy

- 1. Set all data at each visit following the intercurrent event to missing.
- 2. Exclude week 1 data and participants with missing baseline values.
- 3. Generate 1000 multiply imputed datasets using a monotone logistic imputation with augmentation (binary endpoints) or monotone regression imputation (continuous endpoints) including terms for baseline value, all previous visit values, and treatment group, i.e. a model of the form

$$y_i = \alpha_{1i} + \alpha_{2i}base + \alpha_{3i}trt + \beta_{i-1}y_{i-1} + \dots + \beta_1y_1$$
 where  $y_i$  is the result at visit  $i$ 

4. Perform statistical analysis as detailed in Section 7.1.3 and Section 7.2.3.

# 14.10.4. Intermittent Missing Data Multiple Imputation

Under the primary estimand strategy detailed in Section 14.10.1, in the absence of a treatment discontinuation flag at a particular visit, the models will all reduce to a model of the form:

$$y_i = \alpha_{1i} + \alpha_{2i}base + \alpha_{3i}trt + \beta_{i-1}y_{i-1} + \dots + \beta_1y_1$$

where  $y_i$  is the result at visit i, which will satisfy an MAR assumption for intermittent missing data.

Under the supplemental estimand 1 strategy detailed in Section 14.10.2, intermittent missing data will be imputed separately under an MAR assumption.

Under the supplemental estimand 2 strategy detailed in Section 14.10.3, all data, including intermittent missing data, is imputed under an MAR assumption.

# 14.11. Appendix 11: Abbreviations & Trade Marks

# 14.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AAC | All Analysis Complete |
| ACR | American College of Rheumatology |
| ADA | Anti-Drug Antibodies |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | |
| | And verse Event of Special Interest |
| ANCOVA | Analysis of Covariance |
| bDMARD | Biologic Disease-Modifying Anti-Rheumatic Drug |
| BID | Twice a day |
| BMI | Body Mass Index |
| boDMARD | Biological Originator Disease-Modifying Antirheumatic Drug |
| bsDMARD | Biosimilar Disease-Modifying Antirheumatic Drug |
| CDAI | Clinical Disease Activity Index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CIRT | Cenduit Interactive Response Technology |
| CRP | C-Reactive Protein |
| csDMARD | Conventional Synthetic Disease Modifying Antirheumatic Drug |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | Cardiovascular |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DAS | Disease Activity Score |
| DBF | Database Freeze |
| DBR | Database Release |
| DMARD | Disease-Modifying Antirheumatic Drug |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| ESR | Erythrocyte Sedimentation Rate |
| EULAR | European League Against Rheumatism |
| EW | Early Withdrawal |
| FACIT | Functional Assessment of Chronic Illness Therapy - Fatigue |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GM-CSF | Granulocyte-Macrophage Colony-Stimulating Factor |
| GSK | GlaxoSmithKline |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| HDL | Headline Results |
| ICH | International Conference on Harmonization |
| 1011 | international conference on Harmonization |

| Abbreviation | Description |
|--------------|-------------------------------------------------------------|
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IE | Intercurrent Event |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| IWRS | Interactive Web Response System |
| JAKi | Janus Kinase Inhibitor |
| LDA | Low Disease Activity |
| LLOQ | Lower Limit of Quantification |
| LS | Least Squares |
| MACE | Major Adverse Cardiovascular Event |
| MAR | Missing at Random |
| MCID | Minimum Clinically Important Different |
| MCMC | Markov Chain Monte Carlo |
| MCS | Mental Component Score |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| MMRM | Mixed Model Repeated Measures |
| mTSS | Modified Total Sharp Score |
| MTX | Methotrexate |
| NQ | Non-quantifiable |
| NRS | Numerical Rating Scale |
| OR | Odds Ratio |
| PAP | Pulmonary Alveolar Proteinosis |
| PCI | Potential Clinical Importance |
| PCS | Physical Component Score |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PhGA | Physician's Global Assessment of Arthritis Disease Activity |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| PRO | Patient Reported Outcome |
| CCI | |
| PT | Preferred Term |
| PtGA | Patient's Global Assessment of Arthritis Disease Activity |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| QW | Every Week |
| Q2W | Every 2 Weeks |
| RA | Rheumatoid Arthritis |
| RAP | Reporting & Analysis Plan |
| CCI | |
| RF | Rheumatoid Factor |

| Abbreviation | Description |
|--------------|---------------------------------------------------------|
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Events |
| SC | Subcutaneous |
| SDTM | Study Data Tabulation Model |
| SF-36 | 36-Item Short Form Survey |
| SJC | Swollen Joint Count |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| SRT | Safety Review Team |
| TA | Therapeutic Area |
| TB | Mycobacterium Tuberculosis |
| TEAE | Treatment Emergent Adverse Event |
| TFL | Tables, Figures & Listings |
| TJC | Tender Joint Count |
| tsDMARD | Targeted Synthetic Disease Modifying Antirheumatic Drug |
| VAS | Visual Analog Scale |
| WOCBP | Woman of Childbearing Potential |
| WPMI | Within Patient Meaningful Improvement |

# 14.11.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |



# 14.12. Appendix 12: List of Data Displays

All data displays will use the term "subject" rather than "participant" in accordance with CDSIC and GSK Statistical Display Standards.

# 14.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------|------------------|----------------|
| Study Population | 1.1 to 1.30 | 1.1 to 1.2 |
| Japan Study Population | 1.301 to 1.307 | - |
| China Study Population | 1.401 to 1.414 | 1.401 |
| Asia Study Population | 1.501 to 1.508 | - |
| Efficacy | 2.1 to 2.95 | 2.1 to 2.80 |
| Japan Efficacy | 2.301 to 2.320 | - |
| China Efficacy | 2.401 to 2.427 | 2.401 to 2.404 |
| Asia Efficacy | 2.501 to 2.508 | 2.501 |
| Safety | 3.1 to 3.137 | 3.1 to 3.7 |
| Japan Safety | 3.301 to 3.336 | - |
| China Safety | 3.401 to 3.420 - | |
| Asia Safety | 3.501 to 3.512 - | |
| ·CCI | | |
| Japan Pharmacokinetic | 4.301 to 4.302 | - |
| China Pharmacokinetic | 4.401 to 4.402 | - |
| Asia Pharmacokinetic | 4.501 to 4.502 | - |
| CCI | | |
| Section | Listings | |
| ICH Listings | 1 to 14 | |
| Other Listings | 15 to 45 | |

## 14.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in the final version of this document.

## 14.12.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------|
| HDL [1] | Headline Results Complete |
| SAC[2] | Statistical Analysis Complete |
| AAC [3] | All Analysis Complete |
| Asia AAC [4] | Asia All Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# **Study Population Tables**

| | IDSL/ | | | | |
|---|---|---|---|---|---|
| No. | Population | Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ct Disposition | | | | |
| 1.1. | Randomised | Non-<br>Standard<br>POP_T1<br>(Based on<br>ES1) | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT<br>Include Total Column | SAC[2] |
| 1.2. | Randomised | Non-<br>Standard<br>POP_T1<br>(Based on<br>ES1) | Summary of Subject Status and Subject Disposition for Withdrawals due to COVID-19 Pandemic | Only include: • Related to COVID-19 Pandemic This information should be gathered from COVID-19 impact form in eCRF. Include Total Column | SAC[2] |
| 1.3. | Randomised | Non-<br>Standard<br>POP_T2<br>(Based on<br>SD1) | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3<br>Include Total Column | SAC[2] |
| 1.4. | Randomised | Non-<br>Standard<br>POP_T2<br>(Based on<br>SD1) | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment due to COVID-19 Pandemic | Only include: • Related to COVID-19 Pandemic This information should be gathered from COVID-19 impact form in eCRF. Include Total Column | SAC[2] |

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.5. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC[2] |
| 1.6. | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID by Implementation of Pandemic Measures | EudraCT/Clinical Operations Summarise by: Overall Before Implementation of Pandemic Measures After Implementation of Pandemic Measures | SAC[2] |
| Protoc | ol Deviation | | | | |
| 1.7. | ITT | DV1 | Summary of Important Protocol Deviations | ICH E3 Only categories are to be reported in the table. | SAC[2] |
| 1.8. | ITT | DV1 | Summary of Important Protocol Deviations Related to the COVID-19 Pandemic | Only include: • Important related to COVID- 19 Pandemic Only categories are to be reported in the table. | SAC[2] |

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | tion Analysed | | | | |
| 1.9. | Screened | SP1 | Summary of Study Populations | IDSL | SAC[2] |
| 1.10. | Enrolled | SP2 | Summary of Protocol Deviations Leading to Exclusion from the Per Protocol Population(s) | IDSL Include total column. Only categories are to be reported in the table. | SAC[2] |
| Demog | raphic and Bas | seline Characte | eristics | 1 | |
| 1.11. | ITT | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT<br>Add BMI to the output. | HDL[1] |
| 1.12. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC[2] |
| 1.13. | ITT | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC[2] |
| 1.14. | ITT | Non-<br>Standard<br>POP_T3 | Summary of Baseline Efficacy Parameters | Include all efficacy endpoints | HDL[1] |
| 1.15. | ITT | Non-<br>Standard<br>POP_T4 | Summary of Rheumatoid Arthritis Disease History | | HDL[1] |
| 1.16. | ITT | Non-<br>Standard<br>POP_T5 | Summary of History of Tobacco Use and Family History of Cardiovascular Risk Factors | Display by Overall, Age <50 and Age>=50 | SAC[2] |

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitar | nt Medications | | | |
| 1.17. | ITT | AE1 | Summary of Medical Conditions | ICH E3 Include Preferred Terms. | SAC[2] |
| 1.18. | ITT | Non-<br>Standard<br>POP_T6 | Summary of RA Concomitant Medications | Include Total Column. | SAC[2] |
| 1.19. | ITT | CM1 | Summary of All Concomitant Medications | ICH E3 | SAC[2] |
| 1.20. | ITT | Non-<br>Standard<br>POP_T7 | Summary of RA Prior Medications | Include Total Column. | SAC[2] |
| 1.21. | ITT | CM1 | Summary of All Prior Medications | Include Total Column. | SAC[2] |
| 1.22. | ITT | Non-<br>Standard<br>POP_T8 | Summary of RA Medications taken at Baseline (Day 1) | Include Total Column. | SAC[2] |
| 1.23. | ITT | Non-<br>Standard<br>POP_T9 | Summary of Concomitant COVID-19 Vaccines | Include Total Column. | SAC[2] |
| Exposu | re and Treatmer | nt Compliance | | | |
| 1.24. | Safety | Non-<br>Standard<br>POP_T10 | Summary of Exposure to Study Treatment | ICH E3<br>Include Total Column. | SAC[2] |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.25. | Safety | Non-<br>Standard<br>POP_T11 | Summary of Overall Compliance Based on Exposure | Display for compliance with both injections and capsules Include Total Column. | SAC[2] |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| COVID | -19 | | | | |
| 1.26. | ITT | PAN4 | Summary of COVID-19 Visit Impacts | | SAC[2] |
| 1.27. | ITT | DM1 | Summary of Demographic Characteristics by Pre and Post Pandemic Measures | Summarise by: Before Implementation of Pandemic Measures After Implementation of Pandemic Measures | SAC[2] |
| Explora | atory: Pain DE | TECT | | | |
| Tables | for Disclosure | | | | |
| 1.29. | Randomised | Non-<br>Standard<br>POP_T1 | Summary of Subject Disposition for the Subject Conclusion Record (by Randomised Treatment Arm) | Display by randomised treatment arm (i.e. all 6 treatment arms) | AAC[3] |
| 1.30. | ΙΤΤ | DM1 | Summary of Demographic Characteristics (by Randomised Treatment Arm) | Display by randomised treatment arm (i.e. all 6 treatment arms) | AAC[3] |
| Japan | Subgroup | | | | |
| 1.301. | Japanese<br>Randomised | Non-<br>Standard<br>POP_T1<br>(Based on<br>ES1) | Summary of Subject Disposition for the Subject Conclusion Record for Japanese Subjects | Include Total Column. | Asia AAC[4] |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.302. | Japanese<br>ITT | DM1 | Summary of Demographic Characteristics for Japanese Subjects | | Asia AAC[4] |
| 1.303. | Japanese<br>ITT | Non-<br>Standard<br>POP_T3 | Summary of Baseline Efficacy Parameters for Japanese Subjects | Include Total Column. | Asia AAC[4] |
| 1.304. | Japanese<br>ITT | Non-<br>Standard<br>POP_T4 | Summary of Rheumatoid Arthritis Disease History for Japanese Subjects | Include Total Column. | Asia AAC[4] |
| 1.305. | Japanese<br>ITT | Non-<br>Standard<br>POP_T8 | Summary of RA Medications taken at Baseline (Day 1) for Japanese Subjects | Include Total Column. | Asia AAC[4] |
| 1.306. | Japanese<br>Safety | Non-<br>Standard<br>POP_T10 | Summary of Exposure to Study Treatment for Japanese Subjects | Include Total Column. | Asia AAC[4] |
| 1.307. | Japanese<br>Safety | Non-<br>Standard<br>POP_T11 | Summary of Overall Compliance Based on Exposure for Japanese Subjects | Include Total Column. | Asia AAC[4] |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| China | China Subgroup | | | | |
| 1.401. | Chinese<br>Randomised | Non-<br>Standard<br>POP_T1<br>(Based on<br>ES1) | Summary of Subject Disposition for the Subject Conclusion Record for Chinese Subjects | Include Total Column. | Asia AAC[4] |
| 1.402. | Chinese<br>Randomised | Non-<br>Standard<br>POP_T2<br>(Based on<br>SD1) | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment for Chinese Subjects | Include Total Column | Asia AAC[4] |
| 1.403. | Chinese<br>ITT | DV1 | Summary of Important Protocol Deviations for Chinese Subjects | Only categories are to be reported in the table. | Asia AAC[4] |
| 1.404. | Chinese<br>Screened | SP1 | Summary of Study Populations for Chinese Subjects | | Asia AAC[4] |
| 1.405. | Chinese<br>ITT | DM1 | Summary of Demographic Characteristics for Chinese Subjects | | Asia AAC[4] |
| 1.406. | Chinese<br>ITT | Non-<br>Standard<br>POP_T3 | Summary of Baseline Efficacy Parameters for Chinese Subjects | Include Total Column. | Asia AAC[4] |
| 1.407. | Chinese<br>ITT | Non-<br>Standard<br>POP_T4 | Summary of Rheumatoid Arthritis Disease History for Chinese Subjects | Include Total Column. | Asia AAC[4] |

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.408. | Chinese<br>ITT | AE1 | Summary of Medical Conditions for Chinese Subjects | Include Preferred Terms. | Asia AAC[4] |
| 1.409. | Chinese<br>ITT | Non-<br>Standard<br>POP_T6 | Summary of RA Concomitant Medications for Chinese Subjects | Include Total Column. | Asia AAC[4] |
| 1.410. | Chinese<br>Safety | Non-<br>Standard<br>POP_T10 | Summary of Exposure to Study Treatment for Chinese Subjects | Include Total Column. | Asia AAC[4] |
| 1.411. | Chinese<br>Randomised | Non-<br>Standard<br>POP_T1<br>(Based on<br>ES1) | Summary of Subject Status and Subject Disposition for Withdrawals due to COVID-19 Pandemic for Chinese Subjects | Only include: Related to COVID-19 Pandemic This information should be gathered from COVID-19 impact form in eCRF. Include Total Column | Asia AAC[4] |
| 1.412. | Chinese<br>Randomised | Non-<br>Standard<br>POP_T2<br>(Based on<br>SD1) | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment due to COVID-19 Pandemic for Chinese Subjects | Only include: Related to COVID-19 Pandemic This information should be gathered from COVID-19 impact form in eCRF. Include Total Column | Asia AAC[4] |
| 1.413. | Chinese<br>ITT | DV1 | Summary of Important Protocol Deviations Related to the COVID-19 Pandemic for Chinese Subjects | Only include: • Important related to COVID- 19 Pandemic Only categories are to be reported in the table. | Asia AAC[4] |

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.414. | Chinese<br>ITT | PAN4 | Summary of COVID-19 Visit Impacts for Chinese Subjects | | Asia AAC[4] |
| Asia S | ubgroup | | | | |
| 1.501. | Asia<br>Randomised | Non-<br>Standard<br>POP_T1<br>(Based on<br>ES1) | Summary of Subject Disposition for the Subject Conclusion Record for Asia Subjects | Include Total Column. | Asia AAC[4] |
| 1.502. | Asia<br>ITT | DV1 | Summary of Important Protocol Deviations for Asia Subjects | Only categories are to be reported in the table. | Asia AAC[4] |
| 1.503. | Asia<br>Screened | SP1 | Summary of Study Populations for Asia Subjects | | Asia AAC[4] |
| 1.504. | Asia<br>ITT | DM1 | Summary of Demographic Characteristics for Asia Subjects | | Asia AAC[4] |
| 1.505. | Asia<br>ITT | Non-<br>Standard<br>POP_T3 | Summary of Baseline Efficacy Parameters for Asia Subjects | Include Total Column. | Asia AAC[4] |
| 1.506. | Asia<br>ITT | Non-<br>Standard<br>POP_T4 | Summary of Rheumatoid Arthritis Disease History for Asia Subjects | Include Total Column. | Asia AAC[4] |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.507. | Asia<br>ITT | Non-<br>Standard<br>POP_T6 | Summary of RA Concomitant Medications for Asia Subjects | Include Total Column. | Asia AAC[4] |
| 1.508. | Asia<br>Safety | Non-<br>Standard<br>POP_T10 | Summary of Exposure to Study Treatment for Asia Subjects | Include Total Column. | Asia AAC[4] |

# **Study Population Figures**

# **Efficacy Tables**

| Study Population Figures | | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| Subjec | t Disposition | | | | | |
| 1.1. | Randomised | PAN6 | Plot of Recruitment over time by Country Relative to COVID-19 Pandemic Measures | | SAC[2] | |
| COVID | -19 | | | | | |
| 1.2. | ITT | PAN8 | Plot of Visits Impacted by COVID-19 Pandemic | | SAC[2] | |
| China S | Subgroup | | | | | |
| 1.401 | Chinese<br>ITT | PAN8 | Plot of Visits Impacted by COVID-19 Pandemic for Chinese Subjects | | Asia AAC[4] | |
| Efficac | y: Tables | | | | | |
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| ACR20 | | | | | | |
| 2.1. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each Assessment Visit (Primary Estimand) | | HDL[1] | |
| 2.2. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each Assessment Visit (Supplemental Estimand 1) | | SAC[2] | |
| Efficac | Efficacy: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 2.3. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each Assessment Visit (Supplemental Estimand 2) | | AAC[3] | | | |
| 2.4. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR20 Response at Each Assessment Visit | | SAC[2] | | | |
| CDAI-L | DA | | | | | | | |
| 2.5. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit (Primary Estimand) | | HDL[1] | | | |
| 2.6. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit (Supplemental Estimand 1) | | SAC[2] | | | |
| 2.7. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit | | SAC[2] | | | |
| HAQ-D | )[ | | | | | | | |
| 2.8. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) | | HDL[1] | | | |
| 2.9. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in HAQ-DI<br>Score and in Functional Areas of the HAQ-DI Score at<br>Each Assessment Visit | | SAC[2] | | | |

| Efficad | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CDAI | Total Score | | | | |
| 2.10. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in CDAI Total score at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| 2.11. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in CDAI Total score at Each Assessment Visit (Supplemental Estimand 2) | | AAC[3] |
| 2.12. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in CDAI Total Score at Each Assessment Visit | | SAC[2] |
| FACIT | -Fatigue | | | | • |
| 2.13. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in FACIT-Fatigue at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| 2.14. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in FACIT-<br>Fatigue at Each Assessment Visit | | SAC[2] |
| Arthrit | is Pain VAS | | | | • |
| 2.15. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Arthritis Pain VAS Score at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| 2.16. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Arthritis Pain VAS<br>Score at Each Assessment Visit (Supplemental Estimand<br>2) | | AAC[3] |
| 2.17. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Arthritis Pain VAS Score at Each Assessment Visit | | SAC[2] |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ACR50 | )/70 | 1 | | | , |
| 2.18. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR50 Response at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.19. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR70 Response at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.20. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR50/70 Response at Each Assessment Visit | Page by ACR50 and ACR70 | SAC[2] |
| CDAI F | Remission | | | | · |
| 2.21. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI Remission Response (CDAI≤2.8) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.22. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed CDAI Remission (CDAI≤2.8) at Each Assessment Visit | | SAC[2] |
| DAS28 | 3-CRP LDA | | | • | |
| 2.23. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-CRP LDA Response (DAS28-CRP≤3.2) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.24. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-CRP LDA Response (DAS28-CRP≤3.2) at Each Assessment Visit | | SAC[2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DAS28 | B-CRP Remiss | ion | | | |
| 2.25. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-CRP Remission<br>Response (DAS28-CRP<2.6) at Each Assessment Visit<br>(Primary Estimand) | | SAC[2] |
| 2.26. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-CRP Remission Response (DAS28-CRP<2.6) at Each Assessment Visit | | SAC[2] |
| DAS28 | B-ESR LDA | | | | |
| 2.27. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-ESR LDA Response (DAS28-ESR≤3.2) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.28. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-ESR LDA Response (DAS28-ESR≤3.2) at Each Assessment Visit | | SAC[2] |
| DAS28 | B-ESR Remiss | ion | | | |
| 2.29. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-ESR Remission<br>Response (DAS28-ESR<2.6) at Each Assessment Visit<br>(Primary Estimand) | | SAC[2] |
| 2.30. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-ESR Remission Response (DAS28-ESR<2.6) at Each Assessment Visit | | SAC[2] |

| Efficac | cy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Good/ | Moderate EUL | AR Response | | | |
| 2.31. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of Good/Moderate EULAR Response (based on DAS28-CRP) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.32. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed Good/Moderate EULAR Response (based on DAS28-CRP) at Each Assessment Visit | | SAC[2] |
| ACR/E | ULAR Remiss | ion Boolean-bas | sed and Index-based | | · |
| 2.33. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed Index-based ACR/EULAR Remission Response at Each Assessment Visit | | SAC[2] |
| 2.34. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed Boolean-based ACR/EULAR Remission Response at Each Assessment Visit | | SAC[2] |
| Radio | graphic Progre | ession (change f | rom baseline in van der Heijde mTSS score) | | 1 |
| 2.35. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed Proportion of Subjects with Change from Baseline in Van der Heijde mTSS of ≤0 and ≤0.5 at Each Assessment Visit | Page by ≤0 and ≤0.5 | SAC[2] |
| 2.36. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Van der Heijde mTSS at Each Assessment Visit | | SAC[2] |
| Tende | r Joint Counts | 3 | | | |
| 2.37. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in TJC28 at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.38. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in TJC68 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.39. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in TJC28 and TJC68 at Each Assessment Visit | | SAC[2] |
| Swolle | n Joint Count | s | | | |
| 2.40. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in SJC28 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.41. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in SJC66 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.42. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in SJC28 and SJC66 at Each Assessment Visit | | SAC[2] |
| CRP/E | SR | | | | |
| 2.43. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in CRP (mg/L) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.44. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in CRP (mg/L) and ESR (mm/h) at Each Assessment Visit | | SAC[2] |
| 2.45. | ITT | Non-Standard<br>EFF_T5 | Summary of Ratio to Baseline in CRP (mg/L) and ESR (mm/h) at Each Assessment Visit (Log Transformed) | | SAC[2] |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Patien | t's Global Ass | essment | | | |
| 2.46. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Patient's Global<br>Assessment of Arthritis at Each Assessment Visit (Primary<br>Estimand) | | SAC[2] |
| 2.47. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Patient's Global Assessment of Arthritis at Each Assessment Visit | | SAC[2] |
| Physic | ian's Global A | Assessment | | | |
| 2.48. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Physician's Global Assessment of Arthritis at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.49. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Physician's Global Assessment of Arthritis at Each Assessment Visit | | SAC[2] |
| DAS28 | B-CRP | | | | |
| 2.50. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in DAS28-CRP at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.51. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in DAS28-CRP at Each Assessment Visit | | SAC[2] |
| DAS28 | B-ESR | | | | |
| 2.52. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in DAS28-ESR at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.53. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in DAS28-<br>ESR at Each Assessment Visit | | SAC[2] |
| SF-36 | (Physical, Mei | ntal and Individu | al Components) | | |
| 2.54. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Physical Component Score (PCS) of SF-36 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.55. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Physical Component Score (PCS) of SF-36 at Each Assessment Visit | | SAC[2] |
| 2.56. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Mental Component Score (MCS) of SF-36 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.57. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Mental Component Score (MCS) of SF-36 at Each Assessment Visit | | SAC[2] |
| 2.58. | ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Domain Scores of SF-36 at Each Assessment Visit | | SAC[2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |
| - | | | | | |
| _ | | | | | |
| _ | | | | | |
| - | | | | | |
| - | | | | | |
| - | | | | | |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.89. | ITT | Non-Standard<br>EFF_T2 | Summary of Observed Change from Baseline in SF-36 Physical Component Score ≥10 and Mental Component Score≥8 (WPMI) at Each Assessment Visit | | AAC[3] |
| CCI | | | | | |
| Sensit | ivity Analyses | ; | | | |
| 2.92. | Per<br>Protocol | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each Assessment Visit (Primary Estimand) (Per Protocol Population) | | AAC[3] |
| Radiog | raphic Progre | ession (change f | rom baseline in van der Heijde mTSS score) | | |
| 2.93. | ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Van der Heijde mTSS<br>Score at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.94. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of the Proportion of Subjects with Change from Baseline in Van der Heijde mTSS ≤ 0 at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.95. | ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of the Proportion of Subjects with Change from Baseline in Van der Heijde mTSS ≤ 0.5 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| Japan | Subgroup | | | | • |
| 2.301. | Japanese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each<br>Assessment Visit (Primary Estimand) for Japanese<br>Subjects | | Asia AAC[4] |
| 2.302. | Japanese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR20 Response at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.303. | Japanese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit (Primary Estimand) for Japanese Subjects | | Asia AAC[4] |
| 2.304. | Japanese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.305. | Japanese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) for Japanese Subjects | | Asia AAC[4] |
| 2.306. | Japanese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in HAQ-DI Score and in Functional Areas of the HAQ-DI Score at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.307. | Japanese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in CDAI Total score at Each Assessment Visit (Primary Estimand) for Japanese Subjects | | Asia AAC[4] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.308. | Japanese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in CDAI<br>Total Score at Each Assessment Visit for Japanese<br>Subjects | | Asia AAC[4] |
| 2.309. | Japanese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in FACIT-Fatigue at Each Assessment Visit (Primary Estimand) for Japanese Subjects | | Asia AAC[4] |
| 2.310. | Japanese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in FACIT-<br>Fatigue at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.311. | Japanese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Arthritis Pain VAS<br>Score at Each Assessment Visit (Primary Estimand) for<br>Japanese Subjects | | Asia AAC[4] |
| 2.312. | Japanese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Arthritis Pain VAS Score at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.313. | Japanese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR50 Response at Each<br>Assessment Visit (Primary Estimand) for Japanese<br>Subjects | | Asia AAC[4] |
| 2.314. | Japanese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR70 Response at Each<br>Assessment Visit (Primary Estimand) for Japanese<br>Subjects | | Asia AAC[4] |
| 2.315. | Japanese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR50/70 Response at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.316. | Japanese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in DAS28-CRP at Each Assessment Visit (Primary Estimand) for Japanese Subjects | | Asia AAC[4] |
| 2.317. | Japanese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in DAS28-CRP at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.318. | Japanese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in DAS28-ESR at Each Assessment Visit (Primary Estimand) for Japanese Subjects | | Asia AAC[4] |
| 2.319. | Japanese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in DAS28-<br>ESR at Each Assessment Visit for Japanese Subjects | | Asia AAC[4] |
| 2.320. | Japanese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed Proportion of Subjects with Change from Baseline in Van der Heijde mTSS of ≤0 and ≤0.5 at Each Assessment Visit for Japanese Subjects | Page by ≤0 and ≤0.5 | Asia AAC[4] |
| China | Subgroup | | | | · |
| 2.401. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.402. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each<br>Assessment Visit (Supplemental Estimand 1) for Chinese<br>Subjects | | Asia AAC[4] |
| 2.403. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR20 Response at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.404. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI-LDA Response at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.405. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.406. | Chinese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.407. | Chinese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in HAQ-DI<br>Score and in Functional Areas of the HAQ-DI Score at<br>Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.408. | Chinese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in CDAI Total score at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.409. | Chinese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in CDAI Total Score at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.410. | Chinese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in FACIT-Fatigue at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.411. | Chinese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in FACIT-<br>Fatigue at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.412. | Chinese<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in Arthritis Pain VAS<br>Score at Each Assessment Visit (Primary Estimand) for<br>Chinese Subjects | | Asia AAC[4] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.413. | Chinese<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in Arthritis Pain VAS Score at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.414. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR50 Response at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.415. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR70 Response at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.416. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR50/70 Response at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.417. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI Remission Response (CDAI≤2.8) at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.418. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed CDAI Remission (CDAI≤2.8) at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.419. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-CRP LDA Response (DAS28-CRP≤3.2) at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.420. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-CRP LDA Response (DAS28-CRP≤3.2) at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.421. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-CRP Remission<br>Response (DAS28-CRP<2.6) at Each Assessment Visit<br>(Primary Estimand) for Chinese Subjects | | Asia AAC[4] |

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.422. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-CRP Remission Response (DAS28-CRP<2.6) at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.423. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-ESR LDA Response (DAS28-ESR≤3.2) at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.424. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-ESR LDA Response (DAS28-ESR≤3.2) at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.425. | Chinese<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of DAS28-ESR Remission<br>Response (DAS28-ESR<2.6) at Each Assessment Visit<br>(Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.426. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed DAS28-ESR Remission Response (DAS28-ESR<2.6) at Each Assessment Visit for Chinese Subjects | | Asia AAC[4] |
| 2.427. | Chinese<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed Proportion of Subjects with Change from Baseline in Van der Heijde mTSS of ≤0 and ≤0.5 at Each Assessment Visit for Chinese Subjects | Page by ≤0 and ≤0.5 | Asia AAC[4] |
| Asia S | ubgroup | | | <u> </u> | |
| 2.501. | Asia<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of ACR20 Response at Each Assessment Visit (Primary Estimand) for Asia Subjects | | Asia AAC[4] |
| 2.502. | Asia<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed ACR20 Response at Each Assessment Visit for Asia Subjects | | Asia AAC[4] |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.503. | Asia<br>ITT | Non-Standard<br>EFF_T1 | Summary and Analysis of CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit (Primary Estimand) for Asia Subjects | | Asia AAC[4] |
| 2.504. | Asia<br>ITT | Non-Standard<br>EFF_T2 | Summary of Observed CDAI-LDA Response (CDAI ≤10) at Each Assessment Visit for Asia Subjects | | Asia AAC[4] |
| 2.505. | Asia<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) for Asia Subjects | | Asia AAC[4] |
| 2.506. | Asia<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in HAQ-DI<br>Score and in Functional Areas of the HAQ-DI Score at<br>Each Assessment Visit for Asia Subjects | | Asia AAC[4] |
| 2.507. | Asia<br>ITT | Non-Standard<br>EFF_T3 | Analysis of Change from Baseline in CDAI Total score at Each Assessment Visit (Primary Estimand) for Asia Subjects | | Asia AAC[4] |
| 2.508. | Asia<br>ITT | Non-Standard<br>EFF_T4 | Summary of Observed Change from Baseline in CDAI Total Score at Each Assessment Visit for Asia Subjects | | Asia AAC[4] |

## **Efficacy Figures**

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ACR20 | | | | | |
| 2.1. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR20 Response at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| 2.2. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR20 Response at Each Assessment Visit (Supplemental Estimand 1) | | SAC[2] |
| 2.3. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR20 Response at Each Assessment Visit (Supplemental Estimand 2) | | AAC[3] |
| CDAI-L | .DA | | | | |
| 2.4. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving CDAI-LDA (CDAI ≤10) at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| 2.5. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving CDAI-LDA (CDAI ≤10) at Each Assessment Visit (Supplemental Estimand 1) | | SAC[2] |
| HAQ-D | l | | | | |
| 2.6. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| CDAI T | otal Score | | | | |
| 2.7. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in CDAI Total Score at Each Assessment Visit (Primary Estimand) | | HDL[1] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in CDAI Total Score at Each Assessment Visit (Supplemental Estimand 2) | | AAC[3] |
| FACIT- | Fatigue | | | | |
| 2.9. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in FACIT-Fatigue at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| Arthrit | is Pain VAS | | | | |
| 2.10. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Arthritis Pain VAS at Each Assessment Visit (Primary Estimand) | | HDL[1] |
| 2.11. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Arthritis Pain VAS at Each Assessment Visit (Supplemental Estimand 2) | | AAC[3] |
| ACR50 | /70 | | | | |
| 2.12. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR50 Response at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.13. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR70 Response at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| CDAI F | Remission | | | | |
| 2.14. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving CDAI Remission (CDAI≤2.8) at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DAS28 | -CRP LDA | | | | |
| 2.15. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving DAS28-CRP LDA (DAS28-CRP≤3.2) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| DAS28 | -CRP Remiss | ion | | | |
| 2.16. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving DAS28-CRP Remission (DAS28-CRP<2.6) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| DAS28 | -ESR LDA | | | | |
| 2.17. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving DAS28-ESR LDA (DAS28-ESR≤3.2) at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DAS28 | B-ESR Remiss | ion | | | |
| 2.18. | ІТТ | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving DAS28-ESR Remission (DAS28-ESR<2.6) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| Good/l | Moderate EUL | AR Response | | | |
| 2.19. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving Good/Moderate EULAR Response (based on DAS28-CRP) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| Radio | graphic Progre | ession (change f | rom baseline in van der Heijde mTSS score) | | |
| 2.20. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving Change from Baseline in mTSS of ≤0 and ≤0.5 at Each Assessment Visit | | SAC[2] |
| 2.21. | ITT | Non-Standard<br>EFF_F2 | Plot of Change from Baseline in mTSS at Each<br>Assessment Visit | | SAC[2] |
| 2.22. | ITT | Non-Standard<br>EFF_F7 | Cumulative Probability Plots of Individual Subject Changes from Baseline in mTSS at Each Assessment Visit | | SAC[2] |
| Tende | r Joint Counts | 3 | | | |
| 2.23. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in TJC28 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.24. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in TJC68 at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Swolle | Swollen Joint Counts | | | | |
| 2.25. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in SJC28 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.26. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in SJC66 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| CRP | | | | | |
| 2.27. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in CRP (mg/L) at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| Patien | t's Global Ass | essment | | | |
| 2.28. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Patient's Global Assessment at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| Physic | ian's Global <i>A</i> | Assessment | | | |
| 2.29. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Physician's Global Assessment at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| DAS28 | B-CRP | | | | |
| 2.30. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in DAS28-CRP at Each Assessment Visit (Primary Estimand) | | SAC[2] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| DAS28 | -ESR | | | | |
| 2.31. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in DAS28-ESR at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| SF-36 ( | Physical, Mer | ntal and Individu | al Components) | | |
| 2.32. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Physical Component Score (PCS) of SF-36 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.33. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means Change from Baseline in Mental Component Score (MCS) of SF-36 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.34. | ITT | Non-Standard<br>EFF_F3 | Spydergram of Individual Domain Scores of SF-36 at Each Assessment Visit | | SAC[2] |
| Subgro | up: ACR20 | | | | |
| 2.35. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Demographic Subgroup Results for ACR20 – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.36. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Demographic Subgroup Results for ACR20 – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| 2.37. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Disease Characteristic Subgroup Results for ACR20 – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.38. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Disease Characteristic Subgroup Results for ACR20 – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| Subgro | oup: CDAI-LD | A | | | |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.39. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Demographic Subgroup Results for CDAI-<br>LDA – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.40. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Demographic Subgroup Results for CDAI-<br>LDA – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| 2.41. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Disease Characteristic Subgroup Results for CDAI-LDA – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.42. | ITT | Non-Standard<br>EFF_F4 | Forest Plot of Disease Characteristic Subgroup Results for CDAI-LDA – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| Subgro | oup: HAQ-DI | | | | • |
| 2.43. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Demographic Subgroup Results for Change from Baseline in HAQ-DI – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.44. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Demographic Subgroup Results for Change from Baseline in HAQ-DI – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| 2.45. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Disease Characteristic Subgroup Results for Change from Baseline in HAQ-DI – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.46. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Disease Characteristic Subgroup Results for Change from Baseline in HAQ-DI – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| Subgro | oup: CDAI Tot | al | | | |

| Efficad | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.47. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Demographic Subgroup Results for Change from Baseline in CDAI Total Score – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.48. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Demographic Subgroup Results for Change from Baseline in CDAI Total Score – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| 2.49. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Disease Characteristic Subgroup Results for Change from Baseline in CDAI Total Score – Comparison to Placebo at Week 12 | | SAC[2] |
| 2.50. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Disease Characteristic Subgroup Results for Change from Baseline in CDAI Total Score – Comparison to Tofacitinib at Week 24 | | SAC[2] |
| Subgr | oup: Arthritis | Pain VAS | | | |
| 2.51. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Demographic Subgroup Results for Change from Baseline in Arthritis Pain VAS – Comparison to Placebo at Week 12 | | AAC[3] |
| 2.52. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Demographic Subgroup Results for Change from Baseline in Arthritis Pain VAS – Comparison to Tofacitinib at Week 24 | | AAC[3] |
| 2.53. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Disease Characteristic Subgroup Results for Change from Baseline in Arthritis Pain VAS – Comparison to Placebo at Week 12 | | AAC[3] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.54. | ITT | Non-Standard<br>EFF_F5 | Forest Plot of Disease Characteristic Subgroup Results for Change from Baseline in Arthritis Pain VAS – Comparison to Tofacitinib at Week 24 | | AAC[3] |
| Additio | onal Figures S | plitting out Pool | led Placebo Post Week 12 | | |
| 2.55. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR20 Response at Each Assessment Visit (Primary Estimand) Splitting out Pooled Placebo Post Week 12 | Display pooled placebo arm split out after week 12 | AAC[3] |
| 2.56. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving CDAI-LDA (CDAI≤10) at Each Assessment Visit (Primary Estimand) Splitting out Pooled Placebo Post Week 12 | Display pooled placebo arm split out after week 12 | AAC[3] |
| 2.57. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) Splitting out Pooled Placebo Post Week 12 | Display pooled placebo arm split out after week 12 | AAC[3] |
| 2.58. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in CDAI Total Score at Each Assessment Visit (Primary Estimand) Splitting out Pooled Placebo Post Week 12 | Display pooled placebo arm split out after week 12 | AAC[3] |
| 2.59. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Arthritis Pain VAS at Each Assessment Visit (Primary Estimand) Splitting out Pooled Placebo Post Week 12 | Display pooled placebo arm split out after week 12 | AAC[3] |
| 2.60. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR50 Response at Each Assessment Visit (Primary Estimand) Splitting out Pooled Placebo Post Week 12 | Display pooled placebo arm split out after week 12 | AAC[3] |

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CI | | | | | |

| No. P | Population | Example<br>Shell | Title | Programming Notes | [Priority] |
|---|---|---|---|---|---|

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Radiog | graphic Progre | ession (change f | rom baseline in van der Heijde mTSS score) | | |
| 2.78. | ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in Van der Heijde mTSS at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.79. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving Change from Baseline in Van der Heijde mTSS ≤ 0 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| 2.80. | ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving Change from Baseline in Van der Heijde mTSS ≤ 0.5 at Each Assessment Visit (Primary Estimand) | | SAC[2] |
| China | Subgroup | | | | |
| 2.401. | Chinese<br>ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR20 Response at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.402. | Chinese<br>ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving CDAI-LDA (CDAI ≤10) at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| 2.403. | Chinese<br>ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in HAQ-DI Score at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.404. | Chinese<br>ITT | Non-Standard<br>EFF_F2 | Plot of Least Squares Means of Change from Baseline in CDAI Total Score at Each Assessment Visit (Primary Estimand) for Chinese Subjects | | Asia AAC[4] |
| Asia S | ubgroup | | | | |
| 2.501. | Asia<br>ITT | Non-Standard<br>EFF_F1 | Proportion of Subjects Achieving ACR20 Response at Each Assessment Visit (Primary Estimand) for Asia Subjects | | Asia AAC[4] |

## Safety Tables

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events (AEs | s) | | | |
| 3.1. | Safety | AE13 | Overall Summary of Adverse Events (Period 1) | | SAC[2] |
| 3.2. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE13 | Overall Summary of Adverse Events (Period 2) | | SAC[2] |
| 3.3. | Safety | AE13 | Overall Summary of Adverse Events (Period 1+2) | | SAC[2] |
| 3.4. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1) | ICH E3 | SAC[2] |
| 3.5. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 2) | ICH E3 | SAC[2] |
| 3.6. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1+2) | ICH E3 | SAC[2] |
| 3.7. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1) | ICH E3 | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.8. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 2) | ICH E3 | SAC[2] |
| 3.9. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1+2) | ICH E3 | SAC[2] |
| 3.10. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Period 1) | ICH E3 | HDL[1] |
| 3.11. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Period 2) | ICH E3 | SAC[2] |
| 3.12. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Period 1+2) | ICH E3 | HDL[1] |
| 3.13. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1) | IDSL | SAC[2] |
| 3.14. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 2) | IDSL | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.15. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1+2) | IDSL | SAC[2] |
| 3.16. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency (Period 1) | ICH E3 | SAC[2] |
| 3.17. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency (Period 2) | ICH E3 | SAC[2] |
| 3.18. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency (Period 1+2) | ICH E3 | SAC[2] |
| 3.19. | Safety | AE15 | Summary of Common (>=5%) Non-Serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subject and Occurrences) (Period 1) | FDAAA, EudraCT | SAC[2] |
| 3.20. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE15 | Summary of Common (>=5%) Non-Serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subject and Occurrences) (Period 2) | FDAAA, EudraCT | SAC[2] |
| 3.21. | Safety | AE15 | Summary of Common (>=5%) Non-Serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subject and Occurrences) (Period 1+2) | FDAAA, EudraCT | SAC[2] |
| Safety | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.22. | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) (Period 1) | FDAAA, EudraCT | SAC[2] |
| 3.23. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) (Period 2) | FDAAA, EudraCT | SAC[2] |
| 3.24. | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) (Period 1+2) | FDAAA, EudraCT | SAC[2] |
| 3.25. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 1) | ICH E3 | SAC[2] |
| 3.26. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 2) | ICH E3 | SAC[2] |
| 3.27. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 1+2) | ICH E3 | SAC[2] |
| 3.28. | Safety | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 1) | ICH E3 | SAC[2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.29. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 2) | ICH E3 | SAC[2] |
| 3.30. | Safety | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 1+2) | ICH E3 | SAC[2] |
| 3.31. | Safety | AE3 | Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency (Period 1) | PLS Requirements | SAC[2] |
| 3.32. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE3 | Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency (Period 2) | PLS Requirements | SAC[2] |
| 3.33. | Safety | AE3 | Summary of Non-Serious Drug-Related Adverse Events by Overall Frequency (Period 1+2) | PLS Requirements | SAC[2] |
| 3.34. | Safety | AE20 | Summary of Serious Fatal and Non-Fatal Drug-Related Adverse Events by Overall Frequency (Period 1) | PLS Requirements | SAC[2] |
| 3.35. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | AE20 | Summary of Serious Fatal and Non-Fatal Drug-Related Adverse Events by Overall Frequency (Period 2) | PLS Requirements | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.36. | Safety | AE20 | Summary of Serious Fatal and Non-Fatal Drug-Related Adverse Events by Overall Frequency (Period 1+2) | PLS Requirements | SAC[2] |
| 3.37. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for All Adverse Events (Period 1) | | SAC[2] |
| 3.38. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for All Adverse Events (Period 2) | | SAC[2] |
| 3.39. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for All Adverse Events (Period 1+2) | | SAC[2] |
| Advers | se Events of S | pecial Interest ( | AESI) and Other Important AEs | | |
| 3.40. | Safety | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 1) | | HDL[1] |
| 3.41. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 2) | | SAC[2] |
| 3.42. | Safety | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 1+2) | | HDL[1] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.43. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Adverse Events of Special Interest (Period 1) | | SAC[2] |
| 3.44. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Adverse Events of Special Interest (Period 2) | | SAC[2] |
| 3.45. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Adverse Events of Special Interest (Period 1+2) | | SAC[2] |
| 3.46. | Safety | Non-Standard<br>SAFE_T3 | Summary of Other Important Adverse Events (Period 1) | | SAC[2] |
| 3.47. | Safety | Non-Standard<br>SAFE_T3 | Summary of Other Important Adverse Events (Period 2) | | SAC[2] |
| 3.48. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T3 | Summary of Other Important Adverse Events (Period 1+2) | | SAC[2] |
| 3.49. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Other Important Adverse Events (Period 1) | | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.50. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Other Important Adverse Events (Period 2) | | SAC[2] |
| 3.51. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Other Important Adverse Events (Period 1+2) | | SAC[2] |
| 3.52. | Safety | Non-Standard<br>SAFE_T4 | Summary of Adjudicated Cardiovascular Event Categories (Period 1) | | SAC[2] |
| 3.53. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T4 | Summary of Adjudicated Cardiovascular Event Categories (Period 2) | | SAC[2] |
| 3.54. | Safety | Non-Standard<br>SAFE_T4 | Summary of Adjudicated Cardiovascular Event Categories (Period 1+2) | | SAC[2] |
| 3.55. | Safety | ESI1<br>(modified) | Summary of Characteristics of Injection Site Reactions (Period 1) | | SAC[2] |
| 3.56. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | ESI1<br>(modified) | Summary of Characteristics of Injection Site Reactions (Period 2) | | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.57. | Safety | ESI1<br>(modified) | Summary of Characteristics of Injection Site Reactions (Period 1+2) | | SAC[2] |
| 3.58. | Safety | Non-Standard<br>SAFE_T5 | Summary of Injection Site Reactions (Period 1) | | SAC[2] |
| 3.59. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T5 | Summary of Injection Site Reactions (Period 2) | | SAC[2] |
| 3.60. | Safety | Non-Standard<br>SAFE_T5 | Summary of Injection Site Reactions (Period 1+2) | | SAC[2] |
| 3.61. | Safety | Non-Standard<br>SAFE_T6 | Summary of Serious or Adjudicated Opportunistic Infections (Period 1) | | SAC[2] |
| 3.62. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T6 | Summary of Serious or Adjudicated Opportunistic Infections (Period 2) | | SAC[2] |
| 3.63. | Safety | Non-Standard<br>SAFE_T6 | Summary of Serious or Adjudicated Opportunistic Infections (Period 1+2) | | SAC[2] |
| 3.64. | Safety | Non-Standard<br>SAFE_T7 | Summary of Adjudicated Serious Hypersensitivity Reactions (Period 1) | | SAC[2] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.65. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T7 | Summary of Adjudicated Serious Hypersensitivity<br>Reactions (Period 2) | | SAC[2] |
| 3.66. | Safety | Non-Standard<br>SAFE_T7 | Summary of Adjudicated Serious Hypersensitivity Reactions (Period 1+2) | | SAC[2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pulmo | nary Findings | | | | |
| 3.67. | Safety | Non-Standard<br>SAFE_T8 | Summary of Pulmonary Findings (Period 1) | | SAC[2] |
| 3.68. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T8 | Summary of Pulmonary Findings (Period 2) | | SAC[2] |
| 3.69. | Safety | Non-Standard<br>SAFE_T8 | Summary of Pulmonary Findings (Period 1+2) | | SAC[2] |
| 3.70. | Safety | Non-Standard<br>SAFE_T9 | Summary of Pulse Oximetry Results (Period 1) | | SAC[2] |
| 3.71. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T9 | Summary of Pulse Oximetry Results (Period 2) | | SAC[2] |
| 3.72. | Safety | Non-Standard<br>SAFE_T9 | Summary of Pulse Oximetry Results (Period 1+2) | | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | atory: Chemist | ry, Hematology | & Fasting Lipids | | · |
| 3.73. | Safety | LB1 | Summary of Chemistry Changes from Baseline (Period 1) | ICH E3<br>Exclude CRP | SAC[2] |
| 3.74. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB1 | Summary of Chemistry Changes from Baseline (Period 2) | ICH E3<br>Exclude CRP | SAC[2] |
| 3.75. | Safety | LB1 | Summary of Chemistry Changes from Baseline (Period 1+2) | ICH E3<br>Exclude CRP | SAC[2] |
| 3.76. | Safety | LB16A<br>(modified) | Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1) | ICH E3 | SAC[2] |
| 3.77. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB16A<br>(modified) | Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 2) | ICH E3 | SAC[2] |
| 3.78. | Safety | LB16A<br>(modified) | Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1+2) | ICH E3 | SAC[2] |

| Safety | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.79. | Safety | LB1 | Summary of Hematology Changes from Baseline (Period 1) | ICH E3<br>Exclude ESR | SAC[2] |
| 3.80. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB1 | Summary of Hematology Changes from Baseline (Period 2) | ICH E3<br>Exclude ESR | SAC[2] |
| 3.81. | Safety | LB1 | Summary of Hematology Changes from Baseline (Period 1+2) | ICH E3<br>Exclude ESR | SAC[2] |
| 3.82. | Safety | LB16A<br>(modified) | Summary of Worst Case Hematology Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1) | ICH E3 | SAC[2] |
| 3.83. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB16A<br>(modified) | Summary of Worst Case Hematology Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 2) | ICH E3 | SAC[2] |
| 3.84. | Safety | LB16A<br>(modified) | Summary of Worst Case Hematology Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1+2) | ICH E3 | SAC[2] |
| 3.85. | Safety | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 1) | | SAC[2] |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.86. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 2) | | SAC[2] |
| 3.87. | Safety | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 1+2) | | SAC[2] |
| 3.88. | Safety | LB18 | Summary of Laboratory Parameters of Interest CTCAE Worst Grade Shift from Baseline Grade (Period 1) | | SAC[2] |
| 3.89. | Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | LB18 | Summary of Laboratory Parameters of Interest CTCAE<br>Worst Grade Shift from Baseline Grade (Period 2) | | SAC[2] |
| 3.90. | Safety | LB18 | Summary of Laboratory Parameters of Interest CTCAE<br>Worst Grade Shift from Baseline Grade (Period 1+2) | | SAC[2] |
| 3.91. | Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Period 1) | ICH E3 | SAC[2] |
| 3.92. | Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Period 2) | ICH E3 | SAC[2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.93. | Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Period 1+2) | ICH E3 | SAC[2] |
| Labora | tory: Hepatob | oiliary (Liver) | | | |
| 3.94. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting (Period 1) | IDSL | SAC[2] |
| 3.95. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting (Period 2) | IDSL | SAC[2] |
| 3.96. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting (Period 1+2) | IDSL | SAC[2] |
| 3.97. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Period 1) | IDSL | SAC[2] |
| 3.98. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Period 2) | IDSL | SAC[2] |
| 3.99. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Period 1+2) | IDSL | SAC[2] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 3.100. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC[2] |
| 3.101. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit (Period 1) | IDSL | SAC[2] |
| 3.102. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | EG2 | Summary of Change from Baseline in ECG Values by Visit (Period 2) | IDSL | SAC[2] |
| 3.103. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit (Period 1+2) | IDSL | SAC[2] |
| 3.104. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category (Period 1) | IDSL | SAC[2] |
| 3.105. | Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category (Period 2) | IDSL | SAC[2] |
| 3.106. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category (Period 1+2) | IDSL | SAC[2] |
| 3.107. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-<br>Baseline Relative to Baseline by Category (Period 1) | IDSL | SAC[2] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.108. | Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | EG11 | Summary of Maximum Increase in QTc Values Post-<br>Baseline Relative to Baseline by Category (Period 2) | IDSL | SAC[2] |
| 3.109. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-<br>Baseline Relative to Baseline by Category (Period 1+2) | IDSL | SAC[2] |
| Vital Si | gns | | | | · |
| 3.110. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Period 1) | ICH E3 | SAC[2] |
| 3.111. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | VS1 | Summary of Change from Baseline in Vital Signs (Period 2) | ICH E3 | SAC[2] |
| 3.112. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Period 1+2) | ICH E3 | SAC[2] |
| 3.113. | Safety | VS3 | Summary of Worst Case Vital Signs Results Relative to Normal Range Post-Baseline Relative to Baseline (Period 1) | IDSL | SAC[2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.114. | Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | VS3 | Summary of Worst Case Vital Signs Results Relative to Normal Range Post-Baseline Relative to Baseline (Period 1) | IDSL | SAC[2] |
| 3.115. | Safety | VS3 | Summary of Worst Case Vital Signs Results Relative to Normal Range Post-Baseline Relative to Baseline (Period 1+2) | IDSL | SAC[2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | Biomarkers (I | Immunogenicity | | | |
| 3.116. | Safety | Non-Standard<br>SAFE_T10 | Summary of Anti-GSK3196165 Antibodies (ADA) | | AAC[3] |
| 3.117. | Safety | Non-Standard<br>SAFE_T11 | Summary of Binding Antibody at Each Assessment Visit | | AAC[3] |
| 3.118. | Safety | Non-Standard<br>SAFE_T12 | Summary of Neutralising Antibody at Each Assessment Visit | | AAC[3] |
| COVID | -19 | | | | |
| 3.119. | Safety | PAN1 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events (Period 1) | | SAC[2] |
| 3.120. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | PAN1 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events (Period 2) | | SAC[2] |
| 3.121. | Safety | PAN1 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events (Period 1+2) | | SAC[2] |
| 3.122. | Safety | PAN2 | Summary of COVID-19 Additional Assessments for Subjects with COVID-19 Adverse Events (Period 1) | | SAC[2] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.123. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | PAN2 | Summary of COVID-19 Additional Assessments for Subjects with COVID-19 Adverse Events (Period 2) | | SAC[2] |
| 3.124. | Safety | PAN2 | Summary of COVID-19 Additional Assessments for Subjects with COVID-19 Adverse Events (Period 1+2) | | SAC[2] |
| 3.125. | Safety | PAN3 | Summary of COVID-19 Symptoms for Subjects with COVID-19 Adverse Events (Period 1) | Remove "no" and "unknown" rows | SAC[2] |
| 3.126. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | PAN3 | Summary of COVID-19 Symptoms for Subjects with COVID-19 Adverse Events (Period 2) | Remove "no" and "unknown" rows | SAC[2] |
| 3.127. | Safety | PAN3 | Summary of COVID-19 Symptoms for Subjects with COVID-19 Adverse Events (Period 1+2) | Remove "no" and "unknown" rows | SAC[2] |
| 3.128. | Safety | Non-Standard<br>SAFE_T13 | Summary of Adjudicated Serious Cases of COVID-19 Infections (Period 1) | | SAC[2] |
| 3.129. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T13 | Summary of Adjudicated Serious Cases of COVID-19 Infections (Period 2) | | SAC[2] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.130. | Safety | Non-Standard<br>SAFE_T13 | Summary of Adjudicated Serious Cases of COVID-19 Infections (Period 1+2) | | SAC[2] |
| 3.131. | Safety | Non-Standard<br>SAFE_T15 | Summary of COVID-19 Infections (Period 1) | | SAC[2] |
| 3.132. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T15 | Summary of COVID-19 Infections (Period 2) | | SAC[2] |
| 3.133. | Safety | Non-Standard<br>SAFE_T15 | Summary of COVID-19 Infections (Period 1+2) | | SAC[2] |
| Additio | nal Adverse l | Events | | | |
| 3.134. | Safety | Non-Standard<br>SAFE_T14 | Summary of Common (>=2%) Adverse Events by Time from Randomisation | | AAC[3] |
| Exposi | ure Adjusted | SAEs | | | |
| 3.135. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Serious Adverse Events (Period 1) | | SAC[2] |
| 3.136. | Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Serious Adverse Events (Period 2) | | SAC[2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.137. | Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Serious Adverse Events (Period 1+2) | | SAC[2] |
| Japan | subgroup | | | | |
| 3.301. | Japanese<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.302. | Japanese<br>Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.303. | Japanese<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.304. | Japanese<br>Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.305. | Japanese<br>Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.306. | Japanese<br>Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.307. | Japanese<br>Safety | AE1 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Period 1) for Japanese<br>Subjects | | Asia<br>AAC[4] |
| 3.308. | Japanese<br>Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Period 2) for Japanese<br>Subjects | | Asia<br>AAC[4] |
| 3.309. | Japanese<br>Safety | AE1 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Period 1+2) for Japanese<br>Subjects | | Asia<br>AAC[4] |
| 3.310. | Japanese<br>Safety | AE1 | Summary of Adverse Events Leading to Permanent<br>Discontinuation of Study Treatment by System Organ<br>Class and Preferred Term (Period 1) for Japanese<br>Subjects | | Asia<br>AAC[4] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.311. | Japanese<br>Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.312. | Japanese<br>Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.313. | Japanese<br>Safety | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.314. | Japanese<br>Safety –<br>Subjects<br>who<br>Entered<br>Period 2 | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.315. | Japanese<br>Safety | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.316. | Japanese<br>Safety | LB1 | Summary of Chemistry Changes from Baseline (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.317. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB1 | Summary of Chemistry Changes from Baseline (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.318. | Japanese<br>Safety | LB1 | Summary of Chemistry Changes from Baseline (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.319. | Japanese<br>Safety | LB16 | Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.320. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB16 | Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.321. | Japanese<br>Safety | LB16 | Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.322. | Japanese<br>Safety | LB1 | Summary of Hematology Changes from Baseline (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.323. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB1 | Summary of Hematology Changes from Baseline (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.324. | Japanese<br>Safety | LB1 | Summary of Hematology Changes from Baseline (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.325. | Japanese<br>Safety | LB16 | Summary of Worst Case Hematology Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.326. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB16 | Summary of Worst Case Hematology Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.327. | Japanese<br>Safety | LB16 | Summary of Worst Case Hematology Results by Maximum Grade Shift Post-Baseline Relative to Baseline (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.328. | Japanese<br>Safety | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.329. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.330. | Japanese<br>Safety | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.331. | Japanese<br>Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.332. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.333. | Japanese<br>Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.334. | Japanese<br>Safety | VS1 | Summary of Change from Baseline in Vital Signs (Period 1) for Japanese Subjects | | Asia<br>AAC[4] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.335. | Japanese<br>Safety -<br>Subjects<br>who<br>Entered<br>Period 2 | VS1 | Summary of Change from Baseline in Vital Signs (Period 2) for Japanese Subjects | | Asia<br>AAC[4] |
| 3.336. | Japanese<br>Safety | VS1 | Summary of Change from Baseline in Vital Signs (Period 1+2) for Japanese Subjects | | Asia<br>AAC[4] |
| China | Subgroup | | | | |
| 3.401. | Chinese<br>Safety | AE13 | Overall Summary of Adverse Events (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.402. | Chinese<br>Safety | AE13 | Overall Summary of Adverse Events (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.403. | Chinese<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.404. | Chinese<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.405. | Chinese<br>Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.406. | Chinese<br>Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |

| Safety: | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.407. | Chinese<br>Safety | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.408. | Chinese<br>Safety | AE1 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Period 1+2) for Chinese<br>Subjects | | Asia<br>AAC[4] |
| 3.409. | Chinese<br>Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.410. | Chinese<br>Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.411. | Chinese<br>Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.412. | Chinese<br>Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.413. | Chinese<br>Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for All Adverse Events (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.414. | Chinese<br>Safety | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 1) for Chinese Subjects | | Asia<br>AAC[4] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.415. | Chinese<br>Safety | Non-Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest (AESI) (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.416. | Chinese<br>Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Adverse Events of Special Interest (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.417. | Chinese<br>Safety | LB1 | Summary of Chemistry Changes from Baseline (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.418. | Chinese<br>Safety | LB1 | Summary of Hematology Changes from Baseline (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.419. | Chinese<br>Safety | LB1 | Summary of Fasting Lipids Changes from Baseline (Period 1+2) for Chinese Subjects | | Asia<br>AAC[4] |
| 3.420. | Chinese<br>Safety | Non-Standard<br>SAFE_T10 | Summary of Anti-GSK3196165 Antibodies (ADA) for Chinese Subjects | | Asia<br>AAC[4] |
| Asia Sı | ubgroup | | | | · |
| 3.501. | Asia<br>Safety | AE13 | Overall Summary of Adverse Events (Period 1) for Asia Subjects | | Asia<br>AAC[4] |
| 3.502. | Asia<br>Safety | AE13 | Overall Summary of Adverse Events (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |
| 3.503. | Asia<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1) for Asia Subjects | | Asia<br>AAC[4] |
| 3.504. | Asia<br>Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.505. | Asia<br>Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1) for Asia Subjects | | Asia<br>AAC[4] |
| 3.506. | Asia<br>Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |
| 3.507. | Asia<br>Safety | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Period 1) for Asia Subjects | | Asia<br>AAC[4] |
| 3.508. | Asia<br>Safety | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |
| 3.509. | Asia<br>Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1) for Asia Subjects | | Asia<br>AAC[4] |
| 3.510. | Asia<br>Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment by System Organ Class and Preferred Term (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |
| 3.511. | Asia<br>Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for All Adverse Events (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |
| 3.512. | Asia<br>Safety | Non-Standard<br>SAFE_T1 | Summary of Exposure Adjusted Event Rates per 100 Person Years for Adverse Events of Special Interest (Period 1+2) for Asia Subjects | | Asia<br>AAC[4] |

# Safety Figures

| Safety | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | |
| 3.1. | Safety | AE10 | Plot of Relative Risks for Common (>= 5%) Adverse Events | | SAC[2] |
| 3.2. | Safety | AE10 | Plot of Relative Risks for Adverse Events of Special Interest | | SAC[2] |
| Labora | tory: Chemis | try, Hematology | & Fasting Lipids | | |
| 3.3. | Safety | LB9 | Distribution of Laboratory Parameters of Interest by Time and Treatment with Maximum over Time | | SAC[2] |
| Labora | tory: Hepatok | oiliary (Liver) | | | |
| 3.4. | Safety | LIVER14 | Scatter Plot of Maximum vs Baseline for ALT | | SAC[2] |
| 3.5. | Safety | LIVER9 | Scatter Plot of Maximum Total Bilirubin vs Maximum ALT | | SAC[2] |
| Advers | Adverse Events (Treatment Policy Handling Strategy) | | | | |
| 3.6. | Safety | AE10 | Plot of Relative Risks for Common (>= 5%) Adverse Events (Treatment Policy Handling Strategy) | | AAC[3] |
| 3.7. | Safety | AE10 | Plot of Relative Risks for Adverse Events of Special Interest (Treatment Policy Handling Strategy) | | AAC[3] |

#### **Pharmacokinetic Tables**

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Co | ncentration | | | | |
| Japan | Subgroup | | - | 1 | |
| 4.301. | Japanese<br>PK | PK01 | Summary of GSK3196165 Serum Concentrations (ng/mL) by Visit for Japanese Subjects | | Asia AAC[4] |
| 4.302. | Non-<br>Japanese<br>PK | PK01 | Summary of GSK3196165 Serum Concentrations (ng/mL) by Visit for Non-Japanese Subjects | | Asia AAC[4] |
| Chines | se Subgroup | | | | |
| 4.401. | Chinese<br>PK | PK01 | Summary of GSK3196165 Serum Concentrations (ng/mL) by Visit for Chinese Subjects | | Asia AAC[4] |
| 4.402. | Non-<br>Chinese<br>PK | PK01 | Summary of GSK3196165 Serum Concentrations (ng/mL) by Visit for Non-Chinese Subjects | | Asia AAC[4] |
| Asia S | ubgroup | | • | | |
| 4.501. | Asia<br>PK | PK01 | Summary of GSK3196165 Serum Concentrations (ng/mL) by Visit for Asia Subjects | | Asia AAC[4] |
| 4.502. | Non-Asia<br>PK | PK01 | Summary of GSK3196165 Serum Concentrations (ng/mL) by Visit for Non-Asia Subjects | | Asia AAC[4] |

### **Biomarker Tables**

| Bioma | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

#### CONFIDENTIAL

201791 CCI

## **Biomarker Figures**

| 5101116 | arker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |

# ICH Listings

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ct Disposition | | | | · |
| 1. | Randomised | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC[2] |
| 2. | Randomised | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC[2] |
| 3. | ITT | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | SAC[2] |
| Proto | col Deviations | | | | |
| 4. | ITT | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC[2] |
| 5. | ITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC[2] |
| Popul | ations Analyse | d | | | · |
| 6. | Enrolled | SP3 | Listing of Subjects Excluded from Per Protocol Population | ICH E3 | SAC[2] |
| Demo | Demographic and Baseline Characteristics | | | | |
| 7. | ITT | DM2 | Listing of Demographic Characteristics | ICH E3 Include BMI in output. | SAC[2] |
| 8. | ITT | DM9 | Listing of Race | ICH E3 | SAC[2] |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | ure and Treatn | nent Complianc | e | | |
| 9. | Safety | EX3 | Listing of Exposure Data | ICH E3 | SAC[2] |
| Adver | se Events | | | | |
| 10. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | SAC[2] |
| 11. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC[2] |
| 12. | Safety | DD3 | Death Subject Profile | ICH E3 | SAC[2] |
| All Lal | boratory | | | | |
| 13. | Safety | LB5A | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC[2] |
| 14. | Safety | UR2 | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC[2] |

## **Non-ICH Listings**

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ct Disposition | | | | |
| 15. | Screened | ES7 | Listing of Reasons for Screen Failure | BIMO Requirements | SAC[2] |
| Protoc | col Deviations | | | | |
| 16. | ITT | DV2 | Listing of Non-Important COVID-19 related Protocol Deviations | COVID Requirements | SAC[2] |
| Prior a | and Concomita | nt Medications | | | |
| 17. | ITT | CM3 | Listing of Prior and Concomitant Medications | BIMO Requirements Include "medication taken for pain" | SAC[2] |
| 18. | ITT | CM3 | Listing of Intra-Articular Corticosteroids | Add columns for: "medication taken for pain" "Location of dose administration" "Laterality" | SAC[2] |
| Adver | se Events | | | | |
| 19. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | Non-ICH Required | SAC[2] |
| 20. | Safety | AE8XO | Listing of Non-Fatal Serious Adverse Events | Non-ICH Required Include "Action Taken with Background Therapy" | SAC[2] |
| 21. | Safety | AE8XO | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | Non-ICH Required Include "Action Taken with Background Therapy" | SAC[2] |
| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 22. | Safety | AE8XO | Listing of Other Significant Adverse Events | Non-ICH Required<br>Include "Action Taken with<br>Background Therapy" | SAC[2] |
| 23. | Safety | AE8XO | Listing of Adverse Events of Special Interest (AESI) | Include "Action Taken with Background Therapy" | SAC[2] |
| 24. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | BIMO Requirements | SAC[2] |
| 25. | Safety | Non-Standard<br>SAFE_L1 | Listing of Neutrophils and Associated Infections | Select the following subgroup and add under the title: "Subset of Subjects who experienced grade 3 or 4 Neutropenia" | SAC[2] |
| 26. | Safety | Non-Standard<br>SAFE_L1 | Listing of Lymphocytes and Associated Infections | Select the following subgroup and add under the title: "Subset of Subjects who experienced grade 3 or 4 Lymphopenia" | SAC[2] |
| Hepato | obiliary (Liver) | | | | |
| 27. | Safety | LIVER15 | Listing of Liver Event Stopping Profile | Non-ICH Required | SAC[2] |
| All Lab | ooratory | | | | |
| 28. | Safety | LB5A | Listing of All Local Laboratory Data | COVID Requirements | SAC[2] |

| Non-I | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 29. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | BIMO Requirements | SAC[2] |
| 30. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | BIMO Requirements | SAC[2] |
| Vital S | Signs | | | | • |
| 31. | Safety | VS4 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | BIMO Requirements | SAC[2] |
| 32. | Safety | PREG1 | Listing of Subjects Who Became Pregnant During the Study | Non-ICH Required | SAC[2] |
| COVIE | )-19 | | | | |
| 34. | ITT | PAN7 | Listing of All Subjects with Visits and Assessments Impacted by COVID-19 Pandemic | COVID Requirements | SAC[2] |
| 35. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom<br>Assessments for Subjects with COVID-19 Adverse<br>Events | COVID Requirements Include "Serious Event" | SAC[2] |
| 36. | Screened | PAN5 | Listing of Start Dates of COVID-19 Pandemic Measures by Country | COVID Requirements | SAC[2] |

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Cardio | Cardiovascular Event Listings (Conditionally required) | | | | |
| 37. | Safety | ARR1 | Arrhythmia Subject Profile | Non-ICH Required | AAC[3] |
| 38. | Safety | CHF1 | Congestive Heart Failure Subject Profile | Non-ICH Required | AAC[3] |
| 39. | Safety | CVATIA1 | Cerebrovascular Events/Stroke Subject Profile | Non-ICH Required | AAC[3] |
| 40. | Safety | DVT1 | Deep venous Thrombosis/ Pulmonary Embolism Subject Profile | Non-ICH Required | AAC[3] |
| 41. | Safety | MI1 | Myocardial Infarction /Unstable Angina Subject Profile | Non-ICH Required | AAC[3] |
| 42. | Safety | PATE1 | Peripheral Arterial Thrombosis Embolism Subject Profile | Non-ICH Required | AAC[3] |
| 43. | Safety | PUL1 | Pulmonary Hypertension Subject Profile | Non-ICH Required | AAC[3] |
| 44. | Safety | REV1 | Revascularization Subject Profile | Non-ICH Required | AAC[3] |
| 45. | Safety | VAL1 | Valvulopathy Subject Profile | Non-ICH Required | AAC[3] |

## 14.13. Appendix 13: Example Mock Shells for Data Displays

Example: POP\_T1
Protocol: 201791
Population: Safety

ocol: 201791 Page 1 of n

| | Treatment 1 (N=xx) | <pre>Treatment 2 (N=xx)</pre> | <pre>Treatment 3 (N=xx)</pre> | <pre>Treatment 4 (N=xx)</pre> | Treatment 5 (N=xx) | Treatment 6 (N=xx) |
|---|---|---|---|---|---|---|
| Subject Status | | | | | | |
| Completed | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Completed Safety Follow up | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Entered Long Term Extension | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Withdrawn | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Withdrawn in Period 1 [1] | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Withdrawn in Period 2 [2] | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Primary Reason [3] for Study | | | | | | |
| lithdrawal in Period 1 [1] | | | | | | |
| ADVERSE EVENT | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| LACK OF EFFICACY | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PROTOCOL DEVIATION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PROTOCOL-SPECIFIED WITHDRAWAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| CRITERION MET | | | | | | |
| STUDY TERMINATED BY SPONSOR | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| LOST TO FOLLOW-UP | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PHYSICIAN DECISION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| INFORMED CONSENT WITHDRAWN | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| INVESTIGATOR SITE CLOSED | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

201791

Example: POP\_T1 (cntd.)

Population: Safety

Table 1.1

Summary of Subject Status and Subject Disposition for the Study Conclusion Record

| | Treatment 1 (N=xx) | | | Treatment 5 (N=xx) | Treatment 6 (N=xx) | |
|---|---|---|---|---|---|---|
| Primary Reason [3] for Study | | | | | | |
| Withdrawal in Period 2 [2] | | | | | | |
| ADVERSE EVENT | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| LACK OF EFFICACY | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PROTOCOL DEVIATION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PROTOCOL-SPECIFIED WITHDRAWAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| CRITERION MET | | | | | | |
| STUDY TERMINATED BY SPONSOR | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| LOST TO FOLLOW-UP | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PHYSICIAN DECISION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| INFORMED CONSENT WITHDRAWN | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| INVESTIGATOR SITE CLOSED | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Outcome of Adverse Events Which | | | | | | |
| Led to Study Withdrawal in Period 1 [1] | | | | | | |
| NON-FATAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| FATAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Outcome of Adverse Events Which<br>Led to Study Withdrawal in Period 2 [2] | | | | | | |
| NON-FATAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| FATAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

<sup>[1]</sup> Period 1 - up to 12 weeks, defined as time from randomisation and first dose of treatment up to dosing of Period 2 treatment (Week 12) or date of study withdrawal or date of treatment withdrawal plus safety follow up whichever is earlier.

[2] Period 2 - post week 12, defined as time from first dose of treatment of period 2 (week 12) until date of study completion or date of study withdrawal or date of treatment withdrawal plus safety follow up whichever is earlier.

[3] Subjects may have only one primary reason.

201791

Example: POP\_T2
Protocol: 201791
Population: Safety

Protocol: 201791


| | | tment 1<br>=xx) | | ment 2<br>=xx) | | tment 3<br>=xx) | | ment 4<br>xx) | | ment 5<br>xx) | Treatr<br>(N= | nent 6<br>=xx) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Status | | | | | | | | | | | | |
| Prematurely Discontinued Treatment | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Prematurely Discontinued Treatment in Period 1 [1] | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Prematurely Discontinued Treatment in Period 2 [2] | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| Primary Reason [3] for Treatment | | | | | | | | | | | | |
| Discontinuation in Period 1 [1] | | | | | | | | | | | | |
| ADVERSE EVENT | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| LACK OF EFFICACY | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| PROTOCOL DEVIATION | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| PROTOCOL-SPECIFIED WITHDRAWAL CRITERION MET | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| STUDY TERMINATED BY SPONSOR | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| LOST TO FOLLOW-UP | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| PHYSICIAN DECISION | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| WITHDRAWAL BY SUBJECT | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| SPONSOR TERMINATED STUDY TREATMENT | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |
| INVESTIGATOR SITE CLOSED | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) | XX | (xx%) |

201791

Example: POP\_T2 (cntd.)


Population: Safety  ${\tt Table~1.x}$  Summary of Treatment Status and Reasons for Discontinuation of Study Treatment

| | Treatment 1 (N=xx) | Treatment 2 (N=xx) | Treatment 3 (N=xx) | Treatment 4 (N=xx) | Treatment 5 (N=xx) | Treatment 6 (N=xx) |
|---|---|---|---|---|---|---|
| Primary Reason [3] for Treatment | | | | | | |
| Discontinuation in Period 2 [2] | | | | | | |
| ADVERSE EVENT | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| LACK OF EFFICACY | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PROTOCOL DEVIATION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PROTOCOL-SPECIFIED WITHDRAWAL | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| CRITERION MET | | | | | | |
| STUDY TERMINATED BY SPONSOR | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| LOST TO FOLLOW-UP | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PHYSICIAN DECISION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| WITHDRAWAL BY SUBJECT | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| SPONSOR TERMINATED STUDY TREATMENT | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| INVESTIGATOR SITE CLOSED | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

<sup>[1]</sup> Treatment Discontinuation in Period 1- defined as time from first dose of treatment up to date of treatment withdrawal prior to week 12 dosing.

<sup>[2]</sup> Treatment Discontinuation in Period 2- defined as time from first dose of treatment period 2 (week 12) until date of treatment withdrawal post week 12.

<sup>[3]</sup> Subjects may have only one primary reason for treatment discontinuation.

201791


Example: POP\_T3
Protocol: 201791
Population: Intent-to-Treat

Table 1.x Baseline Efficacy Parameters

| | Statistic | Treatment 1 (N=xx) | Treatment 2 (N=xx) | Treatment 3 (N=xx) | Treatment 4 (N=xx) |
|---|---|---|---|---|---|
| Swollen Joint Count 28 | n | XX | xx | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Minimum | xx | XX | XX | XX |
| | Maximum | XX | XX | XX | XX |
| Swollen Joint Count 66 | n | XX | XX | XX | xx |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | xx.xx | xx.xx | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX | XX | XX | XX |
| | Maximum | XX | XX | xx | XX |
| Tender Joint Count 28 | n | xx | XX | xx | xx |
| Tender Joint Count 68 | n | | | | |
| | | XX | XX | XX | XX |
| | <br>n | ··· | ··· | ··· | |
| | n | XX | XX | XX | XX |

Example: POP T4

Population: Intent-to-Treat

Table 1.x
Summary of Rheumatoid Arthritis Disease History

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment 6 |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Time since RA diagnosi | s (years) | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | xxx | XXX | XXX | XXX | XXX | XXX |
| Max. | XXX | XXX | XXX | XXX | XXX | XXX |
| Time since RA diagnosi | S | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| <= 2 years | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >2-5 years | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >5-10 years | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >10 years | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Missing | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| RA functional class | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| I | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| II | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| III | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Time since start of RA | symptoms (years) | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | x.xx | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | xxx | XXX | XXX | XXX | XXX | XXX |
| Max. | xxx | XXX | XXX | XXX | XXX | XXX |

Note: Time since RA diagnosis and start of RA symptoms is calculated up to date of first study medication administration. [1] Stratum information is obtained from IWRS.

Example: POP\_T4 (continued)
Protocol: 201791 Confidential
Population: Intent-to-Treat


| | Treatment 1 N=xx | Treatment 2<br>N=xx | Treatment 3 N=xx | Treatment 4<br>N=xx | Treatment 5<br>N=xx | Treatment 6 |
|---|---|---|---|---|---|---|
| Stratum (Previously failed | | 14 3737 | 14 2727 | 14 222 | 14 7/77 | 14 373 |
| n | XX | XX | XX | XX | XX | XX |
| csDMARD only | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 bDMARD | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 bDMARD | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Baseline Anti-CCP Status | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Positive | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Negative | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Missing | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Baseline RF Status | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Positive | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Negative | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Missing | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Baseline Anti-CCP and RF S | tatus | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| At Least one Positive | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Both Negative | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: Time since RA diagnosis and start of RA symptoms is calculated up to date of first study medication administration.
[1] Stratum information is obtained from IWRS.


Example: POP\_T5
Protocol: 201791

Population: Intent-to-Treat

# Table 1.x Summary of Cardiovascular Risk Factors

Age group: xxxxxx

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| History of Tobacco Use | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Never smoked | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Current Smoker | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Former Smoker | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Unknown | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| If former smoker: Time between last | | | | | | |
| smoking and assessment date (years) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | XXX | XXX | XXX | XXX | XXX | XXX |
| Max. | XXX | XXX | xxx | XXX | XXX | xxx |
| Family history of cardiovascular | | | | | | |
| risk factors [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Unknown | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Angina Pectoris | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Current | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Past | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No Medical History | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: [1] Family history of premature coronary artery disease in women <65 years or men < 55 years in first degree relatives only.

Example: POP\_T5 (continued)
Protocol: 201791


Population: Intent-to-Treat

Table 1.x Summary of Cardiovascular Risk Factors

| And aroun: yyyyyy | Summary Of | Cardiovascura | IL KISK FACTOL | 5 | | |
|---|---|---|---|---|---|---|
| Age group: xxxxxx | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment 6 |
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Diabetes mellitus | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Current | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Past | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No Medical History | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Hyperlipidemia | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Current | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Past | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No Medical History | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Hypertension | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Current | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Past | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No Medical History | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Myocardial Infarction | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Current | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Past | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No Medical History | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Stroke | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Current | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Past | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| No Medical History | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: [1] Family history of premature coronary artery disease in women < 65 years or men < 55 years in first degree relatives only.


Example: POP\_T6
Protocol: 201791

Population: Intent-to-Treat

Table 1.x Summary of RA Concomitant Medications

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment 6 |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| ANY MEDICATION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| DMARDs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Methotrexate | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other csDMARDs (not methotrexate) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| csDMARDs >1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| bsDMARDs/boDMARDs/tsDMARDs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Corticosteroids | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Oral | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Intra-Articular | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other RA medications | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: Concomitant medication is defined as any medication taken after the first dose of study treatment, regardless of whether it was started prior to the first dose of study treatment or not.

Note: For subjects that discontinued treatment, medications taken after the date of treatment discontinuation up to the end of safety follow up are also presented in this table.


Example: POP\_T7
Protocol: 201791

Population: Intent-to-Treat

Table 1.x Summary of RA Prior Medications

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 |
|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx |
| ANY MEDICATION | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| DMARDs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Methotrexate | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other csDMARDs (not methotrexate) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| csDMARDs >1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| bsDMARDs/boDMARDs/tsDMARDs | | | | |
| >=1 of bs/bo/tsDMARDs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| =1 of bs/bo/tsDMARDs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 of bs/bo/tsDMARDs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| <pre>Inadequate response to &gt;=1 bs/boDMARD</pre> | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| <pre>Inadequate response to &gt;=1 tsDMARD</pre> | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Inadequate response to >1 bs/bo/tsDMARD | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Oral corticosteroids | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other RA medications | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: Prior medication is defined as any medication that started before first dose of study treatment.

Example: POP\_T8
Protocol: 201791

Page 1 of n Population: Intent-to-Treat

Table 1.x Summary of RA Medications taken at Baseline (Day 1)

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=XX | N=xx | N=xx | N=xx | N=xx | N=xx |
| Methotrexate | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Other csDMARDs (not methotrexate) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| csDMARDs >1 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Methotrexate dose at baseline | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| No Methotrexate | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| <10mg/week | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >=10mg/week | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Methotrexate dose at baseline (mg/week) | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | XXX | XXX | XXX | XXX | XXX | XXX |
| Max. | XXX | xxx | XXX | xxx | XXX | XXX |
| Corticosteroids [1] | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Corticosteroid dose at baseline (mg/day) [1] | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Min. | XXX | XXX | XXX | XXX | XXX | XXX |
| Max. | XXX | XXX | XXX | XXX | XXX | XXX |

201791


Example: POP\_T9
Protocol: 201791
Population: Intent-to-Treat

Table 1.x Summary of Concomitant COVID-19 Vaccines

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=XX |
| Any Medication | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| PFIZER BIONTECH COVID-19 VACCINE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| MODERNA COVID-19 VACCINE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Example: POP\_T10
Protocol: 201791
Population: Safety


Table 1.x Summary of Exposure to Study Treatment

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Duration of drug exposure | [injections] (days) | | | | | |
| Period 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | xx | xx | XX | XX | XX | XX |
| Period 2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | xx | xx | XX | XX | XX | XX |
| Period 1+2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

Example: POP\_T10 (cntd.)
Protocol: 201791
Population: Safety


Table 1.x Summary of Exposure to Study Treatment

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Number of injections | | | | | | |
| Period 1 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |
| Period 2 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |
| Period 1+2 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | xx | XX | XX | XX | XX | XX |

Example: POP\_T10 (cntd.)
Protocol: 201791
Population: Safety


Table 1.x Summary of Exposure to Study Treatment

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment 6 |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Number of injections | | | | | | |
| Period 1+2 | | | | | | |
| 1 - 12 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 13 - 24 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 25 - 40 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| > 40 | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Number of missed injections | | | | | | |
| Period 1 | | | | | | |
| 0 missed injections | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 missed injection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 missed injection | xx (xx% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Period 2 | | | | | | |
| 0 missed injections | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 missed injection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 missed injection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Period 1+2 | | | | | | |
| 0 missed injections | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 1 missed injection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >1 missed injection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

201791

Example: POP\_T10 (cntd.)
Protocol: 201791
Population: Safety


Table 1.x Summary of Exposure to Study Treatment

| · | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment 6 |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=XX |
| Duration of drug exposure [capsu] | esl (davs) | | | | | |
| Period 1 | - , _ , | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | xx | xx | xx | XX | xx |
| Period 2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | xx | xx | xx | XX | xx |
| Period 1+2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

Example: POP\_T10 (cntd.)
Protocol: 201791
Population: Safety


Table 1.x Summary of Exposure to Study Treatment

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment ( |
|---|---|---|---|---|---|---|
| | N=XX | N=xx | N=XX | N=xx | N=xx | N=xx |
| Number of capsules | | | | | | |
| Period 1 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |
| Period 2 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | XX | xx | XX | xx | xx | XX |
| Period 1+2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | xx | XX | XX | XX | XX | XX |

Example: POP\_T11
Protocol: 201791
Population: Safety


Table 1.x
Summary of Overall Compliance Based on Exposure

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Percent Overall Compliance [inje | ections] | | | | | |
| Period 1 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | xx | XX | XX | XX | XX | XX |
| Period 2 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | xx | XX | XX | XX | XX | XX |
| Period 1+2 | | | | | | |
| n | xx | XX | XX | XX | XX | XX |
| Mean | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | xx | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

201791

Example: POP T11 (cntd.)


Population: Safety

Table 1.x Summary of Overall Compliance Based on Exposure

| | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx | Treatment 5<br>N=xx | Treatment<br>N=xx |
|---|---|---|---|---|---|---|
| ) | | | | | | |
| Overall Compliance Categori | es [Injections] | | | | | |
| Period 1 | | | | | | |
| <80% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 80-105% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >105% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Period 2 | | | | | | |
| <80% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| 80-105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| >105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| Period 1+2 | | | | | | |
| <80% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| 80-105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| >105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |

201791

Example: POP T11 (cntd.)

Population: Safety

Table 1.x
Summary of Overall Compliance Based on Exposure

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Percent Overall Compliance [capsules] | | | | | | |
| Period 1 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |
| Period 2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |
| Period 1+2 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min. | XX | XX | XX | XX | XX | XX |
| Max. | XX | XX | XX | XX | XX | XX |

201791

Example: POP T11 (cntd.)


Population: Safety

Table 1.x Summary of Overall Compliance Based on Exposure

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5 | Treatment |
|---|---|---|---|---|---|---|
| | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Overall Compliance Categori | es [capsules] | | | | | |
| Period 1 | - | | | | | |
| <80% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| 80-105% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| >105% | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Period 2 | | | | | | |
| <80% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| 80-105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| >105% | xx(xx% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| Period 1+2 | | | | | | |
| <80% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| 80-105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| >105% | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |

201791

Example: POP\_T11 (cntd.)
Protocol: 201791

Protocol: 201791
Population: Safety


| | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx | Treatment 5<br>N=xx | Treatment 6<br>N=xx |
|---|---|---|---|---|---|---|
| Overall Compliance (inject | ions and sangulas! >-90% | | | | | |
| Overall Compliance [inject Period 1 | .ions and capsules; >-ou* | | | | | |
| Yes | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| | , , | , | , , | , , | , , | , , |
| No | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Period 2 | | | | | | |
| Yes | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| No | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| Period 1+2 | | | | | | |
| Yes | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |
| No | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) | xx(xx%) |

201791

Example: POP\_T12
Protocol: 201791


Population: Intent-to-Treat

Table 1.x Summary of Neuropathic Pain Component as Identified by the Pain DETECT Questionnaire

| | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx | Treatment 5<br>N=xx | Treatment 6<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|---|---|
| creening Result | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Neuropathic | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| Nociceptive | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |
| Unclear | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx% |

201791

Example: EFF T1


Population: Intent-To-Treat

Table 2.x

Summary and Analysis of the Proportion of Subjects Achieving [ACR20/CDAI-LDA/...] at Each Assessment Visit

Visit: Week X

| Statistic | Pooled PBO (N=xx) | OTI 90mg QW (N=xx) | OTI 150mg QW (N=xx) | TOFA 5mg BID (N=xx) | PBO to OTI<br>90mg QW<br>(N=xx) | PBO to OTI<br>150mg QW<br>(N=xx) | PBO to TOFA 5mg BID (N=xx) |
|---|---|---|---|---|---|---|---|
| %Responders | XX • X | XX . X | XX • X | XX.X | | | |
| SE %Responders | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| Difference vs.<br>Pooled PBO (%) | | XX.X | XX.X | XX.X | | | |
| 95% CI (%) | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | | | |
| Difference vs. | xx.x | xx.x | xx.x | | | | |
| 95% CI (%) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | | | | |
| Odds Ratio vs. | | xx.x | xx.x | xx.x | | | |
| 95% CI (%)<br>p-value | | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | | | |
| Odds Ratio vs.<br>TOFA | xx.x | xx.x | xx.x | xx.x | | | |
| 95% CI (%)<br>p-value | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | | | |

Note: All estimates are produced following multiple imputation specified for the [primary estimand/supplemental estimand 1/supplemental estimand 2].

Note: Positive differences and Odds Ratios >1 indicate an improvement of treatment over placebo or tofacitinib.

Note: 95% confidence intervals for the difference to placebo and tofacitinib are constructed using asymptotic Wald confidence limits without correction.

Note: Odds Ratios and corresponding 95% confidence intervals for odds ratios are generated from the logistic regression model adjusted for [Baseline Value], Treatment Group and Previously Failed Medication Category.

Note: Placebo switch treatment arms will only be displayed after Week 12.

Example: EFF\_T2


Population: Intent-To-Treat

Parameter: XXX [optional]

| | Pooled PBO | OTI 90mg QW (N=xx) | OTI 150mg QW (N=xx) | TOFA 5mg BID (N=xx) | PBO to OTI<br>90mg QW<br>(N=xx) | PBO to OTI<br>150mg QW<br>(N=xx) | PBO to TOFA |
|---|---|---|---|---|---|---|---|
| | (N=xx) | | | | (11 1111) | . , | (N=xx) |
| Week 1 | | | | | | | |
| N | XX | XX | XX | XX | | | |
| n(%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | | | |
| Week 2 | | | | | | | |
| N | XX | XX | XX | XX | | | |
| n(%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | | | |
| Week 3 | | | | | | | |
| N | XX | XX | XX | XX | | | |
| n(%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | | | |
| Week 13 | | | | | | | |
| N | | XX | XX | XX | XX | XX | XX |
| n (%) | | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: N is the number of subjects with non-missing data at that visit

201791

Example: EFF T3


Population: Intent-To-Treat

Table 2.x

Analysis of Change from Baseline in [HAQ-DI/CDAI Total/...] at Each Assessment Visit [(Primary Estimand)]

| Visit: | Week | Χ |
|--------|------|---|
|--------|------|---|

| Statistic | Pooled PBO (N=xx) | OTI 90mg QW (N=xx) | OTI 150mg QW (N=xx) | TOFA 5mg BID (N=xx) | PBO to OTI<br>90mg QW<br>(N=xx) | PBO to OTI<br>150mg QW<br>(N=xx) | PBO to TOFA 5mg BID (N=xx) |
|---|---|---|---|---|---|---|---|
| LS Mean Change | xx.x | XX.X | XX.X | XX.X | | | |
| Standard Error | XX.XX | XX.XX | XX.XX | XX.XX | | | |
| LS Mean Difference<br>from Pooled PBO | | xx.x | xx.x | xx.x | | | |
| 95% CI<br>p-value | | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | | | |
| LS Mean Difference from TOFA | xx.x | XX.X | XX.X | | | | |
| 95% CI<br>p-value | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | | | | |

Note: All estimates are produced following multiple imputation specified for the [primary estimand/supplemental estimand 1/supplemental estimand 2]

Note: All estimates are obtained from an ANCOVA analysis adjusted for Baseline Value, Treatment Group and Previously Failed Medication Category.

Note: Placebo switch treatment arms will only be displayed after Week 12.

201791

Example: EFF T4


Population: Intent-To-Treat

Table 2.x

Summary of Observed [Result/Change from Baseline] in [HAQ-DI/CDAI Total/...] at Each Assessment Visit

Parameter: XXXX [optional]

| Treatment | Visit | n | Mean | SD | 95% CI | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|
| Pooled PBO (N=xx) | Baseline | XX | XX.X | XX.XX | (xx.x,xx.x) | XX.X | XX | XX |
| | Week 1 | XX | XX.X | XX.XX | (xx.x,xx.x) | XX.X | XX | XX |
| TI 90mg QW<br>N=xx) | Baseline | XX | xx.x | xx.xx | (xx.x,xx.x) | xx.x | xx | XX |
| | Week 1 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | Week 13 | XX | XX.X | XX.XX | (xx.x,xx.x) | XX.X | XX | XX |
| | Week 16 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | ••• | | | | | | | |
| BO to OTI 90mg QW<br>N=xx) | Baseline | xx | XX.X | xx.xx | (xx.x,xx.x) | xx.x | xx | XX |
| | Week 13 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | Week 16 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | | | ••• | | | | | ••• |
| • | | | | | | | | |

Example: EFF\_T5

Population: Intent-To-Treat

Table 2.x

Summary of Ratio to Baseline in [CRP] at Each Assessment Visit (Log Transformed)

Parameter: XXXX

| Treatment | Visit | n | Geometric Mean | %CVb | 95% CI | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|
| Pooled PBO (N=xx) | Baseline | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | Week 1 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | | | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| OTI 90mg QW (N=xx) | Baseline | XX | XX.X | xx.xx | (xx.x,xx.x) | XX.X | XX | XX |
| | Week 1 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | | | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | Week 13 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | | | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | Week 16 | XX | xx.x | XX.XX | (xx.x,xx.x) | XX.X | XX | XX |
| | | | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| PBO to OTI 90mg<br>QW (N=xx) | Baseline | XX | XX.X | XX.XX | (xx.x,xx.x) | xx.x | XX | xx |
| | Week 13 | XX | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | | | XX.X | XX.XX | (xx.x, xx.x) | XX.X | XX | XX |
| | Week 16 | xx | xx.x | xx.xx | (xx.x, xx.x) | xx.x | XX | XX |

201791

Example: EFF\_T6
Protocol: 201791 Confidential
Population: Intent-To-Treat Page 1 of n

Table 2.x Summary of Observed [ACR20] Response Within 4/8/12/16/24/>24 Weeks Post Baseline

| Achieved Response | Pooled PBO (N=xx) | OTI 90mg QW<br>(N=xx) | OTI 150mg QW (N=xx) | TOFA 5mg BID (N=xx) |
|---|---|---|---|---|
| Within 4 weeks | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Within 8 weeks n(%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Within 12 weeks n(%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Within 16 weeks n(%) | | xx (xx%) | xx (xx%) | xx (xx%) |
| Within 24 weeks n(%) | | xx (xx%) | xx (xx%) | xx (xx%) |
| Within >24 weeks n(%) | | xx (xx%) | xx (xx%) | xx (xx%) |

201791

Example: EFF T7


Population: Intent-To-Treat

| Maintained Response | OTI 90mg QW<br>(N=xx) | OTI 150mg QW (N=xx) | TOFA 5mg BID (N=xx) |
|---|---|---|---|
| For 12 weeks n(%) | xx (xx%) | xx (xx%) | xx (xx%) |
| For 24 weeks n(%) | xx (xx%) | xx (xx%) | xx (xx%) |
| For 36 weeks n(%) | xx (xx%) | xx (xx%) | xx (xx%) |

Note: If a subject has at most two non-consecutive visits with missing response data within the 12 week window after first occurrence of response and the subject was in response for all other visits, then the subject will be considered to have maintenance of response.

201791

Example: EFF T8


Population: Intent-To-Treat

Table 2.x
Analysis of Time to Onset of [ACR20] Response

| | OTI 90mg QW | OTI 150mg QW | TOFA 5mg BID |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| Jumber of Subjects | | | |
| n | XX | XX | XX |
| Endpoint (ACR20) | xx (xx%) | xx (xx%) | xx (xx%) |
| Censored | xx (xx%) | xx (xx%) | xx (xx%) |
| Early Study Withdrawal | xx (xx%) | xx (xx%) | xx (xx%) |
| Study Completion | xx (xx%) | xx (xx%) | xx (xx%) |
| Estimate for Time to ACR20 (Weeks) [1] 1 <sup>st</sup> Quartile Median 3 <sup>rd</sup> Quartile | xx.x<br>xx.x<br>xx.x | xx.x<br>xx.x | xx.x<br>xx.x<br>xx.x |
| Adjusted Hazard Ratio [2] | | | |
| Estimate | X.XX | X.XX | X.XX |
| 95% CI | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| p-value | 0.xxx | 0.xxx | 0.xxx |
| Estimate for Time to ACR20 (Weeks) [3] | | | |
| 1 <sup>st</sup> Quartile | XX.X | XX.X | xx.x |
| Median | XX.X | XX.X | xx.x |
| 3 <sup>rd</sup> Quartile | XX.X | XX.X | XX.X |

<sup>[1]</sup> Statistics will be missing when the number of events is too low to estimate the values from the survival function.

<sup>[2]</sup> A hazard ratio <1 indicates a lower risk with this treatment compared with tofacitinib. Hazard Ratio is adjusted for [Baseline Value] and Previously Failed Medication Category.

<sup>[3]</sup> Among subjects achieving response.

201791

Example: EFF F1


Population: Intent-to-Treat

Figure 2.x Proportion of Subjects Achieving [ACR20/50/70 Response] at Each Assessment Visit [(Primary Estimand)]



Note: All estimates are produced following multiple imputation specified for the [primary estimand/supplemental estimand 1/supplemental estimand 2]
201791

Example: EFF F2


Population: Intent-to-Treat

Figure 2.x

Plot of Least Squares Means of Change from Baseline in [HAQ-DI/CDAI Total Score/...] at Each Assessment Visit [(Primary Estimand)]



Note: All estimates are produced following multiple imputation specified for the [primary estimand/supplemental estimand 1/supplemental estimand 2]

Note: All estimates are obtained from an ANCOVA analysis adjusted for Baseline Value, Treatment Group and Previously Failed Medication Category.

Example: EFF F3


Population: Intent-to-Treat

Figure 2.x

Spydergram of Individual Domain Scores of SF-36 at Each Assessment Visit

Visit: Week 12



Note: PF=Physical Functioning, RP=Role Physical, BP=Bodily Pain, GH=General Health, VT=Vitality, SF=Social Function, RE=Role Emotional, MH=Mental Health. Note: Values presented are the 0-100 score for each domain.

Note: Baseline presented at each visit as the mean baseline value for each component independent of treatment group.

Example: EFF F4


Population: Intent-to-Treat

Figure 2.x

Forest Plot of [Demographic] Subgroup Results for [ACR20] - Comparison to [Placebo at Week 12]

#### Treatment: OTI 90mg QW

| Subgroup | Pooled PBO<br>% Responders (SE<br>(N=78) | OTI 90mg QW<br>) % Responders (SE<br>(N=157) | OR (95% CI)<br>) | |
|---|---|---|---|---|
| OVERALL | 48.3 (6.01) | 43.1 (4.18) | 0.8 (0.5, 1.5) | <b>├</b> ─ <del> </del> |
| Region | | | | |
| USA and Canada (n=82) | 45.0 (9.30) | 25.6 (6.85) | 0.4 (0.1, 1.2) | <b>├</b> ─── <b>┤</b> |
| Europe (n=85) | 39.5 (9.83) | 45.3 (6.82) | 1.4 (0.5, 3.8) | <del> - </del> |
| Latin America and South Africa (n=51) | 71.8 (12.27) | 66.8 (8.29) | 0.7 (0.1, 2.9) | H |
| Asia (n=17) | 37.5 (26.52) | 38.5 (13.49) | 0.7 (0.0, 12.7) | <del></del> |
| Specific Region (USA, other) | | | | |
| USA (n=81) | 46.5 (9.49) | 25.6 (6.85) | 0.4 (0.1, 1.1) | <del> </del> |
| Other (n=154) | 49.3 (7.68) | 51.4 (5.04) | 1.2 (0.6, 2.5) | <del></del> |
| Specific Region (Europe, other) | | | | |
| Europe (n=85) | 39.5 (9.83) | 45.3 (6.82) | 1.4 (0.5, 3.8) | <del></del> |
| Other (n=150) | 53.0 (7.44) | 41.7 (5.29) | 0.6 (0.3, 1.3) | <del></del> |
| Specific Region (Japan, other) | | | | |
| Japan (n=14) | 37.5 (26.52) | 40.0 (15.49) | 0.6 (0.0, 13.3) | l |
| Other (n=221) | 48.8 (6.14) | 43.3 (4.34) | 0.8 (0.4, 1.5) | <del></del> |
| | | | | 0.1 1 10 |

Note: Odds Ratios (OR) >1 indicate an improvement of treatment over [placebo].

Note: All estimates are produced following multiple imputation specified for the primary estimand.

Note: Odds Ratios and corresponding 95% confidence intervals for odds ratios are generated from the logistic regression model adjusted for [Baseline Value], Treatment Group and Previously Failed Medication Category.

Example: EFF\_F5


Population: Intent-to-Treat

Figure 2.x

Forest Plot of [Demographic] Subgroup Results for Change from Baseline in [HAQ-DI] - Comparison to [Placebo at Week 12]

#### Treatment: OTI 90mg QW

| Subgroup | Pooled PBO<br>LSM (SE)<br>(N=78) | OTI 90mg QW<br>LSM (SE)<br>(N=155) | Diff (95% CI) | |
|---|---|---|---|---|
| OVERALL | -0.4 (0.06) | -0.4 (0.04) | 0.0 (-0.14, 0.16) | H |
| Region | | | | |
| USA and Canada (n=81) | -0.3 (0.10) | -0.3 (0.08) | 0.0 (-0.29, 0.23) | $\vdash$ |
| Europe (n=85) | -0.4 (0.09) | -0.4 (0.07) | -0.1 (-0.27, 0.17) | H |
| Latin America and South Africa (n=50) | -0.8 (0.17) | -0.6 (0.11) | 0.2 (-0.18, 0.59) | H |
| Asia (n=17) | 0.0 (0.21) | -0.1 (0.11) | -0.1 (-0.55, 0.37) | <del></del> |
| Specific Region (USA, other) | | | | |
| USA (n=80) | -0.3 (0.11) | -0.3 (0.08) | 0.0 (-0.26, 0.26) | $\vdash$ |
| Other (n=153) | -0.4 (0.08) | -0.4 (0.05) | 0.0 (-0.17, 0.19) | <del> </del> |
| Specific Region (Europe, other) | | | | |
| Europe (n=85) | -0.4 (0.09) | -0.4 (0.07) | -0.1 (-0.27, 0.17) | H |
| Other (n=148) | -0.4 (0.08) | -0.4 (0.06) | 0.0 (-0.16, 0.23) | $\vdash$ |
| Specific Region (Japan, other) | | | | |
| Japan (n=14) | 0.0 (0.18) | -0.1 (0.11) | -0.1 (-0.48, 0.33) | <del></del> |
| Other (n=219) | -0.4 (0.07) | -0.4 (0.05) | 0.0 (-0.14, 0.17) | $\vdash$ |
| | | | -1.5 -1.0 | 0 -0.5 0.0 0.5 1.0 1.5 |

Note: LSM= Least Squares Means, SE= Standard Error.

Note: All estimates are produced following multiple imputation specified for the primary estimand.

Note: All estimates are obtained from an ANCOVA analysis adjusted for Baseline Value, Treatment Group and Previously Failed Medication Category.

Example: EFF F6


Population: Intent-to-Treat

Figure 2.x Proportion of Subjects Achieving Maintained [ACR50 Response] for At Least 12/24/36 Weeks After the First Occurrence



Note: If a subject has at most two non-consecutive visits with missing response data within the 12 week window after first occurrence of response and the subject was in response for all other visits, then the subject will be considered to have maintenance of response.

201791

Example: EFF F7


Population: Intent-to-Treat

Figure 2.x

Cumulative Probability Plots of Individual Subject Changes from Baseline in [mTSS] at Each Assessment Visit



Example: BIOM T1


Population: Intent-to-Treat

Table 5.x

Summary of Observed [Result/Change from Baseline] in [Pharmacodynamic Biomarkers/...] at Each Assessment Visit

Parameter: XXXX

| Treatment | Visit | n | Mean | SD | Median | (Q1, Q3) | Min | Max |
|---|---|---|---|---|---|---|---|---|
| Pooled PBO (N=xx) | Baseline | XX | XX.X | XX.XX | XX.X | (xx.x, xx.x) | XX | XX |
| | Week 1 | XX | XX.X | XX.XX | XX.X | (xx.x,xx.x) | XX | XX |
| OTI 90mg QW (N=xx) | Baseline | xx | XX.X | xx.xx | xx.x | (xx.x,xx.x) | xx | XX |
| | Week 1 | XX | XX.X | XX.XX | XX.X | (xx.x, xx.x) | XX | XX |
| | Week 13 | XX | XX.X | XX.XX | XX.X | (xx.x,xx.x) | XX | XX |
| | Week 16 | XX | XX.X | XX.XX | XX.X | (xx.x,xx.x) | XX | XX |
| PBO to OTI 90mg QW (N=xx) | Baseline | xx | XX.X | xx.xx | xx.x | (xx.x, xx.x) | XX | XX |
| | Week 13 | XX | XX.X | XX.XX | XX.X | (xx.x, xx.x) | XX | XX |
| | Week 16 | XX | XX.X | XX.XX | XX.X | (xx.x, xx.x) | XX | XX |

Note: Values reported below lower limit of quantification were replaced by one-half the limit of quantification.

Example: BIOM\_T2


Population: Intent-to-Treat

Table 5.x

Repeated Measures Analysis of Change from Baseline in Pharmacodynamic Biomarkers at Each Assessment Visit ([Placebo/Tofacitinib] Comparison)

Biomarker: [Chemokine (C-C Motif) Ligand 17]

Visit: Week 1

| Statistic | Pooled PBO<br>N=xx | OTI 90mg QW<br>N=xx | OTI 150mg QW<br>N=xx | TOFA 5mg BID<br>N=xx |
|---|---|---|---|---|
| n [1] | XX | xx | xx | XX |
| LS Mean Change | XX.X | XX.X | XX.X | XX.X |
| Standard Error | XX.XX | XX.XX | XX.XX | XX.XX |
| LS Mean Difference from Pooled PBO | | xx.x | xx.x | xx.x |
| 95% CI<br>p-value | | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx | (xx.x, xx.x)<br>0.xxxx |

<sup>[1]</sup> Number of subjects with analysable data at the given timepoint.

Note: All estimates are obtained from an MMRM analysis adjusted for Baseline Value, Treatment Group, Previously Failed Medication Category, Visit and Treatment Group by Visit.

201791

Example: BIOM T3


Population: Intent-to-Treat

#### Table 5.x

Repeated Measures Analysis of Change from Baseline in Pharmacodynamic Biomarkers at Each Assessment Visit ([Placebo/Tofacitinib] Comparison) (Log Transformed)

Biomarker: [Chemokine (C-C Motif) Ligand 17]

Visit: Week 1

| Statistic | Pooled PBO<br>N=xx | OTI 90mg QW<br>N=xx | OTI 150mg QW<br>N=xx | TOFA 5mg BID<br>N=xx |
|---|---|---|---|---|
| n [1] | xx | xx | xx | xx |
| LS Geometric Mean | XX.X | XX.X | XX.X | xx.x |
| %CVb | XX.XX | XX.XX | XX.XX | XX.XX |
| Ratio to Pooled PBO | | XX.X | XX.X | XX.X |
| 95% CI | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| p-value | | 0.xxxx | 0.xxxx | 0.xxxx |

<sup>[1]</sup> Number of subjects with analysable data at the given timepoint.

Note: All estimates are obtained from an MMRM analysis adjusted for Baseline Value, Treatment Group, Previously Failed Medication Category, Visit and Treatment Group by Visit.

201791


Example: AE13 (modified)
Protocol: 201791
Population: Safety

Table 3.x Overall Summary of Adverse Events (Period X)

| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 |
|---|---|---|---|---|
| | N=xx | N=XX | N=XX | N=xx |
| ny AE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs related to study treatment | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs leading to discontinuation of study treatment only | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs leading to discontinuation of background therapy only | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs leading to discontinuation of both study treatment and background therapy | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs leading to dose interruption/delay of study treatment | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs leading to dose interruption/delay of background therapy | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| AEs leading to dose reduction of background therapy | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| ny SAE | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| SAEs related to study treatment | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Fatal SAEs | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Fatal SAEs related to study treatment | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| ny SAE excluding COVID-19 Infections | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| SAEs excluding COVID-19 Infections related to study treatment | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Fatal SAEs excluding COVID-19<br>Infections | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Fatal SAEs excluding COVID-19<br>Infections related to study treatment | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

201791

Example: SAFE T1 Protocol: 201791


Table 3.x Summary of Exposure Adjusted Event Rates per 100 years for All Adverse Events (Period X)

| System Organ Class<br>Preferred Term | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx |
|---|---|---|---|---|
| Total Treatment Exposure (person-years) | xx.xx | xx.xx | xx.xx | xx.xx |
| Any Adverse Event | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Infections and Infestations | | | | |
| Any Adverse Event | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Nasopharyngitis | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Upper Respiratory Tract | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Infection | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Bronchitis | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Pharyngitis | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Rhinitis | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Oral Herpes | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |
| Viral Infection | xx.x [xx] | xx.x [xx] | xx.x [xx] | xx.x [xx] |

Note: The rate and number of events "Rate [#]" are reported in this table. #= Number of events.

Note: Rate is event rate per 100 person-years, calculated as the number of events multiplied by 100, divided by the total treatment exposure in years.

201791

Example: SAFE\_T2
Protocol: 201791
Population: Safety


Table 3.x Summary of Adverse Events of Special Interest (AESI) (Period X)

| | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx | Treatment 5<br>N=xx | Treatment 6<br>N=xx |
|---|---|---|---|---|---|---|
| | n (%) [#] | n (%) [#] | n (%) [#] | n (%) [#] | n (%) [#] | n (%) [#] |
| Any AESI | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Serious infections | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Serious infections excluding COVID-19 Infections | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic infections | x(x)[x] | x (x) [x] | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Active TB | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Latent TB | x (x) [x] | x(x)[x] | x (x) [x] | x(x)[x] | x(x)[x] | x(x)[x] |
| TB reactivation | x (x) [x] | x(x)[x] | x (x) [x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Neutropenia | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Persistent cough | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Persistent dyspnoea | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Pulmonary alveolar proteinosis | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Serious Hypersensitivity reactions | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Injection site reaction | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences.

Note: Persistent cough or persistent dyspnoea defined as a cough (CTACE Grade  $\geq$  2) or a dyspnoea (dyspnoea scale Grade  $\geq$  2) for three consecutive weeks ( $\geq$ 21 days).

Note: Neutropenia is defined as AEs/SAEs of neutropenia where the corresponding absolute neutrophil counts are grade 3 or 4 ( $<1.0 \times 10^{9}/L$ ).

Note: Opportunistic infections, Active TB, Latent TB, TB reactivation events, serious hypersensitivity reactions and pulmonary alveolar proteinosis have been adjudicated and only adjudicated events displayed in the summary table.

Example: SAFE T3 Protocol: 201791


Table 3.x

| Samulary or o | - | Adverse Events | | The state of the s |
|---|---|---|---|---|
| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 |
| | N=xx | N=xx | N=xx | N=xx |
| | n (%) [#] | n (%) [#] | n (%) [#] | n (%) [#] |
| Any Other Important AEs | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Adjudicated GI Perforation | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Adjudicated CV Events | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| CV Death | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Myocardial Infarction | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hospitalisation for Unstable Angina | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Stroke | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hospitalisation for Heart Failure | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Deep Vein Thrombosis | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Pulmonary Embolism | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Any Malignancy | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Solid, Excluding Non-melanoma Skin Cancer | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Non-melanoma Skin Cancer | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hematologic | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Lymphoma | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: A subject can have an event in more than one category.

Note: Fatal CV events are captured in two categories, respective CV category and CV death.

201791

Example: SAFE T3 (continued)

Protocol: 201791 Population: Safety

Page 2 of n Table 3.x

| Summary of | Other Important | Adverse Events | s (Period X) | |
|---|---|---|---|---|
| | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 |
| | N=xx<br>n (%) [#] | N=xx<br>n (%) [#] | N=xx<br>n (%) [#] | N=xx<br>n (%) [#] |
| Any malignancy, Excluding Non-melanoma Skin<br>Cancer | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Any Herpes Infection | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Herpes Zoster | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Herpes Simplex | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Non-Specific Herpes Infection | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| All-Cause Mortality | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Serious Pulmonary Infections | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Serious Pulmonary Infections excluding COVID-19 Infections | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Pneumonia (Serious and Non-Serious) | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Pneumonia (Serious and Non-Serious) excluding COVID-19 Infections | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hepatitis B and Hepatitis B Reactivation | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Thromboembolic Events | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences.

Note: A subject can have an event in more than one category.

Note: Fatal CV events are captured in two categories, respective CV category and CV death.

Example: SAFE T4 Protocol: 201791


Table 3.x Summary of Adjudicated Cardiovascular Event Categories (Period X)

| | Treatment 1<br>N=xx<br>n (%) [#] | Treatment 2<br>N=xx<br>n (%) [#] | Treatment 3<br>N=xx<br>n (%) [#] | Treatment 4 N=xx n (%) [#] |
|---|---|---|---|---|
| ny Adjudicated CV Event | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| MACE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Broad MACE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| VTE (DVT and/or PE) | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| DVT only | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| PE only | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| | | | | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences.

Note: MACE=Major Adverse Cardiovascular Event, DVT=Deep Vein Thrombosis, PE= Pulmonary Embolism, VTE=Venous

Thromboembolism.

Note: MACE is defined reported as the following categories - CV death, non-fatal MI and non-fatal stroke.

Note: Broad MACE is defined as reported as the following categories - CV death, MI, hospitalisation for unstable angina,

stroke and hospitalisation for heart failure. A CV event resulting in death is reported as one MACE event.

201791

Example ESI1 (modified)


Period: Period X

| | Treatment 1 (N=100) | | Treatment 2 (N=100) | | Treatment 3 (N=100) | |
|---|---|---|---|---|---|---|
| Number of Subjects with the Event | | (50%) | 40 | (40%) | 40 | (40%) |
| Number of Events | 60 | | 65 | | 55 | |
| Event Characteristics (% based on all subjects)[1] | | | | | | |
| Serious | 10/100 | (10%) | 16/100 | (16%) | 8/100 | (8%) |
| Study treatment related | 25/100 | (25%) | 10/100 | (10%) | 20/100 | (20%) |
| Led to study withdrawal | 5/100 | (5%) | 4/100 | (4%) | 2/100 | (2%) |
| Event Characteristics (% based on subjects with the Event)[1] | | | | | | |
| Serious | 10/50 | (20%) | 16/40 | (40%) | 8/40 | (20%) |
| Study treatment related | 25/50 | (50%) | 10/40 | (25%) | 20/40 | (50%) |
| Led to study withdrawal | 5/50 | (10%) | 4/40 | (10%) | 2/40 | (5%) |

Note: [1] Subjects may be included in more than one category for 'Event Characteristics'.

Note: [2] Outcome worst case hierarchy: Fatal > Not Recovered/Not Resolved > Recovered/Resolved with sequelae > Recovering/Resolving > Recovered/Resolved

Note: [3] Subjects are counted once under each action that was taken.

201791

Example ESI1 (modified)


Population: Safety

 $\label{eq:Table 3.x} \textbf{Summary of Characteristics of Injection Site Reaction}$ 

Study: Period X

| | Treatment 1 | Treatment 2 | |
|---|---|---|---|
| | (N=100) | (N=100) | (N=100) |
| Number of occurrences (% based on all subjects) | | | |
| One | 30/100 (309 | %) 20/100 (20 | 0%) 8/100 (8%) |
| Two | 15/100 (15 | %) 10/100 (10 | 0%) 30/100 (30%) |
| Three or more | 5/100 (59 | %) 10/100 (10 | 0%) 2/100 (2%) |
| Number of occurrences (% based on subjects with the Event) | | | |
| One | 30/50 (609 | %) 20/40 (50 | 0%) 8/40 (20%) |
| Two | 15/50 (309 | %) 10/40 (2) | 5%) 30/40 (75%) |
| Three or more | 5/50 (109 | %) 10/40 (2 | 5%) 2/40 (5%) |
| Outcome (% based on all subjects)[2] | | | |
| Recovered/Resolved | 20/100 (209 | %) 10/100 (10 | 0%) 8/100 (8%) |
| Recovering/Resolving | 10/100 (109 | %) 20/100 (20 | 0%) 30/100 (30%) |
| Not Recovered/Not Resolved | 10/100 (109 | %) 5/100 ( | 5%) 0/100 |
| Recovered/Resolved with sequelae | 5/100 (5 | %) 0/100 | 0/100 |
| Fatal | 5/100 (59 | %) 5/100 ( | 5%) 2/100 (2%) |
| Outcome (% based on subjects with the Event)[2] | | | |
| Recovered/Resolved | 20/50 (409 | %) 10/40 (25 <sup>9</sup> | %) 8/40 (20%) |
| Recovering/Resolving | 10/50 (209 | %) 20/40 (50 | %) 30/40 (75%) |
| Not Recovered/Not Resolved | 10/50 (209 | %) 5/40 (13 | %) 0/40 |
| Recovered/Resolved with sequelae | 5/50 (109 | %) 0/40 | 0/40 |
| Fatal | 5/50 (109 | %) 5/40 (13 | %) 2/40 (5%) |

Note: [1] Subjects may be included in more than one category for 'Event Characteristics'.

Note: [2] Outcome worst case hierarchy: Fatal > Not Recovered/Not Resolved > Recovered/Resolved with sequelae > Recovering/Resolving > Recovered/Resolved

Note: [3] Subjects are counted once under each action that was taken.

201791

Example ESI1 (modified)


Period: Period X

| | Treatment 1 (N=100) | Treatment 2 (N=100) | Treatment 3 (N=100) |
|---|---|---|---|
| Maximum Intensity (% based on all subjects) | | | |
| Mild | 30/100 (30%) | 20/100 (20%) | 8/100 (8%) |
| Moderate | 15/100 (15%) | 10/100 (10%) | 30/100 (30%) |
| Severe | 5/100 (5%) | 10/100 (10%) | 2/100 (2%) |
| Maximum Intensity (% based on subjects with the Event) | | | |
| Mild | 30/50 (60%) | 20/40 (50%) | 8/40 (20%) |
| Moderate | 15/50 (30%) | 10/40 (25%) | 30/40 (75%) |
| Severe | 5/50 (10%) | 10/40 (25%) | 2/40 (5%) |

Note: [1] Subjects may be included in more than one category for 'Event Characteristics'.

Note: [2] Outcome worst case hierarchy: Fatal > Not Recovered/Not Resolved > Recovered/Resolved with sequelae > Recovering/Resolving > Recovered/Resolved

Note: [3] Subjects are counted once under each action that was taken.

Example ESI1 (modified)


Population: Safety

Period: Period X

| | Treatment (N=100) | | Treatm<br>(N=1 | | Treatme:<br>(N=10 | |
|---|---|---|---|---|---|---|
| 7 | | | | | | |
| Action Taken (% based on all subjects)[3] | 00/100 /0 | | | | 0/100 | |
| Study treatment withdrawn | 20/100 (2 | / | 10/100 | , , | 8/100 | (8%) |
| Dose not changed | -, , | (5%) | 0/100 | | 0/100 | (00) |
| Dose interrupted/delayed | 0/100 | 100) | 5/100 | ( / | 2/100 | (2%) |
| Not applicable | 5/100 (1 | 10%) | 0/100 | | 0/100 | |
| Action Taken (% based on subjects with the Event)[3] | | | | | | |
| Study treatment withdrawn | 20/50 (4 | 40%) | 10/40 | (25%) | 8/40 ( | 20%) |
| Dose not changed | 5/50 (1 | 10%) | 0/40 | | 0/40 | |
| Dose interrupted/delayed | 0/50 | | 5/40 | (13%) | 2/40 | (5%) |
| Not applicable | 5/50 (1 | 10%) | 0/40 | | 0/40 | |
| Action Taken with Background Therapy(% based on all | | | | | | |
| subjects)[3] [4] | | | | | | |
| Drug withdrawn | 20/100 (2 | 20%) | 10/100 | (10%) | 8/100 | (8%) |
| Dose reduced | 10/100 (1 | 10%) | 20/100 | (20%) | 30/100 | (30%) |
| Dose not changed | 5/100 ( | (5%) | 0/100 | | 0/100 | |
| Dose interrupted/delayed | 0/100 | | 5/100 | (5%) | 2/100 | (2%) |
| Not applicable | 5/100 (1 | 10%) | 0/100 | | 0/100 | |
| Action Taken (% based on subjects with the Event)[3] | | | | | | |
| Background Therapy [4] withdrawn | 20/50 (4 | 40%) | 10/40 | (25%) | 8/40 ( | 20%) |
| Dose reduced | 10/50 (2 | 20%) | 20/40 | (50%) | 30/40 ( | 75%) |
| Dose not changed | 5/50 (1 | 10%) | 0/40 | | 0/40 | |
| Dose interrupted/delayed | 0/50 | - | 5/40 | (13%) | 2/40 | (5%) |
| Not applicable | 5/50 (1 | 10%) | 0/40 | • | 0/40 | • |

Note: [1] Subjects may be included in more than one category for 'Event Characteristics'.

Note: [2] Outcome worst case hierarchy: Fatal > Not Recovered/Not Resolved > Recovered/Resolved with sequelae > Recovering/Resolving > Recovered/Resolved

Note: [3] Subjects are counted once under each action that was taken.

Example: SAFE\_T5
Protocol: 201791
Population: Safety


Table 3.x Summary of Injection Site Reaction (Period X)

| | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3 N=xx | Treatment 4<br>N=xx |
|---|---|---|---|---|
| | n (%) [#] | n (%) [#] | n (%) [#] | n (%) [#] |
| Any injection site reactions | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| <= 1 Day post injection | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| > 1 Day post injection \$ | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Reported as a non-serious AE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Reported as an SAE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Type of Reactions | | | | |
| Itching/Pruritus | x (x) [x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Redness/Erythema | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Pain | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Bruising | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Swelling/Edema | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Warm to Touch | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences. (\$) until 1 day before next injection.

Example: SAFE\_T6
Protocol: 201791
Population: Safety


| | Treatment 1<br>N=xx<br>n (%) [#] | Treatment 2<br>N=xx<br>n (%) [#] | Treatment 3<br>N=xx<br>n (%) [#] | Treatment 4<br>N=xx<br>n (%) [#] |
|---|---|---|---|---|
| Any serious or opportunistic infections | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Reported as a non-serious AE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Reported as an SAE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Type of Infection | | | | |
| Bacterial - Gram Positive | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Bacterial - Gram Negative | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Bacterial - Atypical | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Bacterial - Unknown | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Bacterial - Other | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Viral - Zoster/shingles | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Viral - Simplex, orogenital | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Viral - EBV | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Viral - HCV | x (x) [x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Viral - HBV | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Viral - HBV Reactivation | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Viral - Unknown | x (x) [x] | x (x) [x] | x (x) [x] | x(x)[x] |
| Viral - Other | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences.

Note: \$ until 1 day before next injection.

Note: Adjudication of serious hypersensitivity reactions was done internally.

201791

Example: SAFE T6 (continued)

Population: Safety

Table 3.x
Summary of Serious or Adjudicated Opportunistic Infections (Period X)

| | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3 N=xx | Treatment 4 |
|---|---|---|---|---|
| | n (%) [#] | n (%) [#] | n (%) [#] | n (%) [#] |
| 'ype of Infection | | | | |
| Opportunistic - Esophageal candidiasis | x (x) [x] | x(x)[x] | x(x)[x] | x(x)[x] |
| Opportunistic - CMV viremia | x (x) [x] | x(x)[x] | x(x)[x] | x (x) [x] |
| Opportunistic - CMV invasive | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Opportunistic - Pneumocystis Jiroveci | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Cryptococcus | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Opportunistic - Disseminated herpes zoster | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - BK virus encephalitis | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Opportunistic - Fungal | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Protozoal/helminthic | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Latent tuberculosis | x (x) [x] | x(x)[x] | x(x)[x] | x (x) [x] |
| Opportunistic - Active tuberculosis | x (x) [x] | x(x)[x] | x(x)[x] | x (x) [x] |
| Opportunistic - Atypical mycobacterial | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Aspergillus | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Fungal non aspergillus | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Fungal non cryptococcal | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Unknown | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Opportunistic - Other | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences.

Note: \$ until 1 day before next injection.

Note: Adjudication of serious hypersensitivity reactions was done internally.

201791

Example: SAFE\_T6 (continued)


Population: Safety

Table 3.x Summary of Serious or Adjudicated Opportunistic Infections (Period X)

| | Treatment 1<br>N=xx<br>n (%) [#] | Treatment 2<br>N=xx<br>n (%) [#] | Treatment 3<br>N=xx<br>n (%) [#] | Treatment 4<br>N=xx<br>n (%) [#] |
|---|---|---|---|---|
| Origin of Infection | (*, ["] | (*) ["] | ( * / [ " ] | (*/ ["] |
| Community | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hospital | x(x)[x] | x (x) [x] | x (x) [x] | x (x) [x] |
| ICU | x(x)[x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Unknown | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Parenteral antibiotics or antimicrobial medication administered | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Culture/swab taken | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Diagnostic imaging or other diagnostic tests performed | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Had grade 3 neutropenia or worse at the time of infection | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences.

Note: \$ until 1 day before next injection.

Note: Adjudication of serious hypersensitivity reactions was done internally.

Example: SAFE\_T7
Protocol: 201791
Population: Safety


Table 3.x Summary of Adjudicated Serious Hypersensitivity Reactions (Period X)

| | Treatment 1<br>N=xx<br>n (%) [#] | Treatment 2<br>N=xx<br>n (%) [#] | Treatment 3<br>N=xx<br>n (%) [#] | Treatment 4<br>N=xx<br>n (%) [#] |
|---|---|---|---|---|
| Any serious hypersensitivity reactions | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| <= 1 Day post injection | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| > 1 Day post injection \$ | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Reported as a non-serious AE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Reported as an SAE | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Type of Systemic Reactions | | | | |
| Headache | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Pruritus | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Urticaria | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Rash | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Angioedema | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Fatigue | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Myalgia | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Arthralgia | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Bronchospasm | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hypotension requiring vasopressors | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Hypotension not requiring vasopressors | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Dizziness | x (x) [x] | x (x) [x] | x(x)[x] | x (x) [x] |
| Syncope | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Crampy abdominal pain | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Respiratory failure requiring intubation | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| ICU Management required | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |
| Other | x (x) [x] | x (x) [x] | x (x) [x] | x (x) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences. (\$) until 1 day before next injection.

201791

Example: SAFE\_T7 (continued)
Protocol: 201791

Population: Safety

| | Treatment 1<br>N=xx<br>n (%) [#] | Treatment 2<br>N=xx<br>n (%) [#] | Treatment 3<br>N=xx<br>n (%) [#] | Treatment 4<br>N=xx<br>n (%) [#] |
|---|---|---|---|---|
| Met anaphylaxis criteria | | | | |
| Criterion 1 | x (x) [x] | x (x) [x] | x (x) [x] | x(x)[x] |
| Criterion 2 | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |
| Criterion 3 | x (x) [x] | x (x) [x] | x(x)[x] | x(x)[x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences. (\$) until 1 day before next injection.

Example: SAFE\_T8
Protocol: 201791
Population: Safety


Table 3.x Summary of Pulmonary Findings (Period X)

| Subjects with at least one event of | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx |
|---|---|---|---|---|
| Cough | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Abnormal lung auscultation | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Dyspnoea | xx (xx) | xx (xx) | xx (xx) | xx (xx) |

Note: Cough includes subjects who reported cough of any grade.

Note: Abnormal lung auscultation includes subjects with any abnormality recorded.

Note: Dyspnoea includes subjects who reported dyspnoea of any grade.

Example: SAFE\_T9
Protocol: 201791
Population: Safety


Table 3.x
Summary of Pulse Oximetry Results (Period X)

| Visit<br>Blood Oxygen | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx | Treatment 4<br>N=xx |
|---|---|---|---|---|
| Baseline | | | | |
| n | XX | XX | XX | XX |
| <80% | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| 80% to <90% | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| >=90% | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| Worst Post-Baseline Result | | | | |
| n | xx | XX | XX | XX |
| <80% | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| 80% to 90% | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| >=90% | xx (xx) | xx (xx) | xx (xx) | xx (xx) |

Example: LB16A (modified)


Population: Safety

Table 3.76

Summary of Worst Case Chemistry Results by Maximum Grade Shift Post-Baseline Relative to Baseline

(Period 1)

Test (units): Alanine Aminotransferase (IU/L)
Term: Alanine aminotransferase increased

| Treatment | Planned Time | Change | Categories [2] | | | |
|---|---|---|---|---|---|---|
| Pooled PBO (N=78) | Baseline | n | Grade 1<br>Grade 2<br>Grade 3<br>Grade 4 | xx | XX<br>XX | (xx%)<br>(xx%)<br>(xx%) |
| | Maximum Grade Shift Post<br>Baseline | n | Worsen to Grade 1 Worsen to Grade 2 Worsen to Grade 3 Worsen to Grade 4 Worsen to Grades 1 to 4 Worsen to Grades 2 to 4 Worsen to Grades 3 to 4 | XX<br>XX<br>XX<br>XX | (xx%)<br>(xx%)<br>(xx%)<br>(xx%)<br>(xx%)<br>(xx%) | |
| OTI 90mg QW (N=157) | Baseline | n | Grade 1<br>Grade 2<br>Grade 3<br>Grade 4 | xx | XX<br>XX | (xx%)<br>(xx%)<br>(xx%) |

Note: A worsening is defined as a worsening in grade relative to baseline grade. Subjects with missing baseline values are assumed to have baseline value of grade 0.

<sup>[1]</sup> Grades were derived based on numeric criteria as defined in CTCAEv5.0 and did not take into consideration of clinical signs or symptoms, concomitant medication usage which is needed for the final grade associated with the adverse event.

<sup>[2]</sup> n = number of subjects with values at the specified planned time.

Example: SAFE\_T10
Protocol: 201791
Population: Safety


Table 3.x Summary of Anti-GSK3196165 Antibodies (ADA)

| | Treatment 1 | Treatment 2 | Treatment 3 |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| aseline ADA results | | | |
| n | XX | xx | xx |
| Negative ADA | xx (xx) | xx (xx) | xx (xx) |
| Confirmed positive ADA | xx (xx) | xx (xx) | xx (xx) |
| At least one confirmed positive ADA that subsequently tested positive for Neutralising Antibodies | xx (xx) | xx (xx) | xx (xx) |
| At least one confirmed positive ADA that subsequently tested negative for Neutralising Antibodies | xx (xx) | xx (xx) | xx (xx) |

Note: A subject is considered to have a positive ADA result if they have a positive screening assay, a positive confirmation assay and a titre value. A baseline ADA result is the closest ADA sample prior to the subject receiving the first dose of GSK3196165. Only confirmed ADA positive samples were tested in the Neutralizing Antibody assay.

201791

Example: SAFE T10 (continued)

Population: Safety

Table 3.x
Summary of Anti-GSK3196165 Antibodies (ADA)

| | Treatment 1 | Treatment 2 | Treatment 3 |
|---|---|---|---|
| | N=xx | N=xx | N=xx |
| t-baseline ADA results | | | |
| n | xx | xx | xx |
| At least one confirmed positive ADA result | xx (xx) | xx (xx) | xx (xx) |
| All negative ADA results | xx (xx) | xx (xx) | xx (xx) |
| Confirmed positive ADA result that are positive for Neutralising Antibodies | xx (xx) | xx (xx) | xx (xx) |
| Confirmed positive ADA result that are negative for Neutralising Antibodies | xx (xx) | xx (xx) | xx (xx) |

Note: A subject is considered to have a positive ADA result if they have a positive screening assay, a positive confirmation assay and a titre value. A baseline ADA result is the closest ADA sample prior to the subject receiving the first dose of GSK3196165. Only confirmed ADA positive samples were tested in the Neutralizing Antibody assay.

201791

Example: SAFE\_T11
Protocol: 201791
Population: Safety


Table 3.x Summary of Binding Antibody at Each Assessment Visit

| Visit | Assay Result | · | Treatment 1 | Treatment 2 | Treatment 3 |
|---|---|---|---|---|---|
| . 1010 | - | | N=xx | N=xx | N=XX |
| Baseline | n | | XX | xx | XX |
| | Negative | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Positive | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Titre Value | Median | XX.X | XX.X | XX.X |
| | | Min. | XX | xx | XX |
| | | Max. | XX | XX | XX |
| Week 2 | n | | XX | XX | xx |
| | Negative | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Positive | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Titre Value | Median | XX.X | XX.X | XX.X |
| | | Min. | XX | xx | XX |
| | | Max. | XX | XX | xx |
| ANY TIME POST<br>BASELINE | n | | xx | xx | XX |
| | Negative | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Positive | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Persistent positive | ) | xx (xx%) | xx (xx%) | xx (xx%) |
| | Transient positive | | xx (xx%) | xx (xx%) | xx (xx%) |
| | Titre Value | Median | XX.X | xx.x | XX.X |
| | | Min. | XX | xx | XX |
| | | Max. | XX | xx | XX |

Note: The values shown at the Any Time post baseline visit are based on each subject's highest post baseline titre.

Note: Any Time Post Baseline would be positive for a subject who had negative and positive post baseline results.

Note: Transient positive is defined as a single positive immunogenic response where the previous visit is negative, that does not occur at the final study assessment and persistent positive is defined as a positive immunogenic response where the previous visit is positive of the final study assessment is positive.

Note: The titre value includes the method sample dilution of 1/10.

201791

Example: SAFE\_T12
Protocol: 201791
Population: Safety


| Visit | Assay Result | Treatment 1<br>N=xx | Treatment 2<br>N=xx | Treatment 3<br>N=xx |
|---|---|---|---|---|
| Baseline | n | XX | XX | XX |
| | Negative | xx (xx%) | xx (xx%) | xx (xx%) |
| | Positive | xx (xx%) | xx (xx%) | xx (xx%) |
| Week 2 | n | xx | XX | xx |
| | Negative | xx (xx%) | xx (xx%) | xx (xx%) |
| | Positive | xx (xx%) | xx (xx%) | xx (xx%) |
| NY TIME POST<br>BASELINE | n | xx | xx | xx |
| | Negative | xx (xx%) | xx (xx%) | xx (xx%) |
| | Positive | xx (xx%) | xx (xx%) | xx (xx%) |

Note: NAb assay result is only presented for subjects with a positive ADA assay.

Note: Any Time Post Baseline would be positive for a subject who had negative and positive post baseline results.

201791

Example: SAFE\_T13
Protocol: 201791

Population: Safety

Table 3.x Summary of Adjudicated Serious Cases of COVID-19 Infections (Period X)

| | Treatment 1<br>N=xx<br>n (%) | Treatment 2<br>N=xx<br>n (%) | Treatment 3 N=xx n (%) | Treatment 4 N=xx n (%) |
|---|---|---|---|---|
| Confirmed Cases of COVID-19 | x (x) | x (x) | x (x) | x (x) |
| Non Hospitalised (WHO grade 1 and 2) | x (x) | x (x) | x (x) | x (x) |
| Hospitalised (WHO grade 3, 4 and 5) | x (x) | x (x) | x (x) | x (x) |
| Hospitalised (WHO grade 6 and 7) | x (x) | x (x) | x (x) | x (x) |
| Death | x (x) | x (x) | x (x) | x (x) |
| Probable Cases of COVID-19 | x (x) | x (x) | x (x) | x (x) |
| Non Hospitalised (WHO grade 1 and 2) | x (x) | x (x) | x (x) | x (x) |
| Hospitalised (WHO grade 3, 4 and 5) | x (x) | x (x) | x (x) | x (x) |
| Hospitalised (WHO grade 6 and 7) | x (x) | x (x) | x (x) | x (x) |
| Death | x (x) | x (x) | x (x) | x (x) |



201791

Example: SAFE T14 Protocol: 201791


Table 1.x Summary of Common (>=2%) Adverse Events by Time from Randomisation

Time From Randomisation : [<=12 weeks / >12 weeks and <=24 weeks / >24 weeks and <=36 weeks / >36 weeks and <=52

weeks / >52 weeks 1

| | Treatment 1 | Treatment | Treatment | Treatment 4 | Treatment 5 | Treatment 6 |
|---|---|---|---|---|---|---|
| | N=xx | 2 | 3 | N=xx | N=xx | N=xx |
| | | N=xx | N=xx | | | |
| Any Adverse Event | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| XXXXX | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

201791

Example: SAFE\_T15
Protocol: 201791
Population: Safety

1:  $201\overline{7}91$  Page 1 of x

Table 3.x
Summary of COVID-19 Infections (Period X)

| | Treatment 1 (N=xx) | Treatment 2 (N=xx) | Treatment 3 (N=xx) | Treatment 4 (N=xx) |
|---|---|---|---|---|
| Any COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Any Non-Serious COVID-19<br>Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Confirmed COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Suspected COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Probable COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Any Serious COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Confirmed COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Suspected COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Probable COVID-19 Infection | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

201791

Example: SAFE\_L1
Protocol: 201791
Population: Safety

rotocol: 201791 Page 1 of n

Listing x

Listing of Neutrophils and Associated Infections Subset of Subjects who experienced grade 3 or 4 Neutropenia

Site=xxx; Subject=xxxxxx.xxxxxx; Arm=xxxxxxxxxxx;

Sex=x; Age(YEARS)=xx; Race Details=xxxxxxxx; Weight(kg)=xx.xx

| | | | | | Neu | trophils | (unit) | Associated Infections |
|---|---|---|---|---|---|---|---|---|
| Treatment/<br>Period | Visit | Analysis<br>Visit | Date | Study<br>Day | Result | Out of<br>Normal | Toxicity<br>Grade | Preferred Term/<br>VERBATIM TEXT |
| Placebo/ | SCREENING | SCREENING | XXXX-XX-XX | Х | X.XX | | | |
| 1 | BASELINE | BASELINE | xxxx-xx-xx | XX | X.XX | XXX | X | |
| | WEEK 1 | WEEK 1 | XXXX-XX-XX | XX | X.XX | XXX | X | |
| | WEEK 2 | WEEK 2 | xxxx-xx-xx | XX | X.XX | | | |
| | UNSCHEDULED | WEEK 2 | xxxx-xx-xx | XX | X.XX | XXX | X | |
| | WEEK 4 | WEEK 4 | xxxx-xx-xx | XX | X.XX | | | |

Note: Lower Limit of Normal: xx, Upper Limit of Normal: xx

# Signature Page for 201791 TMF- 14870227 v 2.0

| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 05-Aug-2022 09:36:57 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 05-Aug-2022 10:08:25 GMT+0000 |

Signature Page for TMF-14870227 v2.0